# Predicting the SURPASS-CVOT Cardiovascular Outcome Trial in Healthcare Claims Data

NCT07099718

30<sup>th</sup> July 2025

| Title | Comparative effectiveness of semaglutide and tirzepatide in patients at low, moderate, and high cardiovascular risk with type 2 diabetes and obesity: Predicting the SURPASS-CVOT Cardiovascular Outcome Trial in Healthcare Claims Data |
|---|---|
| Research question & Objectives | This study is part of a three-stage project evaluating the comparative effectiveness of semaglutide and tirzepatide in patients at low, moderate, and high cardiovascular risk with type 2 diabetes and obesity: The SURPASS-CVOT trial evaluates the effect of tirzepatide vs dulaglutide on the risk of major adverse cardiovascular event (MACE) among patients with type 2 diabetes, overweight, and |
| | an established cardiovascular disease. |
| Protocol version | Version 2 |
| Last update date | July 30, 2025 |
| Contributors | Primary investigators contact information: Dr. Nils Krüger, nkruger1@bwh.harvard.edu Dr. Shirley Wang, swang1@bwh.harvard.edu Contributor names: Dr. Krüger implemented the study design in the Aetion Evidence Platform. He is responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform. |
| Study registration | Site: clinicaltrials.gov Identifier: NCT07088718 |
| Sponsor | Organization: N/A<br>Contact: N/A |
| Conflict of interest | Dr. Krüger has no conflict of interest. Dr. Wang has consulted for Cytel Incs, Exponent Inc, and MITRE an FFRDC for Centers for Medicare and Medicaid for unrelated work. |

# Table of contents

| I. Title Page | 1 |
|---|---|
| 2. Abstract | 4 |
| 3. Amendments and updates | 4 |
| 1. Rationale and background | 5 |
| 5. Research question and objectives | 5 |
| Table 2. Primary and secondary research questions and objectives | 5 |
| 5. Research methods | 7 |
| 6.1 Study design | 7 |
| 6.2 Study design diagram when following the eligibility criteria of the SURPASS-CVOT trial (Figure 1). | 8 |
| 6.3 Setting | 9 |
| 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population | 9 |
| 6.3.2 Context and rationale for study inclusion criteria: | 9 |
| 6.3.3 Context and rationale for study exclusion criteria | 9 |
| 6.4 Variables | 9 |
| 6.4.1 Context and rationale for exposure(s) of interest | 9 |
| 6.4.2 Context and rationale for outcome(s) of interest | 9 |
| 6.4.3 Context and rationale for follow-up | 10 |
| Table 1. Operational Definitions of follow-up | 10 |
| 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications) | 11 |
| Table 2. Operational Definitions of Covariates | 11 |
| 6.5 Data analysis | 40 |
| 6.5.1 Context and rationale for analysis plan | 40 |
| Table 3. Primary, secondary, and subgroup analysis specification | 40 |
| Table 4. Sensitivity analyses – rationale, strengths and limitations | 42 |
| 6.5.2 Comparison of Results Between Database Studies and RCTs | 43 |
| 6.6 Data sources | 43 |
| 6.6.1 Context and rationale for data sources | 43 |
| Table 5. Metadata about data sources and software | 44 |
| 6.7 Data management | 44 |
| 6.8 Quality control | 46 |
| 6.9 Study size and feasibility | 47 |
| 7. Limitation of the methods | 47 |

| 3. Protection of human subjects | 47 |
|---|---|
| 9. References | 47 |
| LO. Appendices | 49 |
| 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment | 49 |
| 2 Code algorithms | 49 |
| 3 Flowchart for cohort assembly | 49 |
| 4 1st feasibility assessment | 49 |
| 5 2nd feasibility assessment | 49 |
| 6 Balance Assessment - PS Distribution and C-Statistic | 49 |
| 7 Balance Assessment - Table 1 | 49 |

## 2. Abstract

This is a non-randomized, non-interventional study that is part of the *Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims*: Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to emulate, as closely as is possible in healthcare insurance claims data, the SURPASS-CVOT trial (NCT04255433) described below. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides guidance on the reference standard treatment effect estimate. However, failure to replicate RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons and does not provide information on the validity of the original RCT finding.

The SURPASS-CVOT trial is a non-inferiority trial that aims to evaluate the effect of tirzepatide, a dual glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 receptor agonist (GLP-1-RA), vs dulaglutide, a GLP-1-RA, on time to first occurrence of any major adverse cardiovascular event (MACE), defined as cardiovascular death, myocardial infarction, or stroke among patients with T2DM and an established cardiovascular disease (CVD). In addition, the trial aims to determine noninferiority with a magnitude of difference that also supports superiority against putative placebo and for superiority to dulaglutide will be performed.¹ With estimated study completion in summer 2025, results of the trial are yet to be announced. Therefore, we aim to predict the results of the SURPASS-CVOT trial by emulating its design with protocol registration and statistical analysis conducted before the results of the trial are made public.²

The database study designed to emulate the SURPASS-CVOT trial will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs dulaglutide on the composite end point of all-cause mortality, myocardial infarction, or stroke. Clinical guidelines during the study period recommended both agents under investigation as second-line options for glucose lowering and were similarly costly.

The study will use two data sources: Optum Clinformatics and Merative MarketScan. Optum: Study period between May 13, 2022 to February 28, 2025.

# 3. Amendments and updates

| Version date | Version number | Section of protocol | Amendment or update | Reason |
|---|---|---|---|---|
| | 2 | 6.4.4 | Added three covariates: Heart failure, acute heart failure, microalbuminuria/proteinuria. Split covariate for "Myocardial infarction" into "Acute myocardial infarction" and "Old myocardial infarction". | These covariates were part of the original analytical framework and were inadvertently omitted/changed in the initial version. Their inclusion corrects this oversight. |
| 15 <sup>th</sup> May 2025 | 1 | All sections | This emulation of SURPASS-CVOT is part of a 3-stage study that aims to compare tirzepatide vs semaglutide in patients at cardiovascular risk with type 2 diabetes and obesity. This project is independent from other projects that have also emulated SURPASS-CVOT for unrelated study objectives. Differences in results between independently conducted SURPASS-CVOT emulations may occur due to the differences in objectives and design/implementation. | |

# 4. Rationale and background

The purpose of this protocol is to specify the emulation of the SURPASS CVOT trial (NCT04255433). Tirzepatide became available on May 13, 2022, when it was approved to treat T2DM.<sup>3</sup> A year later, on November 8, 2023 tirzepatide was approved for chronic weight management in adults with obesity or overweight who also have at least one weight-related comorbid condition, such as hypertension, dyslipidemia, T2DM, obstructive sleep

apnea, or CVD. On December 20 2024, tirzepatide was approved to treat moderate to severe obstructive sleep apnea (OSA) in adults with obesity, to be used in combination with a reduced-calorie diet and increased physical activity.

Dulaglutide was approved on September 18, 2014 to improve glycemic control in adults with T2DM.<sup>4</sup> On February 21, 2020 FDA approved dulaglutide to reduce the risk of major adverse cardiovascular events in adults with T2DM who have established CVD or multiple cardiovascular risk factors.<sup>5</sup> In the same year, on September 9, 2020 an additional dosing regimen was approved.<sup>6</sup> Finally, on November 17, 2022, dulaglutide was approved for use in pediatric patients aged 10 years and older.

The SURPASS-CVOT trial enrolled 13299 participants between May 29, 2020 - June 27, 2022. The event-driven trial has planned a mean follow-up duration of approximately 4 years until at least 1,615 participants experience at least one component of adjudication-confirmed MACE. The primary analysis examines noninferiority of tirzepatide vs dulaglutide with an upper bound of the 95% confidence interval (CI) of the hazard ratio (HR) below 1.05 also indicating superiority of tirzepatide vs a putative placebo. An upper bound of the 95% CI of the HR of ≥1.05 but <1.23 for tirzepatide vs dulaglutide will indicate noninferiority and proven safety of tirzepatide to putative placebo. If the upper 95% CI is <1.05 in the primary analysis, a formal analysis for superiority of tirzepatide vs dulaglutide will be performed. Estimated annualized event rate for MACE in the dulaglutide treatment group was expected to be 3.5%, providing approximately 90% power to establish superiority.¹

# 5. Research question and objectives

#### Table 2. Primary and secondary research questions and objectives

#### A. Primary research questions and objectives

| Objective: | To evaluate the comparative effect of tirzepatide vs dulaglutide on time to first occurrence of |
|---|---|
| | MACE (all-cause mortality, myocardial infarction, or death) in patients with T2DM and an |
| | stablished CVD when following the eligibility criteria of the SURPASS-CVOT trial. |
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to dulaglutide at preventing all-cause |
| | mortality, myocardial infarction, or stroke in individuals with T2DM and an established CVD. In |
| | ddition, superiority to dulaglutide will be tested if non-inferiority is achieved. |
| Population (mention key inclusion-exclusion | Individuals aged 40 years or older with T2DM and an established CVD. |
| criteria): | |
| Exposure: | Tirzepatide. |
| Comparator: | Dulaglutide. |
| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |

| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, |
|---|---|
| | discontinuation (45 days grace and risk window), switch between the arms, nursing home |
| | admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |
| Main measure of effect: | Hazard ratio. |

# **B.** Secondary research questions and objectives

| Objective: | To evaluate the comparative effect of tirzepatide vs dulaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients |
|---|---|
| | meeting the eligibility criteria of the SURPASS-CVOT trial. |
| Hypothesis: | We hypothesize that tirzepatide will be non-inferior to dulaglutide at preventing all-cause mortality, myocardial infarction, or stroke in individuals with T2DM and an established CVD. In addition, superiority to dulaglutide will be tested if non-inferiority is achieved. |
| Population (mention key inclusion-exclusion criteria): | Individuals aged 40 years or older with T2DM and an established CVD. |
| Exposure: | Tirzepatide. |
| Comparator: | Dulagluitde. |
| Outcome: | The individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, and stroke. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured from inpatient hospitalizations and death. |
| Main measure of effect: | Hazard ratio. |

| Objective: | To evaluate the effect of tirzepatide vs dulaglutide on negative control outcomes, including (1) |
|---|---|
| | hernia and (2) lumbar radiculopathy in patients typically treated in clinical practice who are at |
| | cardiovascular risk with type 2 diabetes and overweight. |
| Hypothesis: | We hypothesize that tirzepatide will not have a different effect from dulaglutide. |
| Population (mention key inclusion-exclusion | Individuals aged 40 years or older with T2DM and an established CVD. In addition, patients will |
| criteria): | be excluded with recent hernia or lumbar radiculopathy prior to the follow-up time window (45 |
| | days) when studying the negative outcome hernia or lumbar radiculopathy, respectively. |

| Exposure: | Tirzepatide. |
|---|---|
| Comparator: | Dulaglutide. |
| Outcome: | parate analyses for hernia and lumbar radiculopathy. |
| Time (when follow-up begins and ends): | 1 day after cohort entry date until the first of outcome, disenrollment, end of study period, discontinuation (45 days grace and risk window), switch between the arms, nursing home admission, or start of any other GLP-1-RA. |
| Setting: | The outcome will be measured using diagnosis codes in an inpatient or outpatient setting. |
| Main measure of effect: | Hazard ratio. |

# 6. Research methods

## **6.1 Study design**

Research design (e.g. cohort, case-control, etc.): New user active-comparator cohort study.

**Rationale for study design choice:** The new user active-comparator design is a powerful design that may be able to address confounding by indication. It accomplishes this, in large part, through judicious selection of an appropriate active-comparator group.<sup>7,8</sup> While selection of an appropriate comparator in the design phase is crucial, cohort studies often require additional adjustment of measurable confounders. A common method for adjusting for confounding is via a propensity score.

# **6.2 Study design diagram** when following the eligibility criteria of the SURPASS-CVOT trial (Figure 1).

Figure 1. Exposure-based cohort entry where the cohort entry date is selected after application of exclusion criteria



#### 6.3 Setting

#### 6.3.1 Context and rationale for definition of time 0 (and other primary time anchors) for entry to the study population

Time 0 in the database study was defined to emulate randomization to tirzepatide vs dulaglutide in the trial design. See appendix tables 1 and 2a for operational definitions and detailed code algorithms.

#### **6.3.2** Context and rationale for study inclusion criteria:

Study inclusion criteria were defined to emulate the inclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendix 3.

#### 6.3.3 Context and rationale for study exclusion criteria

Study exclusion criteria were defined to emulate the exclusion criteria for the trial. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. A flowchart of the study cohort assembly is provided in appendix 3.

#### **6.4 Variables**

## **6.4.1** Context and rationale for exposure(s) of interest

The exposure and comparator were defined to emulate the agents compared for the trial, tirzepatide vs dulaglutide (active-comparator). See appendix tables 1 and 2 for operational definitions and detailed code algorithms.

## **Algorithm to define duration of exposure effect:**

Assuming the effect of the drug lasts for 45 days after the last day's supply, we allow a 45 days gap between the dispensation (grace period) and also add 45 days at the end of the last day's supply (exposure risk window).

## 6.4.2 Context and rationale for outcome(s) of interest

The primary outcome for the database study was defined to emulate the primary outcome of the trial, i.e., MACE (composite of cardiovascular death, myocardial infarction, or stroke). Due to the inability to capture cause of death in our emulation, we modified the MACE outcome to capture all-cause mortality, myocardial infarction, or stroke. See appendix tables 1 and 2 for operational definitions and detailed code algorithms. Optum includes death information from the inpatient discharged dead status, social security death master file, and deaths scraped from obituaries or other sources. MarketScan includes information from the inpatient discharged dead status as well as social security death master file. PPV for myocardial infarction

using ICD9 codes was 94%.<sup>9-11</sup> PPV for ischemic stroke using ICD9 codes was 95%. Both of the above ICD9 codes were mapped to ICD10, but no validation study was performed.<sup>12</sup>

Secondary outcomes from the trial that will be evaluated include:

1. Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, and stroke.

Control outcomes of interest include:

- 1. Hernia (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs dulaglutide.
- 2. Lumbar radiculopathy (excluding patients with recent outcome prior to the follow-up time window). This is a negative control outcome where no difference in effect is expected for tirzepatide vs dulaglutide.

#### 6.4.3 Context and rationale for follow-up

Both on-treatment (OT) and intention-to-treat (ITT) analyses will be conducted. Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the OT analysis will be the primary analysis. The OT analysis targets the relative hazard of outcomes while on treatment and may more closely emulate the effect observed in highly adherent trial participants. Both OT and ITT analyses will be conducted with up to 1-year follow-up.

**Table 1. Operational Definitions of follow-up** 

| follow-up start | Day 1 | |
|---|---|---|
| follow-up end¹ | Select<br>all that<br>apply | Specify |
| Date of outcome | Yes | |
| Date of death | Yes | Part of the primary outcome. |
| End of observation in data | Yes | Date of disenrollment. |
| Day X following index date<br>(specify day) | Yes | Day 365. |

| End of study period (specify date) | Yes | Different dates for different databases (Optum: February 28, 2025; MarketScan: December 31, 2023). |
|---|---|---|
| End of exposure<br>(specify operational details,<br>e.g. stockpiling algorithm, grace<br>period) | Yes | 45 days grace window and 45 days risk window. |
| Date of add to/switch from exposure (specify algorithm) | Yes | Date of augmentation or switching from an exposure to a comparator and vice versa. |
| Other date (specify) | Yes | Censor upon nursing home admission or starting any other GLP-1-RA. |

<sup>&</sup>lt;sup>1</sup> follow-up ends at the first occurrence of any of the selected criteria that end follow-up.

# 6.4.4 Context and rationale for covariates (confounding variables and effect modifiers, e.g. risk factors, comorbidities, comedications)

We identified a series of covariates that were likely confounders due to being strong risk factors for the primary outcome that were associated with choice of treatment. These include demographics, disease severity related variables, comorbid conditions, comedications, frailty, healthcare utilization and markers of health seeking behaviour.

**Table 2. Operational Definitions of Covariates** 

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Demographics | | | | | | | | | |
| Age | Cohort entry<br>year – year of<br>birth, (last<br>observed<br>value in the<br>baseline) | Continuous | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | n/a |


| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, 0] | Inpatient | ICD-10-CM | Primary | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pancreatitis | | | | | | | | | |
| | | Binary | [-365, 0] | Inpatient | ICD-10-CM | Primary | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Bowel obstruction | | | | | | | | | |
| | | Binary | [-365, 0] | Any | ICD-10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Gastroparesis | | | | | | | | | |
| Diabetes medication | ons | | | | | | | | |
| Number of antidiabetic drugs on CED | | Continuous | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of metformin | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| insulin | | | | | | | Reference:<br>Dulaglutide | | |
| Concomitant use or initiation of sulfonylureas | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of DPP4i | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of SGLT2i | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Concomitant use or initiation of other glucose-lowering drugs | | Binary | [0, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of metformin | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of insulin | | | | | | | | | |
| Past use of sulfonylureas | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Suronylareas | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of DPP4i | | | | | | | | | |
| | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Past use of SGLT2i | | | | | | | | | |
| Past use of other glucose-lowering drugs | | Binary | [-365, -1] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart failure medic | cations | | | | | | | | |
| ACEi / ARB | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Dulaglutide | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| ARNI | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Thiazides | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Beta-blockers | | | | | | | | | |
| Calcium channel | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| blockers | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Digoxin / Digitoxin | | | | | | | | | |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Loop diuretics | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Other diuretics | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Intravenous diuretics | | | | | | | Daiagianae | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Nitrates | | | | | | | | | |
| Other medications | ; | <b>_</b> | <b>_</b> | , | | | - | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-arrhythmics | | | | | | | | | |
| Statins | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Dulaglutide | | |
| PCSK9 inhibitors<br>and other lipid-<br>lowering drugs | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antiplatelet agents | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Oral<br>anticoagulants | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| COPD/Asthma<br>medication | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| NSAIDs | | | | | | | | | |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Oral | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Osteoporosis agents (incl. bisphosphonates) | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Opioids | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Anti-depressants | | | | | | | | | |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Antipsychotics | | | | | | | | | |
| Anxiolytics/hypnot<br>ics,<br>benzodiazepines | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Medication for dementia | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Urinary tract infections antibiotics | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| | | Binary | [-365, 0] | n/a | generic | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Laxatives | | | | | | | | | |
| Healthcare utilizat | ion markers | | | | | | | | |
| Number of distinct<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of office<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Number of<br>endocrinologist<br>visits, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>cardiologist visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of internal<br>medicine/family<br>medicine visits,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Electrocardiogram<br>s, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>Echocardiograms,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pharmacy out-of-<br>pocket cost,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Unique brand<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Unique generic<br>medications,<br>median (iqr), mean<br>(sd)** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Ratio of unique<br>brand to generic<br>medications,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Healthy behavior n | narkers | | | | | | | | |
| Colonoscopy /<br>Sigmoidoscopy | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Flu vaccine /<br>Pneumococcal<br>vaccine | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Pap smear test | | | | | | | | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| PSA test | | | | | | | | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Fecal occult blood<br>test | | | | | | | Dulagiutide | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Bone mineral density tests | | | | | | | Dulagiutide | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Mammograms | | | | | | | | | |
| | | Binary | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Telemedicine | | | | | | | | | |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Laboratory and dia | gnostic tests | <u> </u> | | , | • | | | , | <del> </del> |
| Number of HbA1c<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of lipid<br>panels, median<br>(iqr), mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>creatinine tests,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of<br>natriuretic peptide<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Number of urine<br>tests, median (iqr),<br>mean (sd) | | Continuous | [-365, 0] | Any | CPT/HCPCS | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Lab values | | | | | | | | | |
| I II- A 1 - ** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| HbA1c** | | 0 1: | 1 205 01 | , | , | , | _ | , | Annandia |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Glucose** | | | | | | | | | |
| | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Creatinine** | | | | | | | | | |
| Systolic blood<br>pressure** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Hoove wat - ** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Heart rate** | | 0 | 1 205 01 | /- | 10/0 | | F | /- | Appendix |
| BMI** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Dulaglutide | | |
| eGFR** | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| LDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| HDL** (mg/dl;<br>mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Total cholesterol**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Triglyceride**<br>(mg/dl; mean, sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| Burden of comorbi | dities | | | | | | | | |
| Combined comorbidity score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Gagne et al.,<br>Sun et al. <sup>13,14</sup> |
| comorbidity score | | Continuous | [-365, 0] | Any | ICD10-CM | Any | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Kim et al. <sup>15</sup> |
| Frailty score | | | | | | | | | |
| Baseline hospitaliz | ations and hos | pital metrics | • | • | | | | | |
| Number of any<br>hospitalization,<br>median (iqr), mean<br>(sd) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 91<br>days; n (%) | | Binary | [-91, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Any hospitalization<br>within prior 92-<br>365 days; n (%) | | Binary | [-365, -92] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |

| Characteristics | Details | Type of<br>variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement<br>characteristics<br>/<br>validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| 0, 1, >1<br>hospitalizations<br>(any) | | Continuous | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Hospitalization for heart failure | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Emergency<br>department visits | | Binary | [-365, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | Appendix,<br>Covariate –<br>Algorithm |
| Calendar year of co | ohort entry | <b>-</b> | 1 | 1 | 1 | 1 | 1 | ı | |
| | , | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | n/a |
| 2022 | | | 10.01 | , | , | , | | , | , |
| 2022 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | n/a |
| 2023 | | | 10.01 | , | | , | | | , |
| 2024 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide | n/a | n/a |

| Characteristics | Details | Type of variable | Assessmen<br>t window | Care<br>Settings <sup>1</sup> | Code Type <sup>2</sup> | Diagnosi<br>s<br>Position <sup>3</sup> | Applied to study populations: | Measurement characteristics / validation | Source for algorithm |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Reference:<br>Dulaglutide | | |
| 2025 | | Categorical | [0, 0] | n/a | n/a | n/a | Exposure:<br>Tirzepatide<br>Reference:<br>Dulaglutide | n/a | n/a |

 $<sup>{}^{1}\</sup>text{IP}$  = inpatient, OP = outpatient, ED = emergency department, OT = other, n/a = not applicable

## 6.5 Data analysis

## **6.5.1 Context and rationale for analysis plan**

The studies will use a propensity score (PS) 1:1 nearest neighbor matching with a caliper of 0.01 on the propensity score scale. The propensity score will be estimated as the probability of initiating tirzepatide vs dulaglutide given the baseline patient characteristics using multivariable logistic regression models. As diagnostics for PS models, the study will evaluate distributional covariate balance using standardized differences and c-statistics post-matching. The study will estimate the hazard ratio for tirzepatide vs dulaglutide on MACE outcome in the matched population using a Cox proportional hazards model.

### Table 3. Primary, secondary, and subgroup analysis specification

#### A. Primary analyses

| Hypothesis: | Tirzepatide does not increase the risk of a composite of death, myocardial infarction, or stroke in patients with |
|---|---|
| | T2DM and an established CVD when following the eligibility criteria of the SURPASS-CVOT trial. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |

<sup>&</sup>lt;sup>2</sup>See appendix for listing of clinical codes for each study parameter

<sup>&</sup>lt;sup>3</sup> Specify whether a diagnosis code is required to be in the primary position (main reason for encounter)

<sup>\*</sup>Available for Optum Clinformatics and Medicare

<sup>\*\*</sup>Not used in the PS model

| Outcome: | Composite of all-cause mortality, myocardial infarction, or stroke. |
|---|---|
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

# **B.** Secondary Analyses

| Hypothesis: | Tirzepatide does not increase the risk of occurrence of the individual components of the primary endpoint, i.e., |
|---|---|
| | all-cause mortality, myocardial infarction, or stroke in patients with T2DM and an established CVD when |
| | following the eligibility criteria of the SURPASS-CVOT trial. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke. |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards for all-cause mortality, Aalen-Johansen estimator for myocardial |
| (provide details or code) | infarction and stroke to account for the competing risk of death. |
| | Follow-up time * status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting |
| | algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity |
| | score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple |
| | imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | List all subgroups |
| | N/A. |

| Hypothesis: | Tirzepatide vs dulaglutide has no effect on risk of negative control outcomes compared to dulaglutide. |
|---|---|
| | Negative control outcomes include (1) hernia and (2) lumbar radiculopathy. |
| Exposure contrast: | Tirzepatide vs dulaglutide. |
| Outcome: | Separate analyses for each negative control outcome, including hernia and lumbar radiculopathy |
| Analytic software: | Aetion, SAS 9.4, R.4.4.0, Python 3.13.3 |
| Model(s): | Outcome model: Cox proportional hazards |
| (provide details or code) | Follow-up time*status(0) = exposure |
| Confounding adjustment method | Name method and provide relevant details, e.g. bivariate, multivariable, propensity score weighting (specify weighting algorithm ratio and caliper), propensity score weighting (specify weight formula, trimming, truncation), propensity score stratification (specify strata definition), other. |
| | 1:1 Propensity score nearest-neighbor matching with a caliper of 0.01 on the propensity score scale. |
| Missing data methods | Name method and provide relevant details, e.g. missing indicators, complete case, last value carried forward, multiple imputation (specify model/variables), other. |
| | Assumption that if no relevant claims diagnoses/procedures are present, the condition is not present. |
| Subgroup Analyses | |

Table 4. Sensitivity analyses – rationale, strengths and limitations

| | What is being varied? How? | Why?<br>(What do you expect to<br>learn?) | Strengths of the sensitivity analysis compared to the primary | Limitations of the sensitivity analysis compared to the primary |
|---|---|---|---|---|
| Negative control outcomes, including hernia, lumbar radiculopathy | We evaluate negative control outcomes of hernia and lumbar radiculopathy, where no causal effect is expected from tirzepatide, or dulaglutide. | We will evaluate the potential impact of residual confounding on this outcome for which there is not expected to be a causal effect | The evaluates the robustness of the interpretation of the primary analysis by evaluating the potential magnitude of unmeasured confounding | This analysis assumes that the confounding structure is the same or similar for the negative control outcome as the outcome of interest |
| Effect estimation in individuals with HbA1c measurement. | The population will be restricted to individuals with a HbA1c measurement in the 120 days before cohort entry. | To assess the impact of restricting to individuals with HbA1c measurement and including HbA1c in the PS model. | Includes baseline glycemic information as captured in laboratory HbA1c measurements. | This approach highly restricts the number of eligible individuals under study and thereby the statistical power of the analysis. |
| As-started analyses | To address potential informative censoring. | We will consider the first-<br>used medication for 365 | Reflects follow-up regimen of RCT. | Persistence of drug use is shorter in clinical practice |

| (observational | days without considering | whereas adherence is typically |
|---|---|---|
| analogue to | drug discontinuation or | higher in RCTs. Therefore, we |
| intention-to-treat) | switching, mimicking an | expect the estimated effects |
| to address | "intention-to-treat" | will be diluted toward the null, |
| potential | approach. | underestimating the true |
| informative | | treatment effect had patients |
| censoring. | | remained on therapy. |

#### 6.5.2 Comparison of Results Between Database Studies and RCTs

We attempt to predict the results of the SURPASS-CVOT trial. Failure to predict the RCT findings is not necessarily indicative of the inadequacy of the healthcare claims data for emulation for a range of possible reasons, nor does failure to predict trial results provide information about the validity of the respective trial. Once trials results are available, assessment of concordance in results between the database study-trial pair will use the metrics previously implemented in the RCT-DUPLICATE initiative, namely statistical significance agreement, estimate agreement, and standardized difference agreement. In this project, "full" statistical significance agreement was defined by estimates and confidence intervals on the same side of null; estimate agreement was defined by whether estimates for the trial emulation fell within the 95% CI for the trial results; standardized difference agreement between treatment effect estimates from trials and emulations was defined by standardized differences |z| < 1.96 ( $z = \frac{(\theta_{BCT}-\theta_{BWE})}{(\sqrt{\theta^2_{BCT}-\theta^2_{BWE})}}$ ) where are the treatment effect estimates and the  $\hat{\sigma}^2$  are associated variances). In addition, "partial" significance agreement was defined as meeting pre-specified non-inferiority criteria even though a more highly powered database study may have indicated superiority. 16,17

#### 6.6 Data sources

#### 6.6.1 Context and rationale for data sources

**Reason for selection:** The study will be conducted in 2 US health care claims databases: Optum Clinformatics (2022-2025), and Merative MarketScan (2022-2023). Data from the Merative MarketScan database will only be included if sufficient sample size can be accrued.

**Strengths of data source(s):** Each data source contains deidentified, longitudinal, date-stamped information on patient enrollment, demographics, inpatient/outpatient diagnosis and procedures, admission and discharge dates, and medication dispensation. The death data is captured in the Optum database from inpatient discharge status, social security death master file, and deaths scraped from obituaries or other sources. The death data in MarketScan is captured from the social security death master file and inpatient discharge status. It is recognized that the social security death master file has high specificity and positive predictive value for deaths. While this data resource has under captured deaths since 2011, the capture of deaths is not expected to be differential between compared exposure groups.

Limitations of data source(s): Patient healthcare encounters are only observable when they are enrolled in an insurance plan that contributes to the database. Patients may change insurance plans for multiple reasons. Both Optum Clinformatics and Merative MarketScan are primarily employer based insurance databases where patients may disenroll with job changes. In claims data, dispensing data for inpatient medication is unavailable. Diagnoses reflect billing practices, therefore algorithms (preferably validated) are needed for accurate phenotyping of patient conditions. Services that are not covered by insurance do not appear in the data. The trial evaluated cardiovascular deaths, however we will evaluate all-cause mortality in the emulation because most deaths in this cohort of patients at high cardiovascular risk will be related to cardiovascular reasons, the cause of death is not recorded for databases not linked to NDI, and the performance of NDI at identifying cardiovascular causes of death may be suboptimal. <sup>18</sup>

### **Data source provenance/curation:**

Information about Optum Clinformatics and Merative MarketScan can be found in data dictionaries and user guides that are provided to clients.

Table 5. Metadata about data sources and software

| | Data 1 | Data 2 |
|---|---|---|
| Data Source(s): | Optum Clinformatics | Merative MarketScan |
| Study Period: | 13 <sup>th</sup> May 2022 | 13 <sup>th</sup> May 2022 |
| Eligible Cohort Entry Period: | February 28, 2025 | December 31, 2023 |
| Data Version (or date of last update): | April 2025 | Mortality Cut Set A<br>Received 2024-03-01 |
| Data sampling/extraction criteria: | n/a | n/a |
| Type(s) of data: | Administrative claims | Administrative claims |
| Data linkage: | n/a | n/a |
| Conversion to CDM*: | n/a | n/a |
| Software for data management: | Aetion Evidence Platform® (2025) | Aetion Evidence Platform® (2025) |

<sup>\*</sup>CDM = Common Data Model

#### **6.7 Data management**

<u>Tracking data:</u> The Data Use Agreement (DUA) Custodian (Principal Investigator) and the Division Operations Manager (Winta Tekle) are responsible for receiving and creating a record of new data associated with the given request. The Operations Manager is responsible for all indexing and archiving of documents and electronic media related to data that the Division receives and will log data location, data contents, and associated DUA and Institutional Review Board (IRB) numbers in the Division's centralized tracking system.

<u>Handling and storage:</u> In-scope data will be stored utilizing Mass General Brigham approved information systems – i.e., Division servers and Mass General Brigham network storage.

Archiving: Data retention and any removal will be executed by the Division Operations Manager (Winta Tekle) and Data Manager (Todd MacGarvey). The Division follows Mass General Brigham enterprise record retention policies and follow the terms of the agreement through which the in-scope data was received.

Information security: The Division follows Mass General Brigham's Enterprise Information Security Program (EISP). The EISP helps by providing assurance that Mass General Brigham information and information systems are protected from unauthorized access, use, disclosure, duplication, modification, or destruction in order to maintain their confidentiality, integrity, and availability. To that end, the EISP policies, standards and procedures create an information security framework that is aligned with the recommendations of the International Organization for Standardization's (ISO) publication 27001 and the National Institute of Standards and Technology's (NIST) publication 800-53 Family of Controls and MGB regulatory and legal requirements (as a HIPAA covered entity).

Mass General Brigham workforce members are required to complete new workforce privacy and information security training upon hire and annually thereafter. Refresh training is provided as appropriate. Mass General Brigham workforce members are required to review and sign a Confidentiality Agreement upon hire and annually thereafter. Additionally, we follow Enterprise Information Security and Privacy policies, including Managing Workforce Members Information Security Responsibilities Policy, which was developed to help assure that Mass General Brigham workforce members are competent and eligible to support the information security responsibilities associated with their role. Mass General Brigham workforce, including Division staff, are required to comply with Enterprise Information Security and Privacy Policies.

<u>Facilities:</u> The research team uses a highly secure, state-of-the-art, computing facility housed at Mass General Brigham's Corporate Data Centers in Needham and Marlborough, Massachusetts as well as Amazon Web Services (AWS). We maintain redundant storage for maximal data integrity and high-speed data access.

The Division uses Mass General Brigham corporate provisioned servers to analyze and store data in connection with this project. There are strict access controls enforced by technical means to ensure that only study staff who have been approved to conduct data analyses and contracted data engineers are able to access data (e.g., Mass General Brigham Authentication (Active Directory) utilized; auditing, logging, and monitoring enabled; firewalls enabled; etc.). All Division servers used in this study are accessible to only authorized staff only through the MGB network and utilizing VPN as appropriate (i.e., users must be on the network and logged into VPN to access). Mass General Brigham has a network information security monitoring team and in-scope servers are enrolled in enterprise security tools (e.g., vulnerability scanning service, antivirus, etc.).

The Division also uses AWS. In-scope AWS services / resources have undergone review and assessment by Mass General Brigham's Information Security Risk Assessment Team / InfoSec Risk Management Team as required and in alignment with NIST 800-30: Guide for Conducting Risk Assessments. In-scope AWS servers are for our exclusive use (reserved instances), are covered under our organization's Business Associate Agreement with AWS. In-scope servers are housed in anonymous facilities that are not branded as AWS facilities. Physical access is strictly controlled both at the perimeter and at building ingress points by professional security staff utilizing video surveillance, intrusion detection systems, and other electronic means.

Security attributes and controls for the Division's use of in-scope AWS in connection with this project include: encryption at rest and in transit (industry standard AES-256 encryption, SSL/TSL), anti-malware, latest OS updates and patches as well as anti-virus; multi-factor authentication (MFA), Identity and Access Management, including SSO; auditing and logging; principle of least privilege, including for traffic and ports (e.g., deny all default configurations), use of VPC enabled Step functions, etc.; separation between environments; minimum necessary (out of the box AWS roles are not used as they can be overly permissive); all data would reside in the US domestic regions – use only US east HIPAA compliant region; performance monitoring enabled and reviewed as per internal processes; passwords compliant with enterprise password policy and, as appropriate, more protective password requirements; etc. Our Division's AWS use is also subject to ongoing evaluation and monitoring as well – e.g., vulnerability scanning and management, access review, etc.

A data file list will be maintained in Amazon S3 and tracked through Cloudtrail and Cloudwatch. Reporting of data file availability for any file stored in an S3 bucket will be controlled by MGB.

Amazon EC2, Amazon EBS, and Amazon VPC are integrated with AWS CloudTrail, a service that provides a record of actions taken by a user, role, or an AWS service in Amazon EC2, Amazon EBS, and Amazon VPC. CloudTrail captures all API calls for Amazon EC2, Amazon EBS, and Amazon VPC as events, including calls from the console and from code calls to the APIs. MGB IT/security staff have full access to CloudTrail to ensure that CloudTrail monitoring is available at all times. Amazon CloudWatch Events delivers a near-real-time stream of system events that describe changes in AWS resources. Amazon CloudTrail can log, continuously monitor, and retain account activity related to actions across the MGB AWS infrastructure. CloudTrail provides event history of MGB AWS account activity. This event history simplifies security analysis, resource change tracking, and troubleshooting and complies with requirements to ensure the data file inventory is controlled by MGB.

<u>Backups:</u> Backups are created using industry recognized Cryptographic mechanisms (e.g., 256-bit AES encryption) as appropriate and required. Data are backed up within the MGB network from the MGB Needham data center to the MGB Marlborough data center via replication/mirroring and volume-level snapshots. AWS Backup supports both instance-level backups as Amazon Machine Images (AMIs) and volume-level backups as separate snapshots based on the resource tags. AMIs allow MGB IT and security staff to create backups of all S3 and EC2 instances.

In addition to the safeguards listed above, the Division follows enterprise privacy and information security policies and maintains internally procedures in connection with this project to safeguard the data in connection with this project as appropriate and required including: Physical Security and Environmental Controls for Electronic Information Policy; IT Access Control Standards for Users policy; Safeguarding Fax Copiers Printers Telephone Use and Pagers; Physical Removal and Transport of Protected Health Information and Personal Information policy, etc.

### **6.8 Quality control**

Senior Programmers and Research Specialists perform QA/QC on raw or common data model converted data via SAS/R/Aetion software. The protocol will be iteratively developed and pre-specified data checks including feasibility counts and balance on baseline covariates will be conducted with outputs reviewed by MGB team members. Team members will review code lists to ensure fidelity to intended algorithms.

#### 6.9 Study size and feasibility

See appendix 4 and appendix 5 (feasibility, weighting on age, sex, comorbidity score as well as all predefined propensity score variables). Propensity score distribution plots with c-statistics are available in appendix 6. Table 1 showing prevalence of baseline characteristics and standardized differences in distribution are available in appendix 7. Additional diagnostic evaluations, including balance assessments of laboratory and clinical examination test results not included in the propensity score as well as assessment of heart failure-related medication after follow-up, will be conducted to assess potential residual confounding and divergence of treatment over time.

#### 7. Limitation of the methods

As we are using secondary data and the data were not collected for research purposes, some important variables may not be collected or will be measured imperfectly. We have selected validated algorithms when possible and we have created proxies for important variables that are not directly captured in the data to reduce confounding by unmeasured factors.

When comparing results from an RCT to a database study that emulates the design, we assume that the findings from the single RCT are internally valid.

Although we plan to emulate the important features of each trial as closely as possible in healthcare claims, there may be some elements of the RCT design that are not emulable with a database study, which means that the real-world evidence obtained from the database study and trial will address slightly different clinical questions. For example, in routine clinical care, adherence to treatment is typically not as high as it is in an RCT with strong measures in place to encourage adherence to the study protocol. This means that there is more discontinuation and short-term medication use in the patients identified in claims databases than trial participants.

Apparent agreement between RCT and database study results could occur if the effects of multiple factors (chance, emulation differences, bias) cancel each other out.

## 8. Protection of human subjects

This study has been approved by the Brigham and Women's Hospital Institutional Review Board.

### 9. References

- 1. Nicholls SJ, Bhatt DL, Buse JB, et al. Comparison of tirzepatide and dulaglutide on major adverse cardiovascular events in participants with type 2 diabetes and atherosclerotic cardiovascular disease: SURPASS-CVOT design and baseline characteristics. *Am Heart J*. 2024;267:1-11. doi:10.1016/j.ahj.2023.09.007
- 2. Gemeinsame Stellungnahme zur Nutzenbewertung gemäß § 35a SGB V von Tirzepatid (Dia- betes mellitus Typ 2). https://www.ddg.info/fileadmin/user\_upload/06\_Gesundheitspolitik/01\_Stellungnahmen/2024/Gemeinsame\_Stellungnahme\_zur\_Nutzenbewertung\_Tirzepatid\_fnl\_2 00103.pdf
- 3. FDA approves Lilly's Mounjaro<sup>™</sup> (tirzepatide) injection, the first and only GIP and GLP-1 receptor agonist for the treatment of adults with type 2 diabetes | Eli Lilly and Company. Accessed July 18, 2025. https://investor.lilly.com/news-releases/news-release-details/fda-approves-lillys-mounjarotm-tirzepatide-injection-first-and
- 4. FDA Approves Trulicity™ (dulaglutide), Lilly's Once-Weekly Therapy for Adults with Type 2 Diabetes | Eli Lilly and Company. Accessed July 23, 2025. https://investor.lilly.com/news-releases/news-release-details/fda-approves-trulicitytm-dulaglutide-lillys-once-weekly-therapy
- 5. Trulicity® (dulaglutide) is the first and only type 2 diabetes medicine approved to reduce cardiovascular events in adults with and without established cardiovascular disease | Eli Lilly and Company. Accessed July 23, 2025. https://investor.lilly.com/news-releases/news-release-details/trulicityr-dulaglutide-first-and-only-type-2-diabetes-medicine
- 6. FDA approves additional doses of Trulicity® (dulaglutide) for the treatment of type 2 diabetes | Eli Lilly and Company. Accessed July 23, 2025. https://investor.lilly.com/news-releases/news-release-details/fda-approves-additional-doses-trulicityr-dulaglutide-treatment
- 7. Schneeweiss S. A basic study design for expedited safety signal evaluation based on electronic healthcare data. *Pharmacoepidemiol Drug Saf.* 2010;19(8):858-868. doi:10.1002/pds.1926
- 8. Ray WA. Evaluating medication effects outside of clinical trials: new-user designs. Am J Epidemiol. 2003;158(9):915-920. doi:10.1093/aje/kwg231
- 9. Kiyota Y, Schneeweiss S, Glynn RJ, Cannuscio CC, Avorn J, Solomon DH. Accuracy of medicare claims-based diagnosis of acute myocardial infarction: estimating positive predictive value on the basis of review of hospital records. *Am Heart J*. 2004;148(1):99-104. doi:10.1016/j.ahj.2004.02.013
- 10. Andrade SE, Harrold LR, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. *Pharmacoepidemiol Drug Saf.* 2012;21 Suppl 1(Suppl 1):100-128. doi:10.1002/pds.2312
- 11. Roumie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. *Pharmacoepidemiol Drug Saf.* 2008;17(1):20-26. doi:10.1002/pds.1518
- 12. Wahl PM, Rodgers K, Schneeweiss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious adverse events in a commercially-insured population. *Pharmacoepidemiol Drug Saf*. 2010;19(6):596-603. doi:10.1002/pds.1924
- 13. Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. *J Clin Epidemiol*. 2011;64(7):749-759. doi:10.1016/j.jclinepi.2010.10.004
- 14. Sun JW, Rogers JR, Her Q, et al. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. *Med Care*. 2017;55(12):1046-1051.

#### doi:10.1097/MLR.0000000000000824

- 15. Kim DH, Schneeweiss S, Glynn RJ, Lipsitz LA, Rockwood K, Avorn J. Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index. *J Gerontol A Biol Sci Med Sci*. 2018;73(7):980-987. doi:10.1093/gerona/glx229
- 16. Wang SV, Schneeweiss S, RCT-DUPLICATE Initiative, et al. Emulation of Randomized Clinical Trials With Nonrandomized Database Analyses: Results of 32 Clinical Trials. *JAMA*. 2023;329(16):1376-1385. doi:10.1001/jama.2023.4221
- 17. Franklin JM, Pawar A, Martin D, et al. Nonrandomized Real-World Evidence to Support Regulatory Decision Making: Process for a Randomized Trial Replication Project. *Clin Pharmacol Ther*. 2020;107(4):817-826. doi:10.1002/cpt.1633
- 18. Olubowale OT, Safford MM, Brown TM, et al. Comparison of Expert Adjudicated Coronary Heart Disease and Cardiovascular Disease Mortality With the National Death Index: Results From the REasons for Geographic And Racial Differences in Stroke (REGARDS) Study. *J Am Heart Assoc*. 2017;6(5):e004966. doi:10.1161/JAHA.116.004966

# 10. Appendices

See accompanying excel files that specify the cohort study.

#### 1 Target Trial Framework, Operational Definitions, and Data Fitness Assessment

### 2 Code algorithms

- 2a Exposure
- 2a Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- **8 Covariate Algorithm Sources**

## **Appendices**

- 1 Target Trial Framework, Operational Definitions and Data Fitness Assessment
- 2 Code algorithms
- 2a Exposure
- 2b Inclusion
- 2c Exclusion
- 2d Outcome
- 3 Flowchart for cohort assembly
- 4 1st feasibility assessment
- 5 2nd feasibility assessment
- 6 Balance Assessment PS Distribution and C-Statistic
- 7 Balance Assessment Table 1
- 8 Covariate Algorithm Sources

| | SURPASS-CVOT | OPTUM | MARKETSCAN | Notes/Questions | Color coding |
|---|---|---|---|---|---|
| Treatment assignment (time 0, index date) | International, double-blind, randomized, active-controlled trial to treatment A vs B | Non-randomized initiation of treatment Tirzepatide vs Dulaglutide (first eligible entry to study population) | Non-randomized initiation of treatment Tirzepatide vs Dulaglutide (first eligible entry to study population) | | Good proxy definition |
| , | | Code type: RX | Code type: RX | | , |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A | | |
| | | Washout window: [-183,-1] | Washout window: [-183,-1] | | |
| | | Incident with respect to: Tirzepatide in any formulation or dose Assessment window: N/A | Incident with respect to: Tirzepatide in any formulation or dose Assessment window: N/A | | |
| | Tirzepatide (subcutaneously once per week) | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | Moderate proxy definition |
| Exposure | once per week) | Code type: RX | Code type: RX | | Moderate proxy definition |
| | | Care setting: N/A Diagnosis position: N/A | Care setting: N/A Diagnosis position: N/A | | |
| | | Washout window: [-183,-1] Incident with respect to: Dulagiutide in any formulation or dose | Washout window: [-183, -1] Incident with respect to: Dulaglutide in any formulation or dose | | |
| | | Assessment window: N/A | Assessment window: N/A | | |
| Compositor | Dulaglutide (subcutaneously once per week) | Source of algorithm: N/A Measurement characteristics: N/A | Source of algorithm: N/A Measurement characteristics: N/A | | Poorly measured in database |
| Comparator | bulagrande (subcatalleously office per week) | Code type: DX,PX | Code type: DX,PX | | 1 oony measured matabase |
| | | Care setting: Inpatient for stroke/MI, any for death Diagnosis position: Primary for Stroke, Any for MI | Care setting: Inpatient for stroke/MI, any for death Diagnosis position: Primary | | |
| | | Washout window: | Washout window: | | |
| | | Source of algorithm: Measurement characteristics: Death includes information from the inpatient discharged dead status, social security death master file, and deaths scraped from | Source of algorithm: Measurement characteristics: Death includes information from the inpatient discharged dead status, social security death master file, and deaths scraped from | | Poorly measured in database and |
| Primary outcome to be emulated | MACE, defined as CV death, MI, or stroke | obituaries or other sources. Code type: DX, PX | obituaries or other sources. Code type: DX, PX | | important |
| | | Care setting: Inpatient for stroke/MI, any for death | Care setting: Inpatient for stroke/MI, any for death | | |
| | | Diagnosis position: Primary for Stroke, Any for MI Washout window: | Diagnosis position: Primary for Stroke, Any for MI Washout window: | | |
| | | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) Measurement characteristics: Death includes information from the inpatient discharged | Source of algorithm: PROMISE Team, Validation studies, (Investigator reviewed codes) Measurement characteristics: Death includes information from the inpatient discharged | | |
| | | dead status, social security death master file, and deaths scraped from obituaries or other | dead status, social security death master file, and deaths scraped from obituaries or other | | |
| | | sources. PPV for ischemic stroke using ICD9 codes was 88% and 95% | sources. PPV for ischemic stroke using ICD9 codes was 88% and 95% | | |
| | - Time to first occurrence of individual components of primary composite | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | [https://pubmed.ncbi.nlm.nih.gov/12364739/ and | | |
| Secondary outcome to be | outcome Hernia (negative control) | https://pubmed.ncbi.nlm.nih.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was | https://pubmed.ncbi.nlm.nih.gov/20140892/] Both of the above ICD9 codes were mapped to ICD10, but no validation study was | | |
| emulated | - Lumbar radiculopathy (negative control) Randomization date | performed. One day after initiation of treatment with tirzepatide or dulaglutide | performed. One day after initiation of treatment with tirzepatide or dulaglutide | | |
| i ollow up start | Nandomizadonidate | Earliest of: Outcome, end of observation in data, end of study period (365 days), | Earliest of: Outcome, end of observation in data, end of study period (365 days), | | |
| Follow up end | Expected mean follow-up: 4 years | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-<br>1-RA. nursing home admission | discontinuation of study drug (45 days grace window and risk-window), switch to other GLP-<br>1-RA, nursing home admission | | |
| | *************************************** | , | , | Algorithm detail: Adherence in clinical practice databases is expected to be much worse than in the trial, therefore the on- | |
| | | | | treatment analysis at 1 year follow-up will be the primary | |
| | Intention-to-treat effect Cox proportional hazards model | On-treatment effect Cox proportional hazards regression model | On-treatment effect Cox proportional hazards regression model | analysis. | |
| Inclusion criteria | | oox proportional nazardo regression model | OOX Proportional nazardo regression model | | |
| | | Applied before/after selection of index date: Before Assessment window: [0, 0] | Applied before/after selection of index date: Before Assessment window: [0, 0] | | |
| | | Assessment window: [0,0] Code type: N/A | Assessment window: [0, 0] Code type: N/A | | |
| | | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A | | |
| | | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A | | |
| | Men and women aged 40 years or older | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before | | |
| | | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX | Assessment window: [0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX | | |
| | | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any | | |
| 1 | Men and women aged 40 years or older | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | | |
| 1 | | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | | |
| 1 | Men and women aged 40 years or older | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-20, 0] | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [20, 0] | Algorithm detail: Not considered in the main cohort due to high missingness of HhAIr measurements. A sensitivity | |
| 1 | Men and women aged 40 years or older | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any | high missingness of HbA1c measurements. A sensitivity<br>analyses on a subset of the cohort with HbA1c | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: 365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: 120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement indow: 120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | Assessment window: [0, 0] Code type: NA Care setting: NA Diagnosis position: N/A Source of algorithm: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement indow: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team | high missingness of HbA1c measurements. A sensitivity | |
| 2 | Men and women aged 40 years or older | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Mapplied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Measurement characteristics: N/A Source of algorithm: PROMISE team Measurement characteristics: N/A Measurement characteristics: N/A Measurement characteristics: N/A | high missingness of HbA1c measurements. A sensitivity<br>analyses on a subset of the cohort with HbA1c<br>measurements will be conducted in the cohort from the | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] | high missingness of HbA1c measurements. A sensitivity analyses on a subset of the cohort with HbA1c measurements will be conducted in the cohort from the Optum database, including the last recorded value in the | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-365, 0] Code type: D/X Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/X Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-365, 0] Code type: D/X Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/X Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | high missingness of HbA1c measurements. A sensitivity analyses on a subset of the cohort with HbA1c measurements will be conducted in the cohort from the Optum database, including the last recorded value in the | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window:[0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before of algorithm: PROMISE team Measurement characteristics: N/A Applied before of algorithm: Any Source of algorithm: Any Source of algorithm: Any Code type: DX Code type: DX. LOINC (7-20,0) Code type: DX. LOINC (7-20,0) Code type: DX. LOINC (7-20,0) Code type: DX. LOINC (7-20,0) Diagnosis position: Any Diagnosis position: Any Code type: DX. LOINC (7-20,0) Diagnosis position: Any | Assessment window.[0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window.[-365,0] Code type: D/A Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window.[-20.0] Code type: D/A Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: D/A Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: D/A, LOINC Care setting: Any Diagnosis position: Any | high missingness of HbA1c measurements. A sensitivity analyses on a subset of the cohort with HbA1c measurements will be conducted in the cohort from the Optum database, including the last recorded value in the | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-365, 0] Code type: D/A Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-20, 0] Code type: D/A Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/A, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: D/A Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/A, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidiation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. | |
| 2 | Men and women aged 40 years or older Type 2 diabetes mellitus | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Pallidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMIH: related (ICD-9-CM and ICD-10-CM administrative, diagnosis position: Any Source of algorithm: Validation of body mass index (BMIH: related (ICD-9-CM and ICD-10-CM administrative, diagnosis codes recorded in US claims data | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Cade type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMII): related (ICD-9-CM and ICD-10-CM administrative, diagnosis position: Any Source of algorithm: Validation of body mass index (BMII): related (ICD-9-CM and ICD-10-CM administrative, diagnosis code recorded in US claims data | high missingness of HbA1c measurements. A sensitivity analyses on a subset of the cohort with HbA1c measurements will be conducted in the cohort from the Optum database, including the last recorded value in the | |
| 1<br>2<br>3<br>4<br>5 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m² Established atherosclerotic cardiovascular disease, either one of: | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-365, 0] Code type: D/A Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-20, 0] Code type: D/A Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/A, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: D/A Care setting: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: D/A Care setting: Any Diagnosis position: Any Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/A, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidiation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 1<br>2<br>3<br>4<br>5 | Men and women aged 40 years or older $Type\ 2\ diabetes\ mellitus$ $HbA1c\ \geq 7\%\ and\ \leq 10.5\%$ $BMI\ \geq 25kg/m2$ | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-365, 0] Code type: D/ Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-120, 0] Code type: D/ Code type: D/ Code type: D/ Code type: D/ Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Code type: D/ Code type: D/ Code type: D/ Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Pallation of beeity-related diagnosis codes inclaims data: Validation of body mass index (RMM:-related ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A | Assessment window. [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-365, 0] Code type: D/ Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window. [-120, 0] Code type: D/ Code type: D/ Code type: D/ Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Care setting: Any Diagnosis position: Any Diagnosis position: Any Code type: D/ Code type: D/ Code type: D/ Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: D/, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Pallidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMM:-related (CD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 1<br>2<br>3 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m² Established atherosclerotic cardiovascular disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-30,0] Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-30,0] Signalia on the poly mass index (BMI): related diagnosis codes inclaims data: Validation of body mass index (BMI): related (ICD-9-CM and ICD-10-CM administrative, diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] | Assessment window:[0,0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: DX Care setting: Any Diagnosis position: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-120,0] Code type: DX Care setting: Any Source of algorithm: Any Source of algor | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 1<br>2<br>3 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m² Established atherosclerotic cardiovascular disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-20,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before after selection of index date: Before Asplied before after selection of index date: Before Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before after selection of index date: Before Asplied before after selection of index date: Before Asplied before after selection of index date: Before Asplied before after selection of index date: Before Asplied before after selection of index date: Before Asplied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before after selection of index date: Before Assessment window: [-30,0] Code type: DX. CONC Code t | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 1<br>2<br>3 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m² Established atherosclerotic cardiovascular disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of obesity-related diagnosis codes in claims data: Validation of body mass index (BMII): related (ICD-9-CM and ICD-10-CM administrative diagnosis code recorded in ICD claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX. Care setting: Any Diagnosis position: Any | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of obesity-related diagnosis codes in claims data: Validation of body mass index (BMII): related (ICD-9-CM and ICD-10-CM administrative diagnosis code recorded in ICS claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX. Care setting: Any Diagnosis position: Any | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 2<br>3<br>4<br>5<br>5.1 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m² Established atherosclerotic cardiovascular disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX. Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of obesity-related diagnosis codes in claims data: Validation of body mass index (BMI): related (ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX. Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 2<br>3<br>4<br>5<br>5.1 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m2 Established atherosclerotic cardiovascular disease, either one of: Coronary artery disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX Care setting: Any Diagnosis position: Any Diag | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Diagnosis position: Any Applied before/after selection of index date: Before Assessment window: [-130, 0] Code type: DX, LOINC Care setting: Any Diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-130, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: If BMI measurement via LOINC code is | |
| 2<br>3<br>4<br>5<br>5.1 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m2 Established atherosclerotic cardiovascular disease, either one of: Coronary artery disease, either one of: | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Care setting: Any Diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-130,0] Code type: DX Code typ | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis codes in claims data: Walidation of hosty mass index (JBMI)-related (J0-9-CM and ICD-10-CM administrative, diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Code type: DX | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. Algorithm detail: If BMI measurement via LOINC code is below 10 or above 100 then measurent is set to missing. | |
| 2<br>3<br>4<br>5<br>5.1 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m2 Established atherosclerotic cardiovascular disease, either one of: Coronary artery disease, either one of: | Assessment window: [0, 0] Code type: N/A Car esetting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-130,0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Measurement characteri | Assessment window: [0, 0] Code type: N/A Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730,0] Code type: DX, LOINC Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Validation of besity-related diagnosis codes in claims data: Validation of body mass index: MBMI-related ICD-9-CM and ICD-10-CM administrative. diagnosis recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, DAY Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Me | high missingness of Hb AL measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propersity score. Algorithm detail: HBMI measurement via LOINC code is below 10 or above 100 then measurent is set to missing. Algorithm detail: ±50% stenosis was proxied by ICD-10 codes, based on the premise that most patients are coded | |
| 1<br>2<br>3<br>4<br>5.1<br>5.1 | Men and women aged 40 years or older Type 2 diabetes mellitus HbA1c ≥7% and ≤ 10.5% BMI ≥ 25kg/m2 Established atherosclerotic cardiovascular disease, either one of: Coronary artery disease, either one of: | Assessment window: [0, 0] Code type: N/A Car esetting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of besity-related diagnosis codes in claims data: Validation of body mass index (BMI)-related (ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | Assessment window: [0, 0] Code type: N/A Car esetting: N/A Diagnosis position: N/A Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-120, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-730, 0] Code type: DX, LOINC Care setting: Any Diagnosis position: Any Source of algorithm: Palidation of obesity-related diagnosis codes in claims data: Validation of body mass index (BMI): related (ICD-9-CM and ICD-10-CM administrative diagnosis codes recorded in US claims data Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any | high missingness of Hb ALC measurements. A sensitivity analyses on a subset of the cohort with Hb ALC measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. Algorithm detail: If BMI measurement via LOINC code is below 10 or above 100 then measurent is set to missing. | |

| 5.1.3 ≥50% stenosis in 2 or more major coronary arteries | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: N/A Source of algorithm: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Any Diagnosis position: N/A Source of algorithm: N/A Source of algorithm: N/A | See 5.1.2 |
|---|---|---|---|
| 5.1.4 History of surgical or percutaneous coronary revascularization procedure 5.2 Cerebrovascular disease, either one of: | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| 5.2.1 Documented history of ischemic stroke | Assessment window: [all available data, 0] Codet type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Assessment window: [all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | |
| Carotid arterial disease with ≥50% stenosis, documented by carotid ultrasound, | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of alsorthm: N/A | |
| 5.2.2 MRI, or angiography | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Anny Diagnosis position: Anny Source of algorithm: N/A | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX, PX Care setting: Anny Diagnosis position: Any Source of algorithm: N/A | See 5.1.2 |
| 5.2.3 History of carotid stenting or surgical revascularization 5.3 Peripheral arterial disease, either one of: | Measurement characteristics: N/A Applied before/after selection of index date: Before | Measurement characteristics: N/A Applied before/after selection of index date: Before | |
| 5.3.1 Intermittent claudication and ankle-brachial index < 0.9 | Assessment window.[-all available data, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window.[all available data, 0] Code type: D/X, P/X Care setting: Any | Assessment window.[-all available data, 0] Code type: DX Car esetting: Any Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window.[all available data, 0] Code type: DX, PX Car esetting: Any | Algorithm detail: Intermittent claudication was proxied by ICD-10-CM codes for peripheral vascular disease. |
| Prior nontraumatic amputation or peripheral vascular procedure (eg., stenting or 5.3.2 surgical revascularization), due to peripheral arterial ischemia | Diagnosis position: Any Source of algorithm: N/A Measurement characteristics: N/A | Diagnosis position: Any<br>Source of algorithm: N/A<br>Measurement characteristics: N/A | |
| Exclusion criteria 6 HbA1c>10.5% | Applied before/after selection of index date: Before Assessment window:[-120,0] X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: PX Care setting: Any | Applied before/after selection of index date: Before Assessment window:[-120,0] X X Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window:[-365,0] Code type: PX Care setting: Any | Algorithm detail: Not considered in the main cohort due to high missingness of HbALc measurements. A sensitivity analyses on a subset of the cohort with HbALc measurements will be conducted in the cohort from the Optum database, including the last recorded value in the propensity score. |
| 7 Planning treatment for diabetic retinopathy and/or macular edema | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A Applied before/after selection of index date: Before | Algorithm detail: Planned treatment will be proxied by a<br>history of treatment (e.g. codes for intravitreal injection of<br>anti-VEGFi OR photocoagulation.) |
| 8 Hospitalized for chronic heart failure within 2 months prior to screening | Assessment window:[-60,0] for HF diagnosis or HHF Code type: DX, RX Care setting: [inpatient Diagnosis position: Primary Source of algorithm: DUPLICATE team, investigator reviewed codes Measurement characteristics: N/A | Assessment window:[-60,0] for HF diagnosis or HHF Code type: DX, RX Care setting: [inpatient Diagnosis position: Primary Source of algorithm: DIPLICATE team, investigator reviewed codes Measurement characteristics: NIA | |
| Chronic New York Heart Association Functional Classification IV heart failure | Can't be measured in claims. | Can't be measured in claims. | Algorithm detail: A proportion of patients with NYHA class IV will be excluded from the cohort by exclusion criterion 8. |
| 10 Planned coronary, carottid, or peripheral artery revascularization 11 History of chronic or acute pancreatitis | Can't be measured inclaims. Applied before/after selection of index date: Before Assessment window: [-183,0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/after selection of index date: Before | Can't be measured in claims. Applied before/lafte selection of index date: Before Assessment window: [-183, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: NIA Applied before/lafter selection of index date: Before | Will be excluded not the color by exclusion circles on b. |
| 12 Known clinically significant gastric emptying abnormality or bariatric surgery | Assessment window:[-365,0] Codet type: DV, Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team, https://pubmed.ncbi.nlm.nih.gov/35857336/, Investigator reviewed codes Measurement characteristics: N/A | Assessment window: [-365,0] Code type: Dy, Care setting: Inpatient Diagnosis position: Any Source of algorithm: PROMISE team, https://pubmed.ncbi.nlm.nin.gov/35857/336/, Investigator reviewed codes Measurement characteristics: N/A | See SUMMIT |

| Liver disease (not including non-alcoholic fatty liver disease [NAFLD]) or ALT level 13 23 X the ULN | Applied before/after selection of index date: Before Assessment window: [183,0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Investigator reviewed codes Measurement characteristics: N/A | Applied before/after selection of Index date: Before Assessment window: [183, 0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: Investigator reviewed codes Measurement characteristics: N/A | Algorithm detail: Based on diagnostic codes rather than laboratory values. |
|---|---|---|---|
| 14 eGFR <15 mL/Min/1/73 m2 or on chronic dialysis | Applied before/after selection of index date: Before Assessment window: [-365.0] Code type DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of Index date: Before Assessment window: [-365,0] Code type: DX, PX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Algorithm detail: Proxied by ICD-10-CM codes for chronic kidney disease stage 5 OR end-stage renal disease OR ICD-10-CM procedure codes for dishysis. |
| Family or personal history of multiple endocrine neoplasia or medullary thyroid 15 carcinoma | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: PROMISE team Measurement characteristics: N/A | Applied before/after selection of index date: Before Assessment window: [all available data, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithms: POMISE team Measurement characteristics: N/A | |
| 16 Elevated serum calcitonin level | Cart be measured in claims. Applied before'after selection of index date: Before Assessment window: [-60, 0] for all except unstable angina [-30, 0] Code type; DX, PX Care setting: inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviewed codes | Can't be measured in claims. Applied befor-lafter selection of index date: Before Assessment window: [-60,0] for all except unstable angina [-30,0] Code type: DX, PX: Care setting: inpatient/ED for MI, Stroke, TIA, inpatient for procedures Diagnosis position: Any Source of algorithm: PROMISE team, Investigator reviewed codes | |
| 17 Cardiovascular event or intervention <60 days prior to screening | Measurement characteristics: N/A Applied before/after selection of index date: Before Assessment window: [-183,0] Code type: RX Care setting: N/A Diagnosis position: N/A Source of algorithm: N/A | Measurement characteristics: NIA Applied before/after selection of index date: Before Assessment window: [-183,0] Code type: RX Care setting: NIA Diagnosis position: NIA Source of algorithm: NIA | |
| 18 GLP-1-RA or pramlintide treatment within 3 months prior to Visit 1 19 Women who are pregnant or breastfeeding | Measurement characteristics: n/a Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: DX Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Measurement characteristics: n/a Applied before/after selection of index date: Before Assessment window: [-365, 0] Code type: D/X Care setting: Any Diagnosis position: Any Source of algorithm: Pregnancy team Measurement characteristics: N/A | Algorithm detail: Proxied by ICD-10-CM codes indicative of pregnancy at baseline. |


TYPE 2 DIABETES MELLITUS WITH SEVERE NONPROLIFERATIVE DIABETIC RETINOPATHY


5.1.1 5.1.1 5.1.1 5.1.1 5.1.1 5.1.1


BYPASS CORONARY ARTERY, ONE ARTERY FROM AORTA WITH ZOOPLASTIC TISSUE,


BYPASS CORONARY ARTERY, ONE ARTERY FROM CORONARY ARTERY, PERCUTANEOUS


BYPASS CORONARY ARTERY, TWO ARTERIES FROM THORACIC ARTERY WITH


BYPASS CORONARY ARTERY, THREE ARTERIES FROM ABDOMINAL ARTERY WITH

BYPASS CORONARY ARTERY, FOUR OR MORE ARTERIES FROM AORTA WITH


BYPASS CORONARY ARTERY, FOUR OR MORE ARTERIES FROM CORONARY VEIN WITH


BYPASS CORONARY ARTERY, FOUR OR MORE ARTERIES FROM LEFT INTERNAL


DILATION OF CORONARY ARTERY, TWO ARTERIES WITH THREE DRUG-ELUTING


DILATION OF CORONARY ARTERY, TWO ARTERIES WITH RADIOACTIVE INTRALUMINAL


DILATION OF CORONARY ARTERY, THREE ARTERIES, BIFURCATION, WITH TWO


DILATION OF CORONARY ARTERY, FOUR OR MORE ARTERIES, BIFURCATION, WITH TWO


| 5.1.4 | History of surgical or percutaneous coronary | 33519 PX | CORONARY ARTERY BYPASS, USING VENOUS GRAFT(S) AND ARTERIAL GRAFT(S); 3 VENOUS GRAFTS (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) | CPT/HCPCS |
|---|---|---|---|---|
| 5.1.4 | History of surgical or percutaneous coronary | 33521 PX | CORONARY ARTERY BYPASS, USING VENOUS GRAFT(S) AND ARTERIAL GRAFT(S); 4 VENOUS GRAFTS (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33522 PX | CORONARY ARTERY BYPASS, USING VENOUS GRAFT(S) AND ARTERIAL GRAFT(S); 5<br>VENOUS GRAFTS (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE)<br>CORONARY ARTERY BYPASS, USING VENOUS GRAFT(S) AND ARTERIAL GRAFT(S); 6 OR | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33523 PX | MORE VENOUS GRAFTS (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) REOPERATION, CORONARY ARTERY BYPASS PROCEDURE OR VALVE PROCEDURE, MORE THAN 1 MONTH AFTER ORIGINAL OPERATION (LIST SEPARATELY IN ADDITION TO CODE | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33530 PX | FOR PRIMARY PROCEDURE) | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33533 PX | CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); SINGLE ARTERIAL GRAFT CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 2 CORONARY ARTERIAL | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33534 PX | GRAFTS CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 3 CORONARY ARTERIAL | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33535 PX | GRAFTS<br>CORONARY ARTERY BYPASS, USING ARTERIAL GRAFT(S); 4 OR MORE CORONARY | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33536 PX | ARTERIAL GRAFTS REPAIR OF POSTINFARCTION VENTRICULAR SEPTAL DEFECT, WITH OR WITHOUT | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33545 PX | MYOCARDIAL RESECTION CORONARY ENDARTERECTOMY, OPEN, ANY METHOD, OF LEFT ANTERIOR DESCENDING, CIRCUMFLEX, OR RIGHT CORONARY ARTERY PERFORMED IN CONJUNCTION WITH | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 33572 PX | CORONARY ARTERY BYPASS GRAFT PROCEDURE, EACH VESSEL (LIST SEPARATELY IN ADDITION TO PRIMARY PROCEDURE) | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92920 PX | PERCUTANEOUS TRANSLUMINAL CORONARY ANGIOPLASTY; SINGLE MAJOR CORONARY ARTERY OR BRANCH PERCUTANEOUS TRANSLUMINAL CORONARY ANGIOPLASTY; EACH ADDITIONAL | CPT/HCPCS |
| | | | BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR | |
| 5.1.4 | History of surgical or percutaneous coronary | 92921 PX | PRIMARY PROCEDURE) PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH CORONARY | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92924 PX | ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR CORONARY ARTERY OR BRANCH | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92925 PX | PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) PERCUTANEOUS TRANSCATHETER PLACEMENT OF INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR CORONARY ARTERY OR | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92928 PX | BRANCH PERCUTANEOUS TRANSCATHETER PLACEMENT OF INTRACORONARY STENT(S), WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92929 PX | PROCEDURE) PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; SINGLE MAJOR CORONARY | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92933 PX | ARTERY OR BRANCH PERCUTANEOUS TRANSLUMINAL CORONARY ATHERECTOMY, WITH INTRACORONARY STENT, WITH CORONARY ANGIOPLASTY WHEN PERFORMED; EACH ADDITIONAL BRANCH OF A MAJOR CORONARY ARTERY (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY | |
| 5.1.4 | History of surgical or percutaneous coronary | 92934 PX | PROCEDURE) PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF OR THROUGH CORONARY ARTERY BYPASS GRAFT (INTERNAL MAMMARY, FREE ARTERIAL, VENOUS), ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY. | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92937 PX | INCLUDING DISTAL PROTECTION WHEN PERFORMED; SINGLE VESSEL PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF OR THROUGH CORONARY ARTERY BYPASS GRAFT (INTERNAL MAMMARY, FREE ARTERIAL, VENOUS), ANY COMBINATION OF INTRACORONARY STENT, ATHERECTOMY AND ANGIOPLASTY, INCLUDING DISTAL PROTECTION WHEN PERFORMED; EACH ADDITIONAL BRANCH | CPT/HCPCS |
| 5.1.4 | History of surgical or percutaneous coronary | 92938 PX | SUBTENDED BY THE BYPASS GRAFT (LIST SEPARATELY IN ADDITION TO CODE FOR PRIMARY PROCEDURE) | CPT/HCPCS |


PERCUTANEOUS TRANSLUMINAL REVASCULARIZATION OF ACUTE TOTAL/SUBTOTAL


DILATION OF RIGHT COMMON CAROTID ARTERY WITH DRUG-ELUTING INTRALUMINAL


DILATION OF RIGHT COMMON CAROTID ARTERY WITH FOUR OR MORE INTRALUMINAL


DILATION OF LEFT COMMON CAROTID ARTERY WITH TWO DRUG-ELUTING


DILATION OF RIGHT INTERNAL CAROTID ARTERY, BIFURCATION, WITH INTRALUMINAL


DILATION OF LEFT INTERNAL CAROTID ARTERY WITH INTRALUMINAL DEVICE, OPEN


DILATION OF LEFT INTERNAL CAROTID ARTERY, BIFURCATION, WITH TWO


ATHEROSCLEROSIS OF NATIVE ARTERIES OF RIGHT LEG WITH ULCERATION OF OTHER


ATHEROSCLEROSIS OF UNSPECIFIED TYPE OF BYPASS GRAFT(S) OF THE RIGHT LEG WITH


ATHEROSCLEROSIS OF OTHER TYPE OF BYPASS GRAFT(S) OF THE RIGHT LEG WITH


BYPASS ABDOMINAL AORTA TO BILATERAL INTERNAL ILIAC ARTERIES WITH


BYPASS ABDOMINAL AORTA TO LEFT INTERNAL ILIAC ARTERY WITH AUTOLOGOUS


BYPASS ABDOMINAL AORTA TO BILATERAL EXTERNAL ILIAC ARTERIES WITH

BYPASS ABDOMINAL AORTA TO LOWER EXTREMITY ARTERY, PERCUTANEOUS


BYPASS LEFT COMMON ILIAC ARTERY TO RIGHT FEMORAL ARTERY WITH AUTOLOGOUS


BYPASS RIGHT INTERNAL ILIAC ARTERY TO BILATERAL FEMORAL ARTERIES WITH


BYPASS LEFT INTERNAL ILIAC ARTERY TO LEFT FEMORAL ARTERY WITH AUTOLOGOUS


BYPASS RIGHT EXTERNAL ILIAC ARTERY TO RIGHT FEMORAL ARTERY WITH SYNTHETIC


BYPASS LEFT EXTERNAL ILIAC ARTERY TO BILATERAL FEMORAL ARTERIES WITH


BYPASS LEFT FEMORAL ARTERY TO BILATERAL FEMORAL ARTERIES WITH SYNTHETIC


BYPASS LEFT FEMORAL ARTERY TO BILATERAL FEMORAL ARTERIES WITH


BYPASS RIGHT POPLITEAL ARTERY TO FOOT ARTERY WITH AUTOLOGOUS ARTERIAL


BYPASS LEFT POPLITEAL ARTERY TO LOWER EXTREMITY VEIN WITH SYNTHETIC


BYPASS LEFT POPLITEAL ARTERY TO LOWER EXTREMITY ARTERY, PERCUTANEOUS


DILATION OF ABDOMINAL AORTA WITH THREE INTRALUMINAL DEVICES,


DILATION OF RIGHT COMMON ILIAC ARTERY, BIFURCATION, WITH TWO INTRALUMINAL


DILATION OF RIGHT COMMON ILIAC ARTERY WITH FOUR OR MORE DRUG-ELUTING


DILATION OF LEFT COMMONILIAC ARTERY, BIFURCATION, WITH THREE DRUG-ELUTING


DILATION OF RIGHT INTERNAL ILIAC ARTERY WITH FOUR OR MORE INTRALUMINAL


DILATION OF LEFT INTERNAL ILIAC ARTERY WITH TWO INTRALUMINAL DEVICES, OPEN


DILATION OF LEFT INTERNAL ILIAC ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE,


DILATION OF LEFT EXTERNAL ILIAC ARTERY WITH DRUG-ELUTING INTRALUMINAL


DILATION OF RIGHT FEMORAL ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL


DILATION OF LEFT FEMORAL ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-


DILATION OF RIGHT POPLITEAL ARTERY USING DRUG-COATED BALLOON, OPEN


DILATION OF RIGHT POPLITEAL ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE,


DILATION OF LEFT POPLITEAL ARTERY, BIFURCATION, WITH DRUG-ELUTING


DILATION OF LEFT POPLITEAL ARTERY WITH TWO INTRALUMINAL DEVICES,


DILATION OF RIGHT ANTERIOR TIBIAL ARTERY WITH FOUR OR MORE DRUG-ELUTING


DILATION OF LEFT ANTERIOR TIBIAL ARTERY, BIFURCATION, WITH DRUG-ELUTING


DILATION OF RIGHT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH FOUR OR MORE


DILATION OF RIGHT POSTERIOR TIBIAL ARTERY WITH TWO INTRALUMINAL DEVICES,


DILATION OF LEFT POSTERIOR TIBIAL ARTERY, BIFURCATION, WITH INTRALUMINAL


DILATION OF RIGHT PERONEAL ARTERY, BIFURCATION, WITH TWO DRUG-ELUTING


DILATION OF LEFT PERONEAL ARTERY, BIFURCATION, WITH FOUR OR MORE


DILATION OF LEFT FOOT ARTERY, BIFURCATION, WITH TWO INTRALUMINAL DEVICES,


DILATION OF LEFT FOOT ARTERY, BIFURCATION, WITH INTRALUMINAL DEVICE,


DILATION OF LOWER ARTERY, BIFURCATION, WITH FOUR OR MORE DRUG-ELUTING


EXTIRPATION OF MATTER FROM RIGHT FEMORAL ARTERY, BIFURCATION,


EXTIRPATION OF MATTER FROM LOWER ARTERY, BIFURCATION, PERCUTANEOUS


BYPASS GRAFT, WITH VEIN; TIBIAL-TIBIAL, PERONEAL-TIBIAL, OR TIBIAL/PERONEAL


REVASCULARIZATION, ENDOVASCULAR, OPEN OR PERCUTANEOUS, FEMORAL,


| Cardiovascular event or intervention < 60 days prior to 17 screening 03120J6 PX BYPASS INNOMINATE ARTERY TO RIGHT UPPER LEG ARTERY WITH SYNTHETICS | SUBSTITU ICD-10-PCS |
|---|---|
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120J7 PX BYPASS INNOMINATE ARTERY TO LEFT UPPER LEG ARTERY WITH SYNTHETIC SI | JBSTITUT ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120J8 PX BYPASS INNOMINATE ARTERY TO BILATERAL UPPER LEG ARTERY WITH SYNTH | ETIC SUBSICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 03120J9 PX BYPASS INNOMINATE ARTERY TO RIGHT LOWER LEG ARTERY WITH SYNTHETIC | |
| Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 03120JB PX BYPASS INNOMINATE ARTERY TO LEFT LOWER LEG ARTERY WITH SYNTHETIC S<br>Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 03120JC PX BYPASS INNOMINATE ARTERY TO BILATERAL LOWER LEG ARTERY WITH SYNTH Cardiovascular event or intervention <60 days prior to | ETIC SUB!ICD-10-PCS |
| 17 screening 03120JD PX BYPASS INNOMINATE ARTERY TO UPPER ARM VEIN WITH SYNTHETIC SUBSTITUTION Cardiovascular event or intervention <60 days prior to | TE, OPEN, ICD-10-PCS |
| 17 screening 03120JF PX BYPASS INNOMINATE ARTERY TO LOWER ARM VEIN WITH SYNTHETIC SUBSTITUTE. | ITE, OPEN ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120JJ PX BYPASS INNOMINATE ARTERY TO RIGHT EXTRACRANIAL ARTERY WITH SYNTHE | TIC SUBS' ICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 03120JK PX BYPASS INNOMINATE ARTERY TO LEFT EXTRACRANIAL ARTERY WITH SYNTHET | IC SUBST ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120K0 PX BYPASS INNOMINATE ARTERY TO RIGHT UPPER ARM ARTERY WITH NONAUTOL | OGOUS TISICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 03120K1 PX BYPASS INNOMINATE ARTERY TO LEFT UPPER ARM ARTERY WITH NONAUTOLC | |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 03120K2 PX BYPASS INNOMINATE ARTERY TO BILATERAL UPPER ARM ARTERY WITH NONAL Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 03120K3 PX BYPASS INNOMINATE ARTERY TO RIGHT LOWER ARM ARTERY WITH NONAUTOL Cardiovascular event or intervention < 60 days prior to | OGOUS TI! ICD-10-PCS |
| 17 screening 03120K4 PX BYPASS INNOMINATE ARTERY TO LEFT LOWER ARM ARTERY WITH NONAUTOLO Cardiovascular event or intervention <60 days prior to | OGOUS TIS ICD-10-PCS |
| 17 screening 03120K5 PX BYPASS INNOMINATE ARTERY TO BILATERAL LOWER ARM ARTERY WITH NONA Cardiovascular event or intervention < 60 days prior to | UTOLOGO ICD-10-PCS |
| 17 screening 03120K6 PX BYPASS INNOMINATE ARTERY TO RIGHT UPPER LEG ARTERY WITH NONAUTOLO | GOUS TIS ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120K7 PX BYPASS INNOMINATE ARTERY TO LEFT UPPER LEG ARTERY WITH NONAUTOLOG | GOUS TISS ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120K8 PX BYPASS INNOMINATE ARTERY TO BILATERAL UPPER LEG ARTERY WITH NONAL | TOLOGOUICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 03120K9 PX BYPASS INNOMINATE ARTERY TO RIGHT LOWER LEG ARTERY WITH NONAUTOL ( 18 STEPPEN OF THE PROPERTY | OGOLIS TIS ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120KB PX BYPASS INNOMINATE ARTERY TO LEFT LOWER LEG ARTERY WITH NONAUTOLO | |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 03120KC PX BYPASS INNOMINATE ARTERY TO BILATERAL LOWER LEG ARTERY WITH NONAL Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 03120KD PX BYPASS INNOMINATE ARTERY TO UPPER ARM VEIN WITH NONAUTOLOGOUS TIS Cardiovascular event or intervention < 60 days prior to | SUE SUBSICD-10-PCS |
| 17 screening 03120KF PX BYPASS INNOMINATE ARTERY TO LOWER ARM VEIN WITH NONAUTOLOGOUS TIS<br>Cardiovascular event or intervention <60 days prior to | SSUE SUB!ICD-10-PCS |
| 17 screening 03120KJ PX BYPASS INNOMINATE ARTERY TO RIGHT EXTRACRANIAL ARTERY WITH NONAU | TOLOGOU! ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120KK PX BYPASS INNOMINATE ARTERY TO LEFT EXTRACRANIAL ARTERY WITH NONAUT | OLOGOUS ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120Z0 PX BYPASS INNOMINATE ARTERY TO RIGHT UPPER ARM ARTERY, OPEN APPROACI | H ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120Z1 PX BYPASS INNOMINATE ARTERY TO LEFT UPPER ARM ARTERY, OPEN APPROACH | ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 0312072 PX BYPASS INNOMINATE ARTERY TO BILATERAL UPPER ARM ARTERY, OPEN APPE | |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 03120Z3 PX BYPASS INNOMINATE ARTERY TO RIGHT LOWER ARM ARTERY, OPEN APPROAC Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 03120Z4 PX BYPASS INNOMINATE ARTERY TO LEFT LOWER ARM ARTERY, OPEN APPROACH Cardiovascular event or intervention < 60 days prior to | ICD-10-PCS |
| 17 screening 03120Z5 PX BYPASS INNOMINATE ARTERY TO BILATERAL LOWER ARM ARTERY, OPEN APPR Cardiovascular event or intervention <60 days prior to | ROACH ICD-10-PCS |
| 17 screening 03120Z6 PX BYPASS INNOMINATE ARTERY TO RIGHT UPPER LEG ARTERY, OPEN APPROACH | ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120Z7 PX BYPASS INNOMINATE ARTERY TO LEFT UPPER LEG ARTERY, OPEN APPROACH | ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120Z8 PX BYPASS INNOMINATE ARTERY TO BILATERAL UPPER LEG ARTERY, OPEN APPRI | DACH ICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 03120Z9 PX BYPASS INNOMINATE ARTERY TO RIGHT LOWER LEG ARTERY, OPEN APPROACH | I ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 03120ZB PX BYPASS INNOMINATE ARTERY TO LEFT LOWER LEG ARTERY, OPEN APPROACH | ICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 03120ZC PX BYPASS INNOMINATE ARTERY TO BILATERAL LOWER LEGARTERY, OPEN APPR | OACH ICD-10-PCS |


| Cardiovascular event or intervention < 60 days prior to 17 screening 051H0KY PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH NONAUTOLOGOUS TISSUE SUBSTITE OF THE PROPERTY OF THE PROPERTY OF THE PROPERTY OF THE PROPERTY OF T | |
|---|---|
| Cardiovascular event or intervention < 60 days prior to | UTE, OHCD-10-PCS |
| 17 screening 051H0ZY PX BYPASS LEFT HAND VEIN TO UPPER VEIN, OPEN APPROACH Cardiovascular event or intervention <60 days prior to | ICD-10-PCS |
| 17 screening 051H47Y PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSUE SUBSTITUTE Cardiovascular event or intervention <60 days prior to | PERCUICD-10-PCS |
| 17 screening 051H49Y PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH AUTOLOGOUS VENOUS TISSUE, PER | RCUTATICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051H4AY PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTERIAL TISSUE, PI | ERCUT ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051H4JY PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTITUTE, PERCUTA | NEOUSICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051H4KY PX BYPASS LEFT HAND VEIN TO UPPER VEIN WITH NONAUTOLOGOUS TISSUE SUBSTIT | UTE, PHCD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 051H4ZY PX BYPASS LEFT HAND VEIN TO UPPER VEIN, PERCUTANEOUS ENDOSCOPIC APPROA: | |
| Cardiovascular event or intervention <60 days prior to 17 screening 051L07Y PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSUE SUBSTIT | |
| Cardiovascular event or intervention <60 days prior to | |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 051L0AY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTERIAL TISSU Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 051L0JY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTITUTE, OPEN Cardiovascular event or intervention <60 days prior to | APPR(ICD-10-PCS |
| 17 screening 051L0KY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH NONAUTOLOGOUS TISSUE SUB Cardiovascular event or intervention <60 days prior to | STITUT ICD-10-PCS |
| 17 screening 051L0ZY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN, OPEN APPROACH Cardiovascular event or intervention <60 days prior to | ICD-10-PCS |
| 17 screening 051L47Y PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSUE SUBSTIT | UTE, PEICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening | PERCLICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051L4AY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTERIAL TISSU | E, PER(ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051L4JY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTITUTE, PERC | UTANE ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051L4KY PX BYPASS INTRACRANIAL VEINTO UPPER VEIN WITH NONAUTOLOGOUS TISSUE SUB | STITUTICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 051L4ZY PX BYPASS INTRACRANIAL VEIN TO UPPER VEIN, PERCUTANEOUS ENDOSCOPIC APPER | ROACH ICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 051M07Y PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSI | |
| Cardiovascular event or intervention <60 days prior to | |
| 17 screening 051M09Y PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS VENC<br>Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 051M0AY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTE Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 051M0JY PX BYPASS RIGHT INTERNAL JUGULAR VEINTO UPPER VEIN WITH SYNTHETIC SUBSTI<br>Cardiovascular event or intervention < 60 days prior to | TUTE, CICD-10-PCS |
| 17 screening 051M0KY PX BYPASS RIGHT INTERNAL JUGULAR VEINTO UPPER VEIN WITH NONAUTOLOGOUS Cardiovascular event or intervention < 60 days prior to | FISSUE ICD-10-PCS |
| 17 screening 051M0ZY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN, OPEN APPROACH Cardiovascular event or intervention < 60 days prior to | ICD-10-PCS |
| 17 screening 051M47Y PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSI Cardiovascular event or intervention < 60 days prior to | JE SUB ICD-10-PCS |
| 17 screening 051M49Y PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS VENC | OUS TIS ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051M4AY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTE | RIAL TICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051M4JY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTI | TUTE, FICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051M4KY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH NONAUTOLOGOUS | FISSUE ICD-10-PCS |
| Cardiovascular event or intervention <60 days prior to 17 screening 051M4ZY PX BYPASS RIGHT INTERNAL JUGULAR VEIN TO UPPER VEIN, PERCUTANEOUS ENDOS | COPIC /ICD-10-PCS |
| Cardiovascular event or intervention < 60 days prior to 17 screening 051N07Y PX BYPASS LEFT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS TISSU | |
| Cardiovascular event or intervention <60 days prior to | |
| Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 051N0AY PX BYPASS LEFT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH AUTOLOGOUS ARTEI Cardiovascular event or intervention < 60 days prior to | |
| 17 screening 051N0JY PX BYPASS LEFT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH SYNTHETIC SUBSTIT Cardiovascular event or intervention < 60 days prior to | UTE, OF ICD-10-PCS |
| 17 screening 051NOKY PX BYPASS LEFT INTERNAL JUGULAR VEIN TO UPPER VEIN WITH NONAUTOLOGOUS TI Cardiovascular event or intervention <60 days prior to | SSUE SICD-10-PCS |
| 17 screening D51NOZY PX BYPASS LEFT INTERNAL JUGULAR VEIN TO UPPER VEIN, OPEN APPROACH | ICD-10-PCS |


CEREBRAL INFARCTION DUE TO THROMBOSIS


CEREBRAL INFARCTION DUE TO EMBOLISM OF


CEREBRAL INFARCTION DUE TO UNSPECIFIED


PARASTOMAL HERNIA WITH OBSTRUCTION,


## Appendix 3. Flowchart for cohort assembly

| OPTUM (May 13, 2022 to Feb 28, 2025) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 95,349,410 |
| Patients meeting cohort entry criteria | | 563,099 |
| Excluded due to insufficient enrollment | -215,765 (38%) | 347,334 |
| Excluded due to prior use of referent | -116,754 (34%) | 230,580 |
| Excluded due to prior use of exposure | -157,852 (68%) | 72,728 |
| Excluded because patient qualified in >1 exposure category | -3 (<1%) | 72,725 |
| Excluded based on 1 - Age | -2,111 (3%) | 70,614 |
| Excluded based on 1 - Gender | -5 (<1%) | 70,609 |
| Excluded based on 2 - Type 2 diabetes mellitus | -4,665 (7%) | 65,944 |
| Excluded based on 4 - BMI ≥ 25kg/m2 (ICD-10) | -10,858 (16%) | 55,086 |
| Excluded based on 4 - BMI ≥ 25kg/m2 (Truncated) | -288 (<1%) | 54,798 |
| Excluded based on 5 - Established atherosclerotic cardiovascular disease | -15,096 (28%) | 39,702 |
| Excluded based on 7 - Planning treatment for diabetic retinopathy and/or macular edema | -582 (1%) | 39,120 |
| Excluded based on 8 - Hospitalized for chronic heart failure within 2 months prior to screening | -97 (<1%) | 39,023 |
| Excluded based on 11 - History of chronic or acute pancreatitis | -156 (<1%) | 38,867 |
| Excluded based on 12 - Known clinically significant gastric emptying abnormality or bariatric surgery | -1,941 (5%) | 36,926 |
| Excluded based on 13 - Liver disease (not including non-alcoholic fatty liver disease [NAFLD]) or ALT level ≥3X the ULN | -188 (<1%) | 36,738 |
| Excluded based on 14 - eGFR <15 mL/Min/1.73 m2 or on chronic dialysis | -260 (<1%) | 36,478 |
| Excluded based on 15 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -53 (<1%) | 36,425 |
| Excluded based on 17 - Cardiovascular event or intervention < 60 days prior to screening | -132 (<1%) | 36,293 |
| Excluded based on 18 - GLP-1-RA or pramlintide treatment within 3 months prior to Visit1 | -1,991 (5%) | 34,302 |
| Excluded based on 19 - Women who are pregnant or breastfeeding | -1 (<1%) | 34,301 |
| Patients in Exposure Group | | 20,311 |
| Patients in Referent Group | | 13,990 |
| Total Patients | | 34.301 |

| MARKETSCAN (May 13, 2022 to Dec 31, 2023) | | |
|---|---|---|
| | Excluded Patients | Remaining Patients |
| Patients in dataset | | 126,118,0 |
| Patients meeting cohort entry criteria | | 319,2 |
| Excluded due to insufficient enrollment | -62,500 (20%) | 256,7 |
| Excluded due to prior use of referent | -107,319 (42%) | 149,3 |
| Excluded due to prior use of exposure | -107,417 (72%) | 41,9 |
| Excluded because patient qualified in >1 exposure category | -6 (<1%) | 41,9 |
| Excluded based on 1 - Age | -4,476 (11%) | 37,4 |
| Excluded based on 1 - Gender | -0 (<1%) | 37,4 |
| Excluded based on 2 - Type 2 diabetes mellitus | -6,233 (17%) | 31,2 |
| Excluded based on 4 - BMI ≥ 25kg/m2 | -7,237 (23%) | 24,0 |
| Excluded based on 5 - Established atherosclerotic cardiovascular disease | -11,218 (47%) | 12,8 |
| Excluded based on 7 - Planning treatment for diabetic retinopathy and/or macular edema | -208 (2%) | 12,6 |
| Excluded based on 8 - Hospitalized for chronic heart failure within 2 months prior to screening | -53 (<1%) | 12,5 |
| Excluded based on 11 - History of chronic or acute pancreatitis | -35 (<1%) | 12,5 |
| Excluded based on 12 - Known clinically significant gastric emptying abnormality or bariatric surgery | -717 (6%) | 11,7 |
| Excluded based on 13 - Liver disease (not including non-alcoholic fatty liver disease [NAFLD]) or ALT level ≥3X the ULN | -42 (<1%) | 11,7 |
| Excluded based on 14 - eGFR <15 mL/Min/1.73 m2 or on chronic dialysis | -60 (<1%) | 11,6 |
| Excluded based on 15 - Family or personal history of multiple endocrine neoplasia or medullary thyroid carcinoma | -29 (<1%) | 11,6 |
| Excluded based on 17 - Cardiovascular event or intervention < 60 days prior to screening | -61 (<1%) | 11,6 |
| Excluded based on 18 - GLP-1-RA or pramlintide treatment within 3 months prior to Visit 1 | -1,154 (10%) | 10,4 |
| Excluded based on 19 - Women who are pregnant or breastfeeding | -5 (<1%) | 10,4 |
| Patients in Exposure Group | | 5,1 |
| Patients in Referent Group | | 5,3 |
| Total Patients | | 10,4 |

## Appendix 4.1st Feasibility Assessment

## Table of Contents

- A. Patient characteristics by treatment group
- B. Summary Parameters of Study Population
- C. Median Follow up Time in Overall Study Population
- D. Reasons for Censoring in Overall Study Population
- E. Initial Power Assessment
- F. Aetion report link
- G. Review by Principal Investigator

In order to complete the initial power analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

OPTUM: Study period from May 13, 2022 to Feb 28, 2025 MARKETSCAN: Study period from May 13, 2022 to Dec 31, 2023

## A. Patient characteristics by treatment group (follow-up start is 1 days after CED, so few patients and dropped, hence table 1 could include sightly fewer patients than the attrition table)

| Before matching | | Optum | | | Marketscan | |
|---|---|---|---|---|---|---|
| Variable | Reference- Dulaglutide | Exposure - Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 13,990 | 20,311 | - (-, -) | 5,329 | 5,116 | - (-, -) |
| Age | | | | | | |
| mean (sd) | 69.14 (9.06) | 66.92 (9.17) | 2.22 (2.02, 2.42) | 63.74 (10.60) | 59.86 (9.36) | 3.88 (3.50, 4.26) |
| median [IQR] | 70.00 [64.00, 75.00] | 68.00 [61.00, 73.00] | - (-, -) | 63.00 [56.00, 72.00] | 59.00 [53.00, 65.00] | - (-, -) |
| Gender | | | | | | |
| Male; n (%) | 6,883 (49.2%) | 9,605 (47.3%) | 1.9% (0.8%, 3.0%) | 2,885 (54.1%) | 2,538 (49.6%) | 4.5% (2.6%, 6.5%) |
| CCI (365 days) | | | | | | |
| mean (sd) | 3.57 (2.92) | 2.99 (2.68) | 0.58 (0.52, 0.64) | 2.34 (2.50) | 1.78 (2.02) | 0.57 (0.48, 0.65) |
| median [IQR] | 3.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | - (-, -) | 2.00 [1.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |

## B. Summary Parameters of Overall Study Population (Step 1)

| | Optum | Marketscan |
|-----------------------------------------------------|-----------|------------|
| Variable | Value | Value |
| Number of patients in full cohort | 34,301 | 10,445 |
| Number of patients dropped as incomplete cases | 0 | 0 |
| Number of patients that did not begin follow-up | 68 | 7 |
| Number of patients in analytic cohort | 34,233 | 10,438 |
| Number of events | 642 | 141 |
| Number of person-years | 16,569.35 | 4,748.51 |
| Number of patients in group: Reference- Sitagliptin | 13,970 | 5,324 |
| Number of patients in group: Exposure - Tirzepatide | 20,263 | 5,114 |
| Risk per 1,000 patients | 18.75 | 13.51 |
| Rate per 1,000 person-years | 38.75 | 29.69 |

## C. Median Follow up Time in Overall Study Population (Step 1)

| | Optum | Marketscan |
|---|---|---|
| Patient Group | Median Follow-Up<br>Time (Days) [IQR] | Median Follow-Up<br>Time (Days) [IQR] |
| Overall Patient Population | 140 [71, 274] | 136 [71, 253] |

## D. Reasons for Censoring in Overall Study Population (Step 1)

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 642 (1.9%) | 141 (1.4%) |
| Start of an additional exposure | 691 (2.0%) | 269 (2.6%) |
| End of index exposure | 14,259 (41.7%) | 2,853 (27.3%) |
| Maximum follow-up time | 5,529 (16.2%) | 1,101 (10.5%) |
| Specified date reached | 1,572 (4.6%) | 4,979 (47.7%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 9,197 (26.9%) | 637 (6.1%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 2,343 (6.8%) | 458 (4.4%) |

## E. Power Assessment

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|--------|------------|
| Number of patients matched | | |
| Reference | 13,990 | 5,329 |
| Exposed | 20,311 | 5,116 |
| Risk per 1,000 patients | 18.75 | 13.51 |
| Assumed HR from RCT | 0.8 | 0.8 |
| Alpha (2-sided) | 0.05 | 0.05 |
| Non-inferiority margin | 1.05 | 1.05 |
| Number of events expected | 643 | 141 |
| Power | 0.93 | 0.37 |

F. Aetion report link
Optum Step 1: https://bwb-dope.aetion.com/project/2905/cwrs/139334
Marketscan Step 1: https://bwh-dope.aetion.com/project/2906/rwrs/139338

## F. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|
|-----------------|-------------|----------------|---------------|

# Appendix 5. 2nd Feasibility Assessment

## Table of Contents

A. Median Follow up Time by Treatment Group

B. Reasons for Censoring by Treatment Group

C. Final Power Assessment

D. Aetion report link

E. Review by Principal Investigator

In order to complete the feasibility analysis, a dummy outcome of a 90-day gap in database enrollment was used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. We completed a PS overlap weighted comparative analysis using this outcome. The PS included all prespecified covariates listed in the protocol. Power calculations are based on the formulas from Chow et al. (2008).

# A. Median Follow Up Time by Treatment Group

| Patient Group | - | Median Follow-Up<br>Time (Days) [IQR] |
|---|---|---|
| Overall Patient Population | 140 [71, 274] | 136 [71, 253] |

# **B.** Reasons for Censoring in Overall Study Population

| | Optum | Marketscan |
|---|---|---|
| Overall | Value | Value |
| Outcome | 642 (1.9%) | 141 (1.4%) |
| Start of an additional exposure | 691 (2.0%) | 269 (2.6%) |
| End of index exposure | 14,259 (41.7%) | 2,853 (27.3%) |
| Maximum follow-up time | 5,529 (16.2%) | 1,101 (10.5%) |
| Specified date reached | 1,572 (4.6%) | 4,979 (47.7%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 9,197 (26.9%) | 637 (6.1%) |
| Switch to other GLP-1-RA (for censoring) / Nursing home admission | 2,343 (6.8%) | 458 (4.4%) |

## **C. Power Assessment**

| Noninferiority Analysis | Optum | Marketscan |
|----------------------------|-------|------------|
| Number of patients matched | | |
| Reference | 13,9 | 90 5,329 |
| Exposed | 20, | 311 5,116 |
| Risk per 1,000 patients | 18 | .75 13.51 |
| Assumed HR from RCT | | 0.8 |
| Alpha (2-sided) | 0 | .05 0.05 |
| Non-inferiority margin | 1 | .05 1.05 |
| Number of events expected | | 141 |
| Power | 0 | .93 0.37 |

# D. Aetion report link

Optum Step 1: https://bwh-dope.aetion.com/project/2905/rwrs/139334

Marketscan Step 1: https://bwh-dope.aetion.com/project/2906/rwrs/139338

# E. Review by principal investigator

Stop analyses until feasibility and power are reviewed by primary investigators.

| Reviewed by PI: | Nils Krüger | Date reviewed: | July 30, 2025 |
|-----------------|-------------|----------------|---------------|

Appendix 6. Balance Assessment - PS Distribution and C-Statistic

C-statistics unadjusted, OPTUM: 0.778



C-statistics adjusted after overlap weighing on the PS, OPTUM: 0.525



C-statistics unadjusted, MARKETSCAN: 0.751



C-statistics adjusted after overlap weighing on the PS, MARKETSCAN: 0.541



1.1

Appendix 7. Balance Assessment - Table 1

| | | | | | | _ |
|---|---|---|---|---|---|---|
| OPTUM | | | | | | |
| Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 13,970 | 20,263 | - (-, -) | 9,525 | 9,525 | - (-, -) |
| Year of Cohort Entry Date | | | | | | |
| 2022; n (%) | 4,345 (31.1%) | 1,352 (6.7%) | 24.4% (23.6%, 25.3%) | 1,298 (13.6%) | 1,293 (13.6%) | 0.1% (-0.9%, 1.0%) |
| 2023; n (%) | 6,094 (43.6%) | 7,976 (39.4%) | 4.3% (3.2%, 5.3%) | 4,859 (51.0%) | 4,821 (50.6%) | 0.4% (-1.0%, 1.8%) |
| 2024; n (%) | 3,495 (25.0%) | 10,644 (52.5%) | -27.5% (-28.5%, -26.5%) | 3,332 (35.0%) | 3,378 (35.5%) | -0.5% (-1.9%, 0.9%) |
| 2025; n (%) | 36 (0.3%) | 291 (1.4%) | -1.2% (-1.4%, -1.0%) | 36 (0.4%) | 33 (0.3%) | 0.0% (-0.1%, 0.2%) |
| Age | | | | | | |
| mean (sd) | 69.14 (9.05) | 66.92 (9.17) | 2.22 (2.03, 2.42) | 68.30 (9.05) | 68.31 (8.86) | -0.01 (-0.26, 0.24) |
| median [IQR] | 70.00 [64.00, 75.00] | 68.00 [61.00, 73.00] | - (-, -) | 69.00 [63.00, 75.00] | 69.00 [63.00, 74.00] | - (-, -) |
| min, max | 40.00, 88.00 | 40.00, 88.00 | - (-, -) | 40.00, 88.00 | 40.00, 88.00 | - (-, -) |
| Gender (male); n (%) | 6,873 (49.2%) | 9,584 (47.3%) | 1.9% (0.8%, 3.0%) | 4,620 (48.5%) | 4,647 (48.8%) | -0.3% (-1.7%, 1.1%) |
| Race (Recategorized) | | | | | | |
| White: n (%) | 6.463 (46.3%) | 10.227 (50.5%) | -4.2% (-5.3%, -3.1%) | 4.522 (47.5%) | 4.584 (48.1%) | -0.7% (-2.1%, 0.8%) |
| Black; n (%) | 2.182 (15.6%) | 2.567 (12.7%) | 3.0% (2.2%, 3.7%) | 1,404 (14,7%) | 1,370 (14,4%) | 0.4% (-0.7%, 1.4%) |
| Unknown / Missing; n (%) | 5,115 (36.6%) | 7,229 (35.7%) | 0.9% (-0.1%, 2.0%) | 3,471 (36.4%) | 3,455 (36.3%) | 0.2% (-1.2%, 1.5%) |
| Others; n (%) | 210 (1.5%) | 240 (1.2%) | 0.3% (0.1%, 0.6%) | 128 (1.3%) | 116 (1.2%) | 0.1% (-0.2%, 0.5%) |
| Region / State | (2070) | | | (2.070) | (1.2.70) | |
| Northest; n (%) | 1,502 (10.8%) | 1,665 (8.2%) | 2.5% (1.9%, 3.2%) | 895 (9.4%) | 912 (9.6%) | -0.2% (-1.0%, 0.7%) |
| | | | 2.3% (1.4%, 3.1%) | | | |
| Midwest / North central; n (%) | 2,830 (20.3%)<br>7,077 (50.7%) | 3,645 (18.0%)<br>12,397 (61.2%) | -10.5% (-11.6%, -9.4%) | 1,865 (19.6%)<br>5,204 (54.6%) | 1,875 (19.7%)<br>5,191 (54.5%) | -0.1% (-1.2%, 1.0%)<br>0.1% (-1.3%, 1.6%) |
| South; n (%) | | | | | | |
| West; n (%) | 2,555 (18.3%) | 2,547 (12.6%) | 5.7% (4.9%, 6.5%) | 1,558 (16.4%) | 1,544 (16.2%) | 0.1% (-0.9%, 1.2%) |
| Missing, n (%) | 6 (0.0%) | 9 (0.0%) | -0.0% (-0.0%, 0.0%) | 3 (0.0%) | 3 (0.0%) | 0.0% (-0.1%, 0.1%) |
| Smoking/Tobacco use; n (%) | 4,385 (31.4%) | 5,928 (29.3%) | 2.1% (1.1%, 3.1%) | 2,903 (30.5%) | 2,940 (30.9%) | -0.4% (-1.7%, 0.9%) |
| Weight | | | | | | |
| Overweight; n (%) | 1,719 (12.3%) | 1,346 (6.6%) | 5.7% (5.0%, 6.3%) | 943 (9.9%) | 932 (9.8%) | 0.1% (-0.7%, 1.0%) |
| Class 1 Obesity; n (%) | 3,478 (24.9%) | 4,061 (20.0%) | 4.9% (3.9%, 5.8%) | 2,221 (23.3%) | 2,226 (23.4%) | -0.1% (-1.3%, 1.2%) |
| Class 2 Obesity; n (%) | 4,497 (32.2%) | 7,185 (35.5%) | -3.3% (-4.3%, -2.2%) | 3,219 (33.8%) | 3,217 (33.8%) | 0.0% (-1.3%, 1.4%) |
| Class 3 Obesity; n (%) | 2,603 (18.6%) | 5,242 (25.9%) | -7.2% (-8.1%, -6.3%) | 1,992 (20.9%) | 1,972 (20.7%) | 0.2% (-1.0%, 1.4%) |
| Unspecified Obesity; n (%) | 1,673 (12.0%) | 2,429 (12.0%) | -0.0% (-0.7%, 0.7%) | 1,150 (12.1%) | 1,178 (12.4%) | -0.3% (-1.2%, 0.6%) |
| Diabetic retinopathy; n (%) | 2,355 (16.9%) | 2,393 (11.8%) | 5.0% (4.3%, 5.8%) | 1,449 (15.2%) | 1,416 (14.9%) | 0.3% (-0.7%, 1.4%) |
| Diabetic neuropathy; n (%) | 6,341 (45.4%) | 7,322 (36.1%) | 9.3% (8.2%, 10.3%) | 4,026 (42.3%) | 4,066 (42.7%) | -0.4% (-1.8%, 1.0%) |
| Diabetic nephropathy; n (%) | 5,201 (37.2%) | 5,712 (28.2%) | 9.0% (8.0%, 10.1%) | 3,229 (33.9%) | 3,239 (34.0%) | -0.1% (-1.5%, 1.3%) |
| Diabetes with other ophthalmic complications; n (%) | 987 (7.1%) | 1,027 (5.1%) | 2.0% (1.5%, 2.5%) | 580 (6.1%) | 593 (6.2%) | -0.1% (-0.8%, 0.6%) |
| Diabetes with peripheral circulatory disorders; n (%) | 4,024 (28.8%) | 4,517 (22.3%) | 6.5% (5.6%, 7.5%) | 2,492 (26.2%) | 2,471 (25.9%) | 0.2% (-1.0%, 1.5%) |
| Diabetic foot; n (%) | 905 (6.5%) | 960 (4.7%) | 1.7% (1.2%, 2.2%) | 556 (5.8%) | 549 (5.8%) | 0.1% (-0.6%, 0.7%) |
| Erectile dysfunction; n (%) | 742 (5.3%) | 1,149 (5.7%) | -0.4% (-0.9%, 0.1%) | 524 (5.5%) | 564 (5.9%) | -0.4% (-1.1%, 0.2%) |
| Hypoglycemia; n (%) | 4,402 (31.5%) | 5,630 (27.8%) | 3.7% (2.7%, 4.7%) | 2,862 (30.0%) | 2,899 (30.4%) | -0.4% (-1.7%, 0.9%) |
| Hyperglycemia/DKA/HONK; n (%) | 8,731 (62.5%) | 10,893 (53.8%) | 8.7% (7.7%, 9.8%) | 5,643 (59.2%) | 5,744 (60.3%) | -1.1% (-2.5%, 0.3%) |
| Skin infections; n (%) | 1,931 (13.8%) | 2,648 (13.1%) | 0.8% (0.0%, 1.5%) | 1,269 (13.3%) | 1,317 (13.8%) | -0.5% (-1.5%, 0.5%) |
| Stable angina; n (%) | 1,649 (11.8%) | 2,452 (12.1%) | -0.3% (-1.0%, 0.4%) | 1,128 (11.8%) | 1,165 (12.2%) | -0.4% (-1.3%, 0.5%) |
| Unstable angina; n (%) | 734 (5.3%) | 1.074 (5.3%) | -0.0% (-0.5%, 0.4%) | 512 (5.4%) | 505 (5.3%) | 0.1% (-0.6%, 0.7%) |
| Hypertension; n (%) | 13.207 (94.5%) | 18.911 (93.3%) | 1.2% (0.7%, 1.7%) | 8,962 (94.1%) | 8,962 (94.1%) | 0.0% (-0.7%, 0.7%) |
| Hypotension; n (%) | 890 (6.4%) | 958 (4.7%) | 1.6% (1.1%, 2.1%) | 525 (5.5%) | 543 (5.7%) | -0.2% (-0.9%, 0.5%) |
| Hyperlipidemia; n (%) | 12,648 (90.5%) | 18,288 (90.3%) | 0.3% (-0.4%, 0.9%) | 8,597 (90.3%) | 8,591 (90.2%) | 0.1% (-0.8%, 0.9%) |
| Atrial fibrillation; n (%) | | | | 1,619 (17.0%) | | |
| | 2,416 (17.3%) | 3,439 (17.0%) | 0.3% (-0.5%, 1.1%) | | 1,597 (16.8%) | 0.2% (-0.8%, 1.3%) |
| Cardiac conduction disorder; n (%) | 1,524 (10.9%) | 1,966 (9.7%) | 1.2% (0.5%, 1.9%) | 947 (9.9%) | 966 (10.1%) | -0.2% (-1.1%, 0.7%) |
| Previous cardiac procedure (CABG, PTCA, Stent); n (%) | 498 (3.6%) | 667 (3.3%) | 0.3% (-0.1%, 0.7%) | 329 (3.5%) | 340 (3.6%) | -0.1% (-0.6%, 0.4%) |
| Ischemic stroke; n (%) | 262 (1.9%) | 213 (1.1%) | 0.8% (0.6%, 1.1%) | 136 (1.4%) | 147 (1.5%) | -0.1% (-0.5%, 0.2%) |
| PVD diagnosis or surgery; n (%) | 3,769 (27.0%) | 4,719 (23.3%) | 3.7% (2.7%, 4.6%) | 2,423 (25.4%) | 2,401 (25.2%) | 0.2% (-1.0%, 1.5%) |
| Other cardiac dysrhythmia; n (%) | 4,213 (30.2%) | 6,097 (30.1%) | 0.1% (-0.9%, 1.1%) | 2,780 (29.2%) | 2,803 (29.4%) | -0.2% (-1.5%, 1.1%) |
| Cardiomyopathy; n (%) | 1,509 (10.8%) | 1,849 (9.1%) | 1.7% (1.0%, 2.3%) | 931 (9.8%) | 962 (10.1%) | -0.3% (-1.2%, 0.5%) |
| Valve disorders; n (%) | 2,716 (19.4%) | 3,780 (18.7%) | 0.8% (-0.1%, 1.6%) | 1,800 (18.9%) | 1,830 (19.2%) | -0.3% (-1.4%, 0.8%) |
| Valve replacement; n (%) | 344 (2.5%) | 465 (2.3%) | 0.2% (-0.2%, 0.5%) | 228 (2.4%) | 230 (2.4%) | -0.0% (-0.5%, 0.4%) |
| TIA; n (%) | 585 (4.2%) | 676 (3.3%) | 0.9% (0.4%, 1.3%) | 348 (3.7%) | 359 (3.8%) | -0.1% (-0.7%, 0.4%) |
| Edema; n (%) | 2,873 (20.6%) | 3,971 (19.6%) | 1.0% (0.1%, 1.8%) | 1,860 (19.5%) | 1,892 (19.9%) | -0.3% (-1.5%, 0.8%) |
| Venous thromboembolism / Pulmonary embolism; n (%) | 721 (5.2%) | 978 (4.8%) | 0.3% (-0.1%, 0.8%) | 458 (4.8%) | 451 (4.7%) | 0.1% (-0.5%, 0.7%) |
| Pulmonary hypertension; n (%) | 692 (5.0%) | 971 (4.8%) | 0.2% (-0.3%, 0.6%) | 455 (4.8%) | 453 (4.8%) | 0.0% (-0.6%, 0.6%) |
| Implantable cardioverter defibrillator; n (%) | 89 (0.6%) | 115 (0.6%) | 0.1% (-0.1%, 0.2%) | 66 (0.7%) | 64 (0.7%) | 0.0% (-0.2%, 0.3%) |

| Hyperkalemia; n (%) | 877 (6.3%) | 845 (4.2%) | 2.1% (1.6%, 2.6%) | 488 (5.1%) | 492 (5.2%) | -0.0% (-0.7%, 0.6%) |
|---|---|---|---|---|---|---|
| Coronary atherosclerosis; n (%) | 6,364 (45.6%) | 8,807 (43.5%) | 2.1% (1.0%, 3.2%) | 4,260 (44.7%) | 4,310 (45.2%) | -0.5% (-1.9%, 0.9%) |
| Cerebrovas cular procedure; n (%) | 50 (0.4%) | 40 (0.2%) | 0.2% (0.0%, 0.3%) | 26 (0.3%) | 30 (0.3%) | -0.0% (-0.2%, 0.1%) |
| Insertion of pacemakers / removal of cardiac lead; n (%) | 45 (0.3%) | 63 (0.3%) | 0.0% (-0.1%, 0.1%) | 31 (0.3%) | 22 (0.2%) | 0.1% (-0.1%, 0.3%) |
| CKD Stage 1-2; n (%) | 1,155 (8.3%) | 1,466 (7.2%) | 1.0% (0.4%, 1.6%) | 760 (8.0%) | 781 (8.2%) | -0.2% (-1.0%, 0.6%) |
| CKD Stage 3-4; n (%) | 4,124 (29.5%) | 4,550 (22.5%) | 7.1% (6.1%, 8.0%) | 2,545 (26.7%) | 2,539 (26.7%) | 0.1% (-1.2%, 1.3%) |
| Unspecified CKD; n (%) | 1,828 (13.1%) | 1,831 (9.0%) | 4.0% (3.4%, 4.7%) | 1,077 (11.3%) | 1,080 (11.3%) | -0.0% (-0.9%, 0.9%) |
| Acute kidney injury; n (%) | 1,815 (13.0%) | 1,747 (8.6%) | 4.4% (3.7%, 5.1%) | 1,033 (10.8%) | 1,032 (10.8%) | 0.0% (-0.9%, 0.9%) |
| Hypertensive nephropathy; n (%) | 3,494 (25.0%) | 3,802 (18.8%) | 6.2% (5.3%, 7.2%) | 2,133 (22.4%) | 2,108 (22.1%) | 0.3% (-0.9%, 1.5%) |
| Urinary tract infections; n (%) | 2,597 (18.6%) | 3,413 (16.8%) | 1.7% (0.9%, 2.6%) | 1,639 (17.2%) | 1,651 (17.3%) | -0.1% (-1.2%, 1.0%) |
| Genital infections; n (%) | 479 (3.4%) | 522 (2.6%) | 0.9% (0.5%, 1.2%) | 287 (3.0%) | 289 (3.0%) | -0.0% (-0.5%, 0.5%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 703 (5.0%) | 1,085 (5.4%) | -0.3% (-0.8%, 0.2%) | 460 (4.8%) | 481 (5.0%) | -0.2% (-0.8%, 0.4%) |
| COPD; n (%) | 2,827 (20.2%) | 3,648 (18.0%) | 2.2% (1.4%, 3.1%) | 1,811 (19.0%) | 1,840 (19.3%) | -0.3% (-1.4%, 0.8%) |
| Asthma; n (%) | 1,646 (11.8%) | 2,760 (13.6%) | -1.8% (-2.6%, -1.1%) | 1,163 (12.2%) | 1,195 (12.5%) | -0.3% (-1.3%, 0.6%) |
| Obstructive sleep apnea; n (%) | 4,591 (32.9%) | 8,250 (40.7%) | -7.9% (-8.9%, -6.8%) | 3,369 (35.4%) | 3,363 (35.3%) | 0.1% (-1.3%, 1.4%) |
| Serious bacterial infections; n (%) | 737 (5.3%) | 711 (3.5%) | 1.8% (1.3%, 2.2%) | 388 (4.1%) | 404 (4.2%) | -0.2% (-0.7%, 0.4%) |
| Pneumonia; n (%) | 1,089 (7.8%) | 1,152 (5.7%) | 2.1% (1.6%, 2.7%) | 598 (6.3%) | 611 (6.4%) | -0.1% (-0.8%, 0.6%) |
| Liver disease; n (%) | 2,680 (19.2%) | 3,932 (19.4%) | -0.2% (-1.1%, 0.6%) | 1,781 (18.7%) | 1,791 (18.8%) | -0.1% (-1.2%, 1.0%) |
| MASH/MASLD; n (%) | 1,113 (8.0%) | 2,040 (10.1%) | -2.1% (-2.7%, -1.5%) | 815 (8.6%) | 820 (8.6%) | -0.1% (-0.9%, 0.8%) |
| Fractures / Falls; n (%) | 1,237 (8.9%) | 1,358 (6.7%) | 2.2% (1.6%, 2.7%) | 724 (7.6%) | 749 (7.9%) | -0.3% (-1.0%, 0.5%) |
| Osteoporosis; n (%) | 896 (6.4%) | 1,117 (5.5%) | 0.9% (0.4%, 1.4%) | 583 (6.1%) | 580 (6.1%) | 0.0% (-0.7%, 0.7%) |
| Osteoarthritis; n (%) | 4,825 (34.5%) | 7,132 (35.2%) | -0.7% (-1.7%, 0.4%) | 3,286 (34.5%) | 3,274 (34.4%) | 0.1% (-1.2%, 1.5%) |
| Depression; n (%) | 3,470 (24.8%) | 4,496 (22.2%) | 2.7% (1.7%, 3.6%) | 2,199 (23.1%) | 2,230 (23.4%) | -0.3% (-1.5%, 0.9%) |
| Dementia; n (%) | 1,295 (9.3%) | 976 (4.8%) | 4.5% (3.9%, 5.0%) | 629 (6.6%) | 625 (6.6%) | 0.0% (-0.7%, 0.8%) |
| Delirium or psychosis; n (%) | 402 (2.9%) | 303 (1.5%) | 1.4% (1.1%, 1.7%) | 204 (2.1%) | 195 (2.0%) | 0.1% (-0.3%, 0.5%) |
| Anxiety; n (%) | 3,037 (21.7%) | 4,782 (23.6%) | -1.9% (-2.8%, -1.0%) | 2,079 (21.8%) | 2,112 (22.2%) | -0.3% (-1.5%, 0.8%) |
| Sleep disorders; n (%) | 5,422 (38.8%) | 8,113 (40.0%) | -1.2% (-2.3%, -0.2%) | 3,661 (38.4%) | 3,711 (39.0%) | -0.5% (-1.9%, 0.9%) |
| Anemia; n (%) | 3,828 (27.4%) | 4,932 (24.3%) | 3.1% (2.1%, 4.0%) | 2,457 (25.8%) | 2,455 (25.8%) | 0.0% (-1.2%, 1.3%) |
| Influenza; n (%) | 252 (1.8%) | 381 (1.9%) | -0.1% (-0.4%, 0.2%) | 177 (1.9%) | 175 (1.8%) | 0.0% (-0.4%, 0.4%) |
| COVID; n (%) | 1,860 (13.3%) | 2,345 (11.6%) | 1.7% (1.0%, 2.5%) | 1,144 (12.0%) | 1,143 (12.0%) | 0.0% (-0.9%, 0.9%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 4,034 (28.9%) | 6,266 (30.9%) | -2.0% (-3.0%, -1.1%) | 2,758 (29.0%) | 2,808 (29.5%) | -0.5% (-1.8%, 0.8%) |
| Hypothyroidism; n (%) | 3,264 (23.4%) | 4,979 (24.6%) | -1.2% (-2.1%, -0.3%) | 2,227 (23.4%) | 2,239 (23.5%) | -0.1% (-1.3%, 1.1%) |
| Nephrotic syndrome; n (%) | 27 (0.2%) | 27 (0.1%) | 0.1% (-0.0%, 0.2%) | 15 (0.2%) | 19 (0.2%) | -0.0% (-0.2%, 0.1%) |
| Urinary incontinence; n (%) | 1,224 (8.8%) | 1,486 (7.3%) | 1.4% (0.8%, 2.0%) | 760 (8.0%) | 782 (8.2%) | -0.2% (-1.0%, 0.6%) |
| Biliary disease; n (%) | 27 (0.2%) | 26 (0.1%) | 0.1% (-0.0%, 0.2%) | 17 (0.2%) | 18 (0.2%) | -0.0% (-0.1%, 0.1%) |
| Pancreatitis; n (%) | 10 (0.1%) | 10 (0.0%) | 0.0% (-0.0%, 0.1%) | 6 (0.1%) | 6 (0.1%) | 0.0% (-0.1%, 0.1%) |
| Bowel obstruction; n (%) | 24 (0.2%) | 39 (0.2%) | -0.0% (-0.1%, 0.1%) | 17 (0.2%) | 22 (0.2%) | -0.1% (-0.2%, 0.1%) |
| Gastroparesis; n (%) | 181 (1.3%) | 217 (1.1%) | 0.2% (-0.0%, 0.5%) | 108 (1.1%) | 113 (1.2%) | -0.1% (-0.4%, 0.3%) |
| Number of antidiabetic drugs on CED | | | | | | |
| mean (sd) | 2.39 (1.00) | 2.14 (0.99) | 0.25 (0.23, 0.27) | 2.31 (0.99) | 2.31 (1.02) | -0.01 (-0.04, 0.02) |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| min, max | 1.00, 7.00 | 1.00, 7.00 | - (-, -) | 1.00, 7.00 | 1.00, 7.00 | - (-, -) |
| Concomitant use or initiation of Metformin; n (%) | 6,322 (45.3%) | 8,597 (42.4%) | 2.8% (1.8%, 3.9%) | 4,267 (44.8%) | 4,268 (44.8%) | -0.0% (-1.4%, 1.4%) |
| Concomitant use or initiation of Insulins; n (%) | 4,659 (33.4%) | 4,855 (24.0%) | 9.4% (8.4%, 10.4%) | 2,816 (29.6%) | 2,887 (30.3%) | -0.7% (-2.1%, 0.6%) |
| Concomitant use or initiation of Sulfonylureas; n (%) | 3,225 (23.1%) | 3,076 (15.2%) | 7.9% (7.0%, 8.8%) | 1,929 (20.3%) | 1,961 (20.6%) | -0.3% (-1.5%, 0.8%) |
| Concomitant use or initiation of DPP-4i; n (%) | 1,147 (8.2%) | 1,256 (6.2%) | 2.0% (1.4%, 2.6%) | 681 (7.1%) | 663 (7.0%) | 0.2% (-0.5%, 0.9%) |
| Concomitant use or initiation of SGLT-2i; n (%) | 3,167 (22.7%) | 4,141 (20.4%) | 2.2% (1.3%, 3.1%) | 2,157 (22.6%) | 2,145 (22.5%) | 0.1% (-1.1%, 1.3%) |
| Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 879 (6.3%) | 1,205 (5.9%) | 0.3% (-0.2%, 0.9%) | 593 (6.2%) | 599 (6.3%) | -0.1% (-0.8%, 0.6%) |
| Past use of Metformin; n (%) | 8,549 (61.2%) | 11,782 (58.1%) | 3.1% (2.0%, 4.1%) | 5,756 (60.4%) | 5,743 (60.3%) | 0.1% (-1.3%, 1.5%) |
| Past use of Insulins; n (%) | 6,082 (43.5%) | 6,333 (31.3%) | 12.3% (11.2%, 13.3%) | 3,690 (38.7%) | 3,754 (39.4%) | -0.7% (-2.1%, 0.7%) |
| Past use of Sulfonylureas; n (%) | 4,475 (32.0%) | 4,483 (22.1%) | 9.9% (8.9%, 10.9%) | 2,729 (28.7%) | 2,772 (29.1%) | -0.5% (-1.7%, 0.8%) |
| Past use of DPP-4i; n (%) | 1,790 (12.8%) | 1,961 (9.7%) | 3.1% (2.4%, 3.8%) | 1,060 (11.1%) | 1,052 (11.0%) | 0.1% (-0.8%, 1.0%) |
| Past use of SGLT-2i; n (%) | 4,480 (32.1%) | 5,757 (28.4%) | 3.7% (2.7%, 4.7%) | 3,014 (31.6%) | 2,991 (31.4%) | 0.2% (-1.1%, 1.6%) |
| Past use of Any other glucose-lowering drugs; n (%) | 1,344 (9.6%) | 1,757 (8.7%) | 0.9% (0.3%, 1.6%) | 893 (9.4%) | 904 (9.5%) | -0.1% (-1.0%, 0.7%) |
| ACE-is/ARB's; n (%) | 10,492 (75.1%) | 14,817 (73.1%) | 2.0% (1.0%, 2.9%) | 7,111 (74.7%) | 7,102 (74.6%) | 0.1% (-1.2%, 1.3%) |
| ARNI; n (%) | 474 (3.4%) | 773 (3.8%) | -0.4% (-0.8%, -0.0%) | 350 (3.7%) | 354 (3.7%) | -0.0% (-0.6%, 0.5%) |
| Thiazides; n (%) | 4,386 (31.4%) | 6,881 (34.0%) | -2.6% (-3.6%, -1.5%) | 3,068 (32.2%) | 3,028 (31.8%) | 0.4% (-0.9%, 1.8%) |
| Beta-blockers; n (%) | 8,625 (61.7%) | 11,807 (58.3%) | 3.5% (2.4%, 4.5%) | 5,764 (60.5%) | 5,765 (60.5%) | -0.0% (-1.4%, 1.4%) |
| Calcium channel blockers; n (%) | 5,569 (39.9%) | 7,505 (37.0%) | 2.8% (1.8%, 3.9%) | 3,674 (38.6%) | 3,723 (39.1%) | -0.5% (-1.9%, 0.9%) |
| Calciant Charlier Blockers, 11(70) | | | | | | |
| Digoxin / Digitoxin; n (%) | 165 (1.2%) | 182 (0.9%) | 0.3% (0.1%, 0.5%) | 96 (1.0%) | 92 (1.0%) | 0.0% (-0.2%, 0.3%) |
| | 165 (1.2%)<br>4,225 (30.2%) | 182 (0.9%)<br>5,742 (28.3%) | 0.3% (0.1%, 0.5%)<br>1.9% (0.9%, 2.9%) | 96 (1.0%)<br>2,780 (29.2%) | 92 (1.0%)<br>2,772 (29.1%) | 0.0% (-0.2%, 0.3%) |

| Intravanaus diuratios: n (9/) | 343 (2.5%) | 450 (2.2%) | 0.2% (-0.1%, 0.6%) | 232 (2.4%) | 231 (2.4%) | 0.0% (-0.4%, 0.5%) |
|---|---|---|---|---|---|---|
| Intravenous diuretics; n (%) Nitrates: n (%) | 2.066 (14.8%) | 2.667 (13.2%) | 1.6% (0.9%, 2.4%) | 1,354 (14,2%) | 1,369 (14,4%) | -0.2% (-0.4%, 0.5%) |
| | | 7 | | | 7 | |
| Anti-arrhythmics; n (%) | 508 (3.6%) | 850 (4.2%) | -0.6% (-1.0%, -0.1%) | 351 (3.7%) | 361 (3.8%) | -0.1% (-0.7%, 0.4%) |
| Statins; n (%) | 12,221 (87.5%)<br>2,428 (17.4%) | 16,727 (82.5%)<br>3,905 (19.3%) | 4.9% (4.2%, 5.7%)<br>-1.9% (-2.7%, -1.1%) | 8,183 (85.9%) | 8,206 (86.2%)<br>1,772 (18.6%) | -0.2% (-1.2%, 0.8%)<br>-0.4% (-1.5%, 0.7%) |
| PCSK9 inhibitors and other lipid-lowering drugs; n (%) | | | | 1,737 (18.2%) | | |
| Antiplatelet medications; n (%) | 3,199 (22.9%) | 4,204 (20.7%) | 2.2% (1.3%, 3.1%) | 2,098 (22.0%) | 2,119 (22.2%) | -0.2% (-1.4%, 1.0%) |
| Oral anticoagulants; n (%) | 2,428 (17.4%) | 3,374 (16.7%) | 0.7% (-0.1%, 1.5%) | 1,589 (16.7%) | 1,571 (16.5%) | 0.2% (-0.9%, 1.3%) |
| COPD/Asthma medications; n (%) | 5,367 (38.4%) | 8,430 (41.6%) | -3.2% (-4.2%, -2.1%) | 3,762 (39.5%) | 3,769 (39.6%) | -0.1% (-1.5%, 1.3%) |
| NSAIDS; n (%) | 3,989 (28.6%) | 6,317 (31.2%) | -2.6% (-3.6%, -1.6%) | 2,793 (29.3%) | 2,770 (29.1%) | 0.2% (-1.1%, 1.5%) |
| Oral corticosteroids; n (%) | 3,202 (22.9%) | 5,850 (28.9%) | -5.9% (-6.9%, -5.0%) | 2,347 (24.6%) | 2,327 (24.4%) | 0.2% (-1.0%, 1.4%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 520 (3.7%) | 663 (3.3%) | 0.5% (0.0%, 0.9%) | 332 (3.5%) | 343 (3.6%) | -0.1% (-0.7%, 0.4%) |
| Opioids; n (%) | 3,569 (25.5%) | 5,416 (26.7%) | -1.2% (-2.1%, -0.2%) | 2,483 (26.1%) | 2,473 (26.0%) | 0.1% (-1.2%, 1.4%) |
| Anti-depressants; n (%) | 5,785 (41.4%) | 8,545 (42.2%) | -0.8% (-1.8%, 0.3%) | 3,930 (41.3%) | 3,942 (41.4%) | -0.1% (-1.5%, 1.3%) |
| Antipsychotics; n (%) | 800 (5.7%) | 935 (4.6%) | 1.1% (0.6%, 1.6%) | 479 (5.0%) | 479 (5.0%) | 0.0% (-0.6%, 0.6%) |
| Anxiolytics / hypnotics, benzos; n (%) | 2,785 (19.9%) | 4,920 (24.3%) | -4.3% (-5.2%, -3.5%) | 2,015 (21.2%) | 2,046 (21.5%) | -0.3% (-1.5%, 0.8%) |
| Dementia medications; n (%) | 524 (3.8%) | 410 (2.0%) | 1.7% (1.4%, 2.1%) | 262 (2.8%) | 274 (2.9%) | -0.1% (-0.6%, 0.4%) |
| Urinary tract infections antibiotics; n (%) | 6,916 (49.5%) | 10,578 (52.2%) | -2.7% (-3.8%, -1.6%) | 4,761 (50.0%) | 4,749 (49.9%) | 0.1% (-1.3%, 1.6%) |
| Laxatives; n (%) | 595 (4.3%) | 808 (4.0%) | 0.3% (-0.2%, 0.7%) | 393 (4.1%) | 392 (4.1%) | 0.0% (-0.6%, 0.6%) |
| Number of distinct medications | | | | | | |
| mean (sd) | 16.99 (7.03) | 16.34 (7.03) | 0.65 (0.50, 0.80) | 16.70 (7.01) | 16.74 (6.99) | -0.04 (-0.24, 0.16) |
| median [IQR] | 16.00 [12.00, 21.00] | 15.00 [11.00, 20.00] | - (-, -) | 16.00 [12.00, 21.00] | 16.00 [12.00, 21.00] | - (-, -) |
| min, max | 1.00, 64.00 | 1.00, 61.00 | - (-, -) | 1.00, 59.00 | 1.00, 61.00 | - (-, -) |
| Number of office visits | | | | | | |
| mean (sd) | 11.31 (7.61) | 11.86 (7.62) | -0.55 (-0.72, -0.39) | 11.50 (7.72) | 11.52 (7.32) | -0.02 (-0.23, 0.20) |
| median [IQR] | 10.00 [6.00, 15.00] | 10.00 [6.00, 16.00] | - (-, -) | 10.00 [6.00, 15.00] | 10.00 [6.00, 15.00] | - (-, -) |
| min, max | 0.00, 96.00 | 0.00, 80.00 | - (-, -) | 0.00.75.00 | 0.00, 80.00 | - (-, -) |
| Number of endocrinologist visits | , | 1 | , , | | | |
| mean (sd) | 0.63 (1.74) | 0.55 (1.52) | 0.08 (0.04, 0.12) | 0.61 (1.72) | 0.59 (1.60) | 0.01 (-0.03, 0.06) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 38.00 | 0.00, 36.00 | - (-, -) | 0.00, 38.00 | 0.00, 29.00 | - (-, -) |
| Number of cardiologist visits | 0.00, 30.00 | 0.00, 30.00 | (, ) | 0.00, 30.00 | 0.00, 23.00 | ( , / |
| mean (sd) | 2.70 (4.57) | 2.75 (4.24) | -0.05 (-0.15, 0.04) | 2.69 (4.59) | 2.73 (4.32) | -0.04 (-0.17, 0.08) |
| median [IQR] | 1.00 [0.00, 4.00] | 1.00 [0.00, 4.00] | - (-, -) | 1.00 [0.00, 4.00] | 1.00 [0.00, 4.00] | -() |
| min, max | 0.00, 90.00 | 0.00, 67.00 | - (-, -) | 0.00, 90.00 | 0.00, 67.00 | - (-, -)<br>- (-, -) |
| | 0.00, 90.00 | 0.00, 67.00 | - (-, -) | 0.00, 90.00 | 0.00, 67.00 | - (-, -) |
| Number of internal/family medicine visits | 10.10 (11.07) | 0.20 (0.02) | 1.04 (1.61.2.07) | 0.07/10.24) | 0.13 (10.06) | 0.00 ( 0.35, 0.33) |
| mean (sd) | 10.10 (11.87) | 8.26 (8.93) | 1.84 (1.61, 2.07) | 9.07 (10.24) | 9.13 (10.06) | -0.06 (-0.35, 0.22) |
| median [IQR] | 6.00 [3.00, 12.00] | 6.00 [3.00, 10.00] | - (-, -) | 6.00 [3.00, 11.00] | 6.00 [3.00, 11.00] | - (-, -) |
| min, max | 0.00, 281.00 | 0.00, 146.00 | - (-, -) | 0.00, 156.00 | 0.00, 146.00 | - (-, -) |
| Number of electrocardiograms (ECG/EKG) | | | | | | |
| mean (sd) | 1.48 (2.25) | 1.41 (1.96) | 0.07 (0.03, 0.12) | 1.43 (2.25) | 1.43 (1.93) | 0.00 (-0.06, 0.06) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 100.00 | 0.00, 59.00 | - (-, -) | 0.00, 100.00 | 0.00, 49.00 | - (-, -) |
| Number of echocardiograms | | | | | | |
| mean (sd) | 0.47 (0.85) | 0.46 (0.75) | 0.01 (-0.01, 0.03) | 0.46 (0.85) | 0.47 (0.75) | -0.01 (-0.03, 0.01) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 33.00 | 0.00, 9.00 | - (-, -) | 0.00, 33.00 | 0.00, 9.00 | - (-, -) |
| Out-of-pocket medication cost | | | | | | |
| mean (sd) | 697.86 (897.38) | 703.26 (992.89) | -5.40 (-25.61, 14.81) | 698.58 (924.58) | 700.52 (793.05) | -1.95 (-26.41, 22.52) |
| median [IQR] | 381.83 [126.64, 982.81] | 422.78 [150.35, 971.64] | - (-, -) | 387.10 [130.20, 974.48] | 420.00 [147.87, 986.68] | - (-, -) |
| min, max | 0.00, 19,723.93 | 0.00, 81,633.89 | - (-, -) | 0.00, 19,723.93 | 0.00, 13,088.53 | - (-, -) |
| Unique brand medicines | | | | | | |
| mean (sd) | 17.36 (7.33) | 16.62 (7.26) | 0.74 (0.58, 0.90) | 17.02 (7.28) | 17.07 (7.26) | -0.04 (-0.25, 0.16) |
| median [IQR] | 16.00 [12.00, 21.00] | 16.00 [11.00, 21.00] | - (-, -) | 16.00 [12.00, 21.00] | 16.00 [12.00, 21.00] | - (-, -) |
| min, max | 1.00, 66.00 | 1.00, 64.00 | - (-, -) | 1.00, 60.00 | 1.00, 64.00 | - (-, -) |
| Unique generic medicines | | | | | | |
| mean (sd) | 16.99 (7.03) | 16.34 (7.03) | 0.65 (0.50, 0.80) | 16.70 (7.01) | 16.74 (6.99) | -0.04 (-0.24, 0.16) |
| median [IQR] | 16.00 [12.00, 21.00] | 15.00 [11.00, 20.00] | - (-, -) | 16.00 [12.00, 21.00] | 16.00 [12.00, 21.00] | - (-, -) |
| min. max | 1.00, 64.00 | 1.00, 61.00 | - (-, -) | 1.00. 59.00 | 1.00, 61.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 1,453 (10.4%) | 2,364 (11.7%) | -1.3% (-1.9%, -0.6%) | 1,034 (10.9%) | 1,026 (10.8%) | 0.1% (-0.8%, 1.0%) |
| Flu Pneumococcal vaccine; n (%) | 5,059 (36.2%) | 6,428 (31.7%) | 4.5% (3.5%, 5.5%) | 3,285 (34.5%) | 3,305 (34.7%) | -0.2% (-1.6%, 1.2%) |
| Pap smear; n (%) | 505 (3.6%) | 1,096 (5.4%) | -1.8% (-2.2%, -1.3%) | 385 (4.0%) | 395 (4.1%) | -0.1% (-0.7%, 0.5%) |
| 1 ap 3 mour, n (70) | JUJ (J.U /U) | 1,000 (J.T /0) | 1.0 /0 (-2.2 /0, -1.3 /0) | JUJ (T.U /U) | JJJ (T.1/0) | U.170 (-U.170, U.J70) |

| PSA test: n (%) | 3,312 (23.7%) | 5,402 (26.7%) | -3.0% (-3.9%, -2.0%) | 2,373 (24.9%) | 2.408 (25.3%) | -0.4% (-1.6%, 0.9%) |
|---|---|---|---|---|---|---|
| Fecal occult blood test; n (%) | 724 (5.2%) | 877 (4.3%) | 0.9% (0.4%, 1.3%) | 441 (4.6%) | 464 (4.9%) | -0.2% (-0.9%, 0.4%) |
| Bone mineral density tests; n (%) | 1,132 (8.1%) | 1,800 (8.9%) | -0.8% (-1.4%, -0.2%) | 791 (8.3%) | 813 (8.5%) | -0.2% (-1.0%, 0.6%) |
| Mammograms; n (%) | 3,012 (21.6%) | 5,293 (26.1%) | -4.6% (-5.5%, -3.6%) | 2,215 (23.3%) | 2,192 (23.0%) | 0.2% (-1.0%, 1.4%) |
| Telemedicine; n (%) | 3,299 (23.6%) | 4,875 (24.1%) | -0.4% (-1.4%, 0.5%) | 2,167 (22.8%) | 2,165 (22.7%) | 0.0% (-1.2%, 1.2%) |
| HbA1c tests | 3,233 (23.070) | 4,073 (24.170) | 0.470 ( 1.470, 0.370) | 2,107 (22.070) | 2,103 (22.170) | 0.070 ( 1.270, 1.270) |
| mean (sd) | 2.63 (1.40) | 2.47 (1.40) | 0.16 (0.13, 0.19) | 2.58 (1.38) | 2.58 (1.45) | 0.00 (-0.04, 0.04) |
| median [IQR] | 3.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) | 3.00 [2.00, 3.00] | 3.00 [2.00, 3.00] | - (-, -) |
| min, max | 0.00, 24.00 | 0.00, 44.00 | - (-, -) | 0.00, 24.00 | 0.00, 44.00 | - (-, -)<br>- (-, -) |
| Lipid panels | 0.00, 24.00 | 0.00, 44.00 | - (-, -) | 0.00, 24.00 | 0.00, 44.00 | - (-, -) |
| mean (sd) | 1.71 (1.25) | 1.81 (1.27) | -0.10 (-0.12, -0.07) | 1.74 (1.25) | 1.76 (1.25) | -0.01 (-0.05, 0.02) |
| median [IQR] | 2.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | - (-, -) |
| min, max | 0.00, 15.00 | 0.00, 26.00 | - (-, -) | 0.00, 12.00 | 0.00, 11.00 | - (-, -)<br>- (-, -) |
| | 0.00, 15.00 | 0.00, 26.00 | - (-, -) | 0.00, 12.00 | 0.00, 11.00 | - (-, -) |
| Creatinine tests | 2.02 (4.17) | 2.55 (2.47) | 0.20 (0.20 0.47) | 2.70 (2.00) | 2.74 (2.06) | 0.04 ( 0.07, 0.10) |
| mean (sd) | 3.93 (4.17)<br>3.00 [2.00, 5.00] | 3.55 (3.47)<br>3.00 [2.00, 5.00] | 0.38 (0.30, 0.47) | 3.78 (3.88) | 3.74 (3.96) | 0.04 (-0.07, 0.16) |
| median [IQR] | | | - (-, -) | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | - (-, -) |
| min, max | 0.00, 181.00 | 0.00, 127.00 | - (-, -) | 0.00, 177.00 | 0.00, 127.00 | - (-, -) |
| Natriuretic peptide tests | 0.00 (0.00) | 0.07/0.00 | 0.00/0.00.00# | 0.00 (0.00) | 0.00 (0.70) | 0.01 / 0.00 0.00 |
| mean (sd) | 0.29 (0.86) | 0.27 (0.83) | 0.02 (-0.00, 0.04) | 0.28 (0.86) | 0.28 (0.79) | 0.01 (-0.02, 0.03) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 28.00 | 0.00, 28.00 | - (-, -) | 0.00, 28.00 | 0.00, 15.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.31 (1.89) | 1.30 (1.84) | 0.01 (-0.03, 0.05) | 1.28 (1.89) | 1.30 (1.84) | -0.01 (-0.07, 0.04) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 34.00 | 0.00, 24.00 | - (-, -) | 0.00, 34.00 | 0.00, 23.00 | - (-, -) |
| Combined comorbidity score | | | | | | |
| mean (sd) | 3.56 (2.91) | 2.99 (2.68) | 0.57 (0.51, 0.64) | 3.27 (2.72) | 3.29 (2.80) | -0.02 (-0.10, 0.06) |
| median [IQR] | 3.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | - (-, -) | 3.00 [1.00, 5.00] | 3.00 [1.00, 5.00] | - (-, -) |
| min, max | -1.00, 20.00 | -2.00, 21.00 | - (-, -) | -1.00, 17.00 | -2.00, 21.00 | - (-, -) |
| Frailty Score | | | | | | |
| mean (sd) | 0.20 (0.07) | 0.19 (0.06) | 0.01 (0.01, 0.01) | 0.19 (0.06) | 0.19 (0.06) | -0.00 (-0.00, 0.00) |
| median [IQR] | 0.19 [0.15, 0.23] | 0.18 [0.15, 0.22] | - (-, -) | 0.18 [0.15, 0.22] | 0.18 [0.15, 0.22] | - (-, -) |
| min, max | 0.06, 0.57 | 0.06, 0.61 | - (-, -) | 0.06, 0.54 | 0.06, 0.61 | - (-, -) |
| Number of Hospitalizations | | | | | | |
| mean (sd) | 0.38 (0.97) | 0.25 (0.70) | 0.13 (0.12, 0.15) | 0.30 (0.82) | 0.31 (0.80) | -0.00 (-0.03, 0.02) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 17.00 | 0.00, 12.00 | - (-, -) | 0.00, 15.00 | 0.00, 12.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 986 (7.1%) | 855 (4.2%) | 2.8% (2.3%, 3.4%) | 522 (5.5%) | 520 (5.5%) | 0.0% (-0.6%, 0.7%) |
| Any hospitalization within prior 92-365 days; n (%) | 2,508 (18.0%) | 2,773 (13.7%) | 4.3% (3.5%, 5.1%) | 1,466 (15.4%) | 1,504 (15.8%) | -0.4% (-1.4%, 0.6%) |
| Number of hospitalizations (0, 1, 2 or more) | | | | | | |
| < 1; n (%) | 10,923 (78.2%) | 17,004 (83.9%) | -5.7% (-6.6%, -4.9%) | 7,755 (81.4%) | 7,726 (81.1%) | 0.3% (-0.8%, 1.4%) |
| 1 - <2; n (%) | 1,900 (13.6%) | 2,235 (11.0%) | 2.6% (1.9%, 3.3%) | 1,171 (12.3%) | 1,185 (12.4%) | -0.1% (-1.1%, 0.8%) |
| >= 2; n (%) | 1,147 (8.2%) | 1,024 (5.1%) | 3.2% (2.6%, 3.7%) | 599 (6.3%) | 614 (6.4%) | -0.2% (-0.9%, 0.5%) |
| Heart failure hospitalization; n (%) | 1,013 (7.3%) | 1,059 (5.2%) | 2.0% (1.5%, 2.6%) | 592 (6.2%) | 591 (6.2%) | 0.0% (-0.7%, 0.7%) |
| ED visit; n (%) | 5,921 (42.4%) | 7,218 (35.6%) | 6.8% (5.7%, 7.8%) | 3,741 (39.3%) | 3,779 (39.7%) | -0.4% (-1.8%, 1.0%) |
| Acute MI; n (%) | 340 (2.4%) | 388 (1.9%) | 0.5% (0.2%, 0.8%) | 204 (2.1%) | 198 (2.1%) | 0.1% (-0.4%, 0.5%) |
| Old MI; n (%) | 1,672 (12.0%) | 1,938 (9.6%) | 2.4% (1.7%, 3.1%) | 1,028 (10.8%) | 1,059 (11.1%) | -0.3% (-1.2%, 0.6%) |
| Heart failure; n (%) | 3,768 (27.0%) | 4,852 (23.9%) | 3.0% (2.1%, 4.0%) | 2,398 (25.2%) | 2,428 (25.5%) | -0.3% (-1.6%, 0.9%) |
| Acute heart failure; n (%) | 926 (6.6%) | 1,032 (5.1%) | 1.5% (1.0%, 2.1%) | 558 (5.9%) | 564 (5.9%) | -0.1% (-0.7%, 0.6%) |
| Microalbuminuria or proteinuria; n (%) | 1,309 (9.4%) | 1,586 (7.8%) | 1.5% (0.9%, 2.2%) | 867 (9.1%) | 843 (8.9%) | 0.3% (-0.6%, 1.1%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.02 (0.03) | 0.00 (0.00, 0.01) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.03] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.86, 1.46 | 0.91, 1.40 | - (-, -) | 0.92, 1.43 | 0.91, 1.40 | - (-, -) |

Appendix 7. Balance Assessment - Table 1

| | | | ı | ı | I | |
|---|---|---|---|---|---|---|
| MARKETSCAN | | | | | | |
| Variable | Reference: Dulaglutide | Exposure: Tirzepatide | Difference | Reference: Dulaglutide | Exposure: Tirzepatide | Difference |
| Number of patients | 5,324 | 5,114 | - (-, -) | 3,297 | 3,297 | - (-, -) |
| Year of Cohort Entry Date | | | | | | |
| 2022; n (%) | 2,327 (43.7%) | 855 (16.7%) | 27.0% (25.3%, 28.7%) | 788 (23.9%) | 812 (24.6%) | -0.7% (-2.8%, 1.4%) |
| 2023; n (%) | 2,997 (56.3%) | 4,259 (83.3%) | -27.0% (-28.7%, -25.3%) | 2,509 (76.1%) | 2,485 (75.4%) | 0.7% (-1.4%, 2.8%) |
| Age | | | | | | |
| mean (sd) | 63.74 (10.60) | 59.86 (9.36) | 3.88 (3.50, 4.26) | 61.27 (9.90) | 61.28 (9.70) | -0.02 (-0.49, 0.45) |
| median [IQR] | 63.00 [56.00, 72.00] | 59.00 [53.00, 65.00] | - (-, -) | 61.00 [54.00, 68.00] | 61.00 [55.00, 68.00] | - (-, -) |
| min, max | 40.00, 95.00 | 40.00, 96.00 | - (-, -) | 40.00, 95.00 | 40.00, 96.00 | - (-, -) |
| Gender (male); n (%) | 2,882 (54.1%) | 2,537 (49.6%) | 4.5% (2.6%, 6.5%) | 1,720 (52.2%) | 1,712 (51.9%) | 0.2% (-2.2%, 2.7%) |
| Region / State | | | | | | |
| .Northeast; n (%) | 635 (11.9%) | 538 (10.5%) | 1.4% (0.2%, 2.6%) | 367 (11.1%) | 374 (11.3%) | -0.2% (-1.8%, 1.3%) |
| .Widwest / North central; n (%) | 2,215 (41.6%) | 1,352 (26.4%) | 15.2% (13.4%, 17.0%) | 1,100 (33.4%) | 1,099 (33.3%) | 0.0% (-2.3%, 2.3%) |
| South: n (%) | 2.179 (40.9%) | 2,974 (58.2%) | -17.2% (-19.1%, -15.3%) | 1,650 (50.0%) | 1.649 (50.0%) | 0.0% (-2.4%, 2.5%) |
| West: n(%) | 289 (5.4%) | 244 (4.8%) | 0.7% (-0.2%, 1.5%) | 176 (5.3%) | 171 (5,2%) | 0.2% (-1.0%, 1.3%) |
| Missing; n (%) | 6 (0.1%) | 6 (0.1%) | -0.0% (-0.1%, 0.1%) | 4 (0.1%) | 4 (0.1%) | 0.0% (-0.2%, 0.2%) |
| imoking / Tobacco use; n (%) | 808 (15.2%) | 697 (13.6%) | 1.5% (0.2%, 2.9%) | 466 (14.1%) | 481 (14.6%) | -0.5% (-2.2%, 1.3%) |
| Veight | 000 (10.270) | 33. (13.070) | 2.0 ,0 (0.2 /0, 2.3 /0) | .55 (17.170) | 102 (17.070) | 5.570 ( Z.Z/0, 1.370) |
| Overweight; n (%) | 813 (15.3%) | 440 (8.6%) | 6.7% (5.4%, 7.9%) | 352 (10.7%) | 347 (10.5%) | 0.2% (-1.4%, 1.7%) |
| | 569 (10.7%) | 425 (8.3%) | 2.4% (1.2%, 3.5%) | 312 (9.5%) | 302 (9.2%) | |
| Class 1 Obesity; n (%) | , , | | | | | 0.3% (-1.1%, 1.7%) |
| Class 2 Obesity; n (%) | 326 (6.1%) | 342 (6.7%) | -0.6% (-1.5%, 0.4%) | 223 (6.8%) | 220 (6.7%) | 0.1% (-1.1%, 1.3%) |
| Class 3 Obesity; n (%) | 1,205 (22.6%) | 990 (19.4%) | 3.3% (1.7%, 4.9%) | 691 (21.0%) | 689 (20.9%) | 0.1% (-1.9%, 2.1%) |
| Unspecified Obesity; n (%) | 2,411 (45.3%) | 2,917 (57.0%) | -11.8% (-13.7%, -9.8%) | 1,719 (52.1%) | 1,739 (52.7%) | -0.6% (-3.0%, 1.8%) |
| biabetic retinopathy; n (%) | 706 (13.3%) | 494 (9.7%) | 3.6% (2.4%, 4.8%) | 360 (10.9%) | 361 (10.9%) | -0.0% (-1.6%, 1.5%) |
| iabetic neuropathy; n (%) | 1,830 (34.4%) | 1,283 (25.1%) | 9.3% (7.5%, 11.0%) | 966 (29.3%) | 953 (28.9%) | 0.4% (-1.8%, 2.6%) |
| iabetic nephropathy; n (%) | 1,327 (24.9%) | 837 (16.4%) | 8.6% (7.0%, 10.1%) | 620 (18.8%) | 621 (18.8%) | -0.0% (-1.9%, 1.9%) |
| iabetes with other opthalmic complications; n (%) | 152 (2.9%) | 114 (2.2%) | 0.6% (0.0%, 1.2%) | 77 (2.3%) | 88 (2.7%) | -0.3% (-1.1%, 0.5%) |
| iabetes with peripheral circulatory disorders; n (%) | 975 (18.3%) | 702 (13.7%) | 4.6% (3.2%, 6.0%) | 515 (15.6%) | 498 (15.1%) | 0.5% (-1.3%, 2.3%) |
| liabetic foot; n (%) | 223 (4.2%) | 151 (3.0%) | 1.2% (0.5%, 2.0%) | 120 (3.6%) | 116 (3.5%) | 0.1% (-0.8%, 1.0%) |
| rectile dysfunction; n (%) | 246 (4.6%) | 247 (4.8%) | -0.2% (-1.0%, 0.6%) | 158 (4.8%) | 169 (5.1%) | -0.3% (-1.4%, 0.7%) |
| lypoglycemia; n (%) | 1,231 (23.1%) | 1,038 (20.3%) | 2.8% (1.2%, 4.4%) | 722 (21.9%) | 698 (21.2%) | 0.7% (-1.3%, 2.7%) |
| Hyperglycemia/DKA/HONK; n (%) | 3,122 (58.6%) | 2,649 (51.8%) | 6.8% (4.9%, 8.8%) | 1,816 (55.1%) | 1,811 (54.9%) | 0.2% (-2.3%, 2.6%) |
| ikin infections; n (%) | 680 (12.8%) | 585 (11.4%) | 1.3% (0.1%, 2.6%) | 388 (11.8%) | 380 (11.5%) | 0.2% (-1.3%, 1.8%) |
| stable angina; n (%) | 507 (9.5%) | 400 (7.8%) | 1.7% (0.6%, 2.8%) | 274 (8.3%) | 288 (8.7%) | -0.4% (-1.8%, 1.0%) |
| Instable angina; n (%) | 270 (5.1%) | 200 (3.9%) | 1.2% (0.3%, 2.0%) | 144 (4.4%) | 145 (4.4%) | -0.0% (-1.0%, 1.0%) |
| Typertension; n (%) | 4,842 (90.9%) | 4,556 (89.1%) | 1.9% (0.7%, 3.0%) | 2,960 (89.8%) | 2,955 (89.6%) | 0.2% (-1.3%, 1.6%) |
| Typotension; n (%) | 211 (4.0%) | 104 (2.0%) | 1.9% (1.3%, 2.6%) | 79 (2.4%) | 84 (2.5%) | -0.2% (-0.9%, 0.6%) |
| Typerlipidemia; n (%) | 4,642 (87.2%) | 4,451 (87.0%) | 0.2% (-1.2%, 1.5%) | 2,859 (86.7%) | 2,882 (87.4%) | -0.7% (-2.3%, 1.0%) |
| trial fibrillation; n (%) | 755 (14.2%) | 556 (10.9%) | 3.3% (2.0%, 4.6%) | 391 (11.9%) | 390 (11.8%) | 0.0% (-1.6%, 1.6%) |
| Cardiac conduction disorder; n (%) | 432 (8.1%) | 266 (5.2%) | 2.9% (1.9%, 3.9%) | 191 (5.8%) | 197 (6.0%) | -0.2% (-1.3%, 1.0%) |
| revious cardiac procedure (CABG, PTCA, Stent); n (%) | 220 (4.1%) | 155 (3.0%) | 1.1% (0.4%, 1.8%) | 115 (3.5%) | 117 (3.5%) | -0.1% (-1.0%, 0.9%) |
| schemic stroke: n (%) | 144 (2.7%) | 78 (1.5%) | 1.2% (0.6%, 1.7%) | 64 (1.9%) | 60 (1.8%) | 0.1% (-0.6%, 0.8%) |
| VD diagnosis or surgery; n (%) | 928 (17.4%) | 733 (14.3%) | 3.1% (1.7%, 4.5%) | 507 (15.4%) | 519 (15.7%) | -0.4% (-2.1%, 1.4%) |
| | 1,367 (25.7%) | 1,202 (23.5%) | 2.2% (0.5%, 3.8%) | 773 (23.4%) | 775 (23.5%) | , , |
| Other cardiac dysrhythmia; n (%) | | | | | | -0.1% (-2.1%, 2.0%) |
| Cardiomyopathy; n (%) | 452 (8.5%) | 339 (6.6%) | 1.9% (0.8%, 2.9%) | 243 (7.4%) | 245 (7.4%) | -0.1% (-1.4%, 1.2%) |
| /alve disorders; n (%) | 796 (15.0%) | 622 (12.2%) | 2.8% (1.5%, 4.1%) | 432 (13.1%) | 430 (13.0%) | 0.1% (-1.6%, 1.7%) |
| /alve replacement; n (%) | 88 (1.7%) | 50 (1.0%) | 0.7% (0.2%, 1.1%) | 40 (1.2%) | 41 (1.2%) | -0.0% (-0.6%, 0.5% |
| TA; n (%) | 176 (3.3%) | 148 (2.9%) | 0.4% (-0.3%, 1.1%) | 96 (2.9%) | 91 (2.8%) | 0.2% (-0.7%, 1.0%) |
| dema; n (%) | 708 (13.3%) | 597 (11.7%) | 1.6% (0.3%, 2.9%) | 390 (11.8%) | 396 (12.0%) | -0.2% (-1.8%, 1.4%) |
| enous thromboembolism / Pulmonary embolism; n (%) | 229 (4.3%) | 172 (3.4%) | 0.9% (0.2%, 1.7%) | 121 (3.7%) | 129 (3.9%) | -0.2% (-1.2%, 0.7%) |
| ulmonary hypertension; n (%) | 130 (2.4%) | 104 (2.0%) | 0.4% (-0.2%, 1.0%) | 66 (2.0%) | 60 (1.8%) | 0.2% (-0.5%, 0.9%) |
| nplantable cardioverter defibrillator, n (%) | 37 (0.7%) | 20 (0.4%) | 0.3% (0.0%, 0.6%) | 17 (0.5%) | 15 (0.5%) | 0.1% (-0.3%, 0.4%) |
| yperkalemia; n (%) | 180 (3.4%) | 82 (1.6%) | 1.8% (1.2%, 2.4%) | 66 (2.0%) | 63 (1.9%) | 0.1% (-0.6%, 0.8%) |
| oronary atherosclerosis; n (%) | 2,104 (39.5%) | 1,695 (33.1%) | 6.4% (4.5%, 8.2%) | 1,182 (35.9%) | 1,174 (35.6%) | 0.2% (-2.1%, 2.6%) |
| erebrovascular procedure; n (%) | 11 (0.2%) | 7 (0.1%) | 0.1% (-0.1%, 0.2%) | 5 (0.2%) | 5 (0.2%) | 0.0% (-0.2%, 0.2%) |
| nsertion of pacemakers / removal of cardiac lead; n (%) | 15 (0.3%) | 2 (0.0%) | 0.2% (0.1%, 0.4%) | 4 (0.1%) | 2 (0.1%) | 0.1% (-0.1%, 0.2%) |
| KD stage 1-2; n (%) | 188 (3.5%) | 151 (3.0%) | 0.6% (-0.1%, 1.3%) | 109 (3.3%) | 112 (3.4%) | -0.1% (-1.0%, 0.8%) |
| CKD stage 3-4; n (%) | 879 (16.5%) | 480 (9.4%) | 7.1% (5.8%, 8.4%) | 378 (11.5%) | 381 (11.6%) | -0.1% (-1.7%, 1.5%) |
| Inspecified CKD; n (%) | | 160 (3.1%) | 2.6% (1.8%, 3.4%) | 130 (3.9%) | 127 (3.9%) | 0.1% (-0.9%, 1.1%) |
| mapeomeu GND, IT (70) | JUJ (J.170) | 100 (3.170) | Z.U /0 (1.0 70, J.4 70) | 100 (3.270) | 121 (3.370) | 0.170 (-0.370, 1.170) |

| Acute kidney injury; n (%) | 433 (8.1%) | 207 (4.0%) | 4.1% (3.2%, 5.0%) | 168 (5.1%) | 164 (5.0%) | 0.1% (-1.0%, 1.2%) |
|---|---|---|---|---|---|---|
| Hypertensive nephropathy: n (%) | 743 (14.0%) | 421 (8,2%) | 5.7% (4.5%, 6.9%) | 338 (10.3%) | 321 (9.7%) | 0.5% (-1.0%, 2.0%) |
| Urinary tract infections; n (%) | 656 (12.3%) | 626 (12.2%) | 0.1% (-1.2%, 1.4%) | 389 (11.8%) | 374 (11.3%) | 0.5% (-1.1%, 2.0%) |
| Genital infections; n (%) | 175 (3.3%) | 161 (3.1%) | 0.1% (-0.6%, 0.8%) | 114 (3.5%) | 117 (3.5%) | -0.1% (-1.0%, 0.8%) |
| Urolithiasis (Kidney and urinary stone); n (%) | 237 (4.5%) | 223 (4.4%) | 0.1% (-0.7%, 0.9%) | 138 (4.2%) | 138 (4.2%) | 0.0% (-1.0%, 1.0%) |
| COPD; n (%) | 583 (11.0%) | 448 (8.8%) | 2.2% (1.0%, 3.4%) | 311 (9.4%) | 310 (9.4%) | 0.0% (-1.4%, 1.5%) |
| Asthma; n (%) | 494 (9.3%) | 541 (10.6%) | -1.3% (-2.5%, -0.1%) | 330 (10.0%) | 312 (9.5%) | 0.5% (-0.9%, 2.0%) |
| Obstructive sleep apnea; n (%) | 1,820 (34.2%) | 1,974 (38.6%) | -4.4% (-6.3%, -2.6%) | 1,204 (36.5%) | 1,176 (35.7%) | 0.8% (-1.5%, 3.2%) |
| Serious bacterial infections; n (%) | 290 (5.4%) | 167 (3.3%) | 2.2% (1.4%, 3.0%) | 134 (4.1%) | 115 (3.5%) | 0.6% (-0.4%, 1.5%) |
| Pneumonia: n (%) | 294 (5.5%) | 202 (3.9%) | 1.6% (0.7%, 2.4%) | 150 (4.5%) | 133 (4.0%) | 0.5% (-0.5%, 1.5%) |
| Liver disease; n (%) | 763 (14.3%) | 799 (15.6%) | -1.3% (-2.7%, 0.1%) | 445 (13.5%) | 469 (14.2%) | -0.7% (-2.4%, 1.0%) |
| MASH/MASLD; n (%) | 367 (6.9%) | 438 (8.6%) | -1.7% (-2.7%, -0.6%) | 238 (7.2%) | 246 (7.5%) | -0.2% (-1.5%, 1.0%) |
| Fractures / Falls; n (%) | 300 (5.6%) | 201 (3.9%) | 1.7% (0.9%, 2.5%) | 148 (4.5%) | 150 (4.5%) | -0.1% (-1.1%, 1.0%) |
| Osteoporosis; n (%) | 138 (2.6%) | 95 (1.9%) | 0.7% (0.2%, 1.3%) | 78 (2.4%) | 70 (2.1%) | 0.2% (-0.5%, 1.0%) |
| Osteoarthritis; n (%) | 1,372 (25.8%) | 1,268 (24.8%) | 1.0% (-0.7%, 2.7%) | 841 (25.5%) | 824 (25.0%) | 0.5% (-1.6%, 2.6%) |
| Depression; n (%) | 880 (16.5%) | 803 (15.7%) | 0.8% (-0.6%, 2.3%) | 515 (15.6%) | 520 (15.8%) | -0.2% (-1.9%, 1.6%) |
| Dementia; n (%) | 251 (4.7%) | 97 (1.9%) | 2.8% (2.1%, 3.5%) | 75 (2.3%) | 82 (2.5%) | -0.2% (-1.0%, 0.6%) |
| Delirium or psychosis; n (%) | 49 (0.9%) | 25 (0.5%) | 0.4% (0.1%, 0.8%) | 23 (0.7%) | 20 (0.6%) | 0.1% (-0.3%, 0.5%) |
| Anxiety; n (%) | 937 (17.6%) | 1,053 (20.6%) | -3.0% (-4.5%, -1.5%) | 613 (18.6%) | 624 (18.9%) | -0.3% (-2.2%, 1.6%) |
| Sleep disorders; n (%) | 1,410 (26.5%) | 1,502 (29.4%) | -2.9% (-4.6%, -1.1%) | 901 (27.3%) | 917 (27.8%) | -0.5% (-2.7%, 1.7%) |
| Anemia; n (%) | 1,166 (21.9%) | 1,029 (20.1%) | 1.8% (0.2%, 3.4%) | 652 (19.8%) | 656 (19.9%) | -0.1% (-2.1%, 1.8%) |
| Influenza; n (%) | 83 (1.6%) | 136 (2.7%) | -1.1% (-1.7%, -0.5%) | 63 (1.9%) | 57 (1.7%) | 0.2% (-0.5%, 0.9%) |
| COVID: n (%) | 790 (14.8%) | 748 (14.6%) | 0.2% (-1.2%, 1.6%) | 487 (14.8%) | 470 (14.3%) | 0.5% (-1.2%, 2.2%) |
| Hyperthyroidism and other thyroid gland disorders; n (%) | 1,328 (24.9%) | 1,400 (27.4%) | -2.4% (-4.1%, -0.7%) | 839 (25.4%) | 860 (26.1%) | -0.6% (-2.8%, 1.5%) |
| Hypothyroidism; n (%) | 1,014 (19.0%) | 1,067 (20.9%) | -1.8% (-3.4%, -0.3%) | 639 (19.4%) | 675 (20.5%) | -1.1% (-3.1%, 0.9%) |
| Nephrotic syndrome; n (%) | 7 (0.1%) | 1(0.0%) | 0.1% (-0.0%, 0.2%) | 2 (0.1%) | 1 (0.0%) | 0.0% (-0.1%, 0.2%) |
| Urinary incontinence; n (%) | 257 (4.8%) | 191 (3.7%) | 1.1% (0.3%, 1.9%) | 134 (4.1%) | 121 (3.7%) | 0.4% (-0.6%, 1.4%) |
| Biliary disease; n (%) | 30 (0.6%) | 11 (0.2%) | 0.3% (0.1%, 0.6%) | 7 (0.2%) | 7 (0.2%) | 0.0% (-0.2%, 0.2%) |
| Pancreatitis; n (%) | 2 (0.0%) | 4 (0.1%) | -0.0% (-0.2%, 0.1%) | 2 (0.1%) | 1 (0.0%) | 0.0% (-0.1%, 0.2%) |
| Bowel obstruction; n (%) | 22 (0.4%) | 10 (0.2%) | 0.2% (-0.0%, 0.4%) | 10 (0.3%) | 10 (0.3%) | 0.0% (-0.3%, 0.3%) |
| Gastroparesis; n (%) | 38 (0.7%) | 48 (0.9%) | -0.2% (-0.6%, 0.1%) | 24 (0.7%) | 27 (0.8%) | -0.1% (-0.5%, 0.4%) |
| Number of antidiabetic drugs on CED | | , , | | | | |
| mean (sd) | 2.32 (1.05) | 2.18 (1.01) | 0.15 (0.11, 0.19) | 2.27 (1.03) | 2.27 (1.03) | -0.00 (-0.05, 0.05) |
| median [IQR] | 2.00 [2.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [2.00, 3.00] | 2.00 [2.00, 3.00] | - (-, -) |
| | | 2.00 [1.00, 3.00]<br>1.00, 7.00 | - (-, -)<br>- (-, -) | 2.00 [2.00, 3.00]<br>1.00, 6.00 | 2.00 [2.00, 3.00]<br>1.00, 7.00 | |
| median [IQR] | 2.00 [2.00, 3.00] | | | | | - (-, -) |
| median [IQR]min, max | 2.00 [2.00, 3.00]<br>1.00, 6.00 | 1.00, 7.00 | - (-, -) | 1.00, 6.00 | 1.00, 7.00 | - (-, -)<br>- (-, -) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2,418 (45.4%) | 1.00, 7.00<br>2,402 (47.0%) | - (-, -)<br>-1.6% (-3.5%, 0.4%) | 1.00, 6.00<br>1,564 (47.4%) | 1.00, 7.00<br>1,570 (47.6%) | - (-, -)<br>- (-, -)<br>-0.2% (-2.6%, 2.3%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2,418 (45.4%)<br>1,554 (29.2%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%) | - (-, -)<br>- (-, -)<br>-0.2% (-2.6%, 2.3%)<br>0.2% (-1.9%, 2.3%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1,554 (29.2%)<br>984 (18.5%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%) | - (-, -)<br>- (-, -)<br>-0.2% (-2.6%, 2.3%)<br>0.2% (-1.9%, 2.3%)<br>0.2% (-1.5%, 2.0%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%) | -(-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%) | - (-, -)<br>- (-, -)<br>-0.2% (-2.6%, 2.3%)<br>0.2% (-1.9%, 2.3%)<br>0.2% (-1.5%, 2.0%)<br>-0.1% (-1.5%, 1.3%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4I; n (%) Concomitant use or initiation of SGLT-2I; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1.320 (24.8%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%) | - (-, -)<br>- (-, -)<br>- 0.2% (-2.6%, 2.3%)<br>0.2% (-1.5%, 2.3%)<br>0.2% (-1.5%, 2.3%)<br>-0.1% (-1.5%, 1.3%)<br>-0.3% (-2.5%, 1.8%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4!; n (%) Concomitant use or initiation of SGLT-2!; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%) | -(-, -)<br>-(-, -)<br>-0.2% (-2.6%, 2.3%)<br>0.2% (-1.9%, 2.3%)<br>0.2% (-1.5%, 2.0%)<br>-0.1% (-1.5%, 1.3%)<br>-0.3% (-2.5%, 1.8%)<br>0.1% (-1.0%, 1.1%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1,554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%) | 1.00, 7.00<br>2,402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1.296 (25.3%)<br>217 (4.2%)<br>3,263 (63.8%) | -(-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%) | - (-, -)<br>- (-, -)<br>- 0.2% (-2.6%, 2.3%)<br>0.2% (-1.5%, 2.3%)<br>0.2% (-1.5%, 2.0%)<br>- 0.1% (-1.5%, 1.3%)<br>- 0.3% (-2.5%, 1.8%)<br>0.1% (-1.0%, 1.1%)<br>- 0.4% (-2.7%, 2.0%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%) | 1.00, 7.00<br>2,402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1.296 (25.3%)<br>217 (4.2%)<br>3.263 (63.8%)<br>1,421 (27.8%) | -(-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%)<br>12.4% (10.6%, 14.2%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%) | - (·, ·)<br>- (·, ·)<br>-0.2% (-2.6%, 2.3%)<br>0.2% (-1.5%, 2.3%)<br>0.2% (-1.5%, 1.3%)<br>-0.1% (-1.5%, 1.3%)<br>-0.3% (-2.5%, 1.8%)<br>0.1% (-1.0%, 1.1%)<br>-0.4% (-2.7%, 2.0%)<br>0.2% (-2.1%, 2.5%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1,554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%)<br>1,414 (26.6%) | 1.00, 7.00<br>2.402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1.296 (25.3%)<br>217 (4.2%)<br>3.263 (63.8%)<br>1,421 (27.8%)<br>889 (17.4%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%)<br>12.4% (10.6%, 14.2%)<br>9.2% (7.6%, 10.8%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%)<br>699 (21.2%) | - (·, ·) - (·, ·) - (·, ·) - (·, ·) - 0.2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.3%) 0.2% (-1.5%, 1.3%) - 0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) - 0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-2.1%, 2.5%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of DPP-4i; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%)<br>1,414 (26.6%)<br>775 (14.6%) | 1.00, 7.00<br>2,402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%)<br>3,263 (63.8%)<br>1,421 (27.8%)<br>889 (17.4%)<br>661 (12.9%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%)<br>12.4% (10.6%, 14.2%)<br>9.2% (7.6%, 10.8%)<br>1.6% (0.3%, 3.0%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%)<br>699 (21.2%)<br>459 (13.9%) | -(-, -) -(-, - |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; n (%) Past use of SGLT-2i; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%)<br>1,414 (26.6%)<br>775 (14.6%)<br>1,794 (33.7%) | 1.00, 7.00<br>2.402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%)<br>3,263 (63.8%)<br>1,421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1,674 (32.7%) | - (-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%)<br>12.4% (10.6%, 14.2%)<br>9.2% (7.6%, 10.8%)<br>1.6% (0.3%, 3.0%)<br>1.0% (-0.9%, 2.8%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1.100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1.139 (34.5%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1.094 (33.2%)<br>699 (21.2%)<br>459 (13.9%)<br>1,150 (34.9%) | -(-, -) -(-, -) -(-, -) -(2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.0%) 0.2% (-1.5%, 2.0%) -0.1% (-1.5%, 1.3%) -0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) -0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-1.8%, 2.8%) 0.1% (-1.6%, 1.8%) -0.3% (-2.7%, 2.0%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of SGLT-2i; n (%) Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1.320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%)<br>1,414 (26.6%)<br>775 (14.6%)<br>1,794 (33.7%)<br>414 (7.8%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%)<br>3,263 (63.8%)<br>1,421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1,674 (32.7%)<br>303 (5.9%) | -(-, -)<br>-1.6% (-3.5%, 0.4%)<br>7.9% (6.2%, 9.6%)<br>6.9% (5.5%, 8.3%)<br>0.9% (-0.2%, 2.0%)<br>-0.5% (-2.2%, 1.1%)<br>1.1% (0.3%, 1.9%)<br>0.8% (-1.1%, 2.6%)<br>12.4% (10.6%, 1.4.2%)<br>9.2% (7.6%, 10.8%)<br>1.6% (0.3%, 3.0%)<br>1.0% (-0.9%, 2.8%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%)<br>699 (21.2%)<br>459 (13.9%)<br>1,150 (34.9%)<br>218 (6.6%) | -(-, -) -(-, - |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; n (%) Past use of SPP-4i; n (%) Past use of SPP-4i; n (%) Past use of SPP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1,320 (24.8%)<br>285 (5.4%)<br>3.437 (64.6%)<br>2,139 (40.2%)<br>1,414 (26.6%)<br>775 (14.6%)<br>1,794 (33.7%)<br>414 (7.8%)<br>3,923 (73.7%) | 1.00, 7.00<br>2,402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%)<br>3,263 (63.8%)<br>1,421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1,674 (32.7%)<br>303 (5.9%)<br>3,642 (71.2%) | - (-, -) -1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 11%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 1.4.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 1.9% (0.9%, 2.8%) 2.5% (0.7%, 4.2%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>2,392 (72.6%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%)<br>699 (21.2%)<br>459 (13.9%)<br>1,150 (34.9%)<br>218 (6.6%)<br>2,363 (71.7%) | -(·,·) -(·,·) -(·,·) -(·,·) -0.2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.0%) -0.1% (-1.5%, 1.3%) -0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) -0.4% (-2.7%, 2.0%) 0.2% (-1.1%, 2.5%) 0.2% (-1.1%, 2.5%) 0.3% (-2.7%, 2.0%) -0.3% (-2.7%, 2.0%) -0.2% (-1.4%, 1.0%) 0.9% (-1.3%, 3.1%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SoLT-2; n (%) Concomitant use or initiation of SoLT-2; n (%) Concomitant use or initiation of SoLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of DPP-4; n (%) Past use of DPP-4; n (%) Past use of SoLT-2; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) | 2.00 [2.00, 3.00]<br>1.00, 6.00<br>2.418 (45.4%)<br>1.554 (29.2%)<br>984 (18.5%)<br>481 (9.0%)<br>1.320 (24.8%)<br>285 (5.4%)<br>3,437 (64.6%)<br>2,139 (40.2%)<br>1.414 (26.6%)<br>775 (14.6%)<br>1,794 (33.7%)<br>414 (7.8%)<br>3,923 (73.7%)<br>188 (3.5%) | 1.00, 7.00<br>2.402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1.296 (25.3%)<br>217 (4.2%)<br>3.263 (63.8%)<br>1.421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1.674 (32.7%)<br>303 (5.9%)<br>3,642 (71.2%)<br>168 (3.3%) | - (-, -) -1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 1.9% (0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1.100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>2,392 (72.6%)<br>110 (3.3%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1.094 (33.2%)<br>699 (21.2%)<br>459 (13.9%)<br>1.150 (34.9%)<br>218 (6.6%)<br>2,363 (71.7%)<br>119 (3.6%) | -(·,·) -(·,·) -(·,·) -(·,·) -(·,·) -0.2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.3%) 0.2% (-1.5%, 2.0%) -0.1% (-1.5%, 1.3%) -0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) -0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-1.8%, 2.2%) 0.1% (-1.6%, 1.8%) -0.3% (-2.7%, 2.0%) 0.2% (-1.4%, 1.0%) 0.9% (-1.3%, 3.1%) -0.3% (-1.2%, 0.6%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of DPP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2,418 (45.4%) 1,554 (29.2%) 984 (18.5%) 481 (9.0%) 1,320 (24.8%) 285 (5.4%) 3,437 (64.6%) 2,139 (40.2%) 1,414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3,923 (73.7%) 188 (3.5%) 1,700 (31.9%) | 1.00, 7.00<br>2.402 (47.0%)<br>1.089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1.296 (25.3%)<br>217 (4.2%)<br>3.263 (63.8%)<br>1.421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1.674 (32.7%)<br>303 (5.9%)<br>3.642 (71.2%)<br>168 (3.3%)<br>1,753 (34.3%) | - (·, ·) -1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 1.9% (0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) -2.3% (-4.2%, -0.5%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>22392 (72.6%)<br>110 (3.3%)<br>1,076 (32.6%) | 1.00, 7.00<br>1,570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2,144 (65.0%)<br>1,094 (33.2%)<br>459 (13.9%)<br>1,150 (34.9%)<br>218 (6.6%)<br>2,363 (71.7%)<br>119 (3.6%)<br>1,089 (33.0%) | - (-, -) - (-, -) - (-, -) - (-, -) - (-, -) - (-) (-2.6%, 2.3%) 0.2% (-1.9%, 2.3%) 0.2% (-1.5%, 2.3%) 0.1% (-1.5%, 1.3%) - 0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) - 0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-1.8%, 2.2%) 0.1% (-1.6%, 1.8%) - 0.3% (-2.7%, 2.0%) - 0.2% (-1.4%, 1.0%) 0.9% (-1.3%, 3.1%) - 0.3% (-1.2%, 0.6%) - 0.4% (-2.7%, 1.9%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of SUlfonylureas; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1.414 (26.6%) 775 (14.6%) 1.794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) | 1.00, 7.00<br>2.402 (47.0%)<br>1,089 (21.3%)<br>592 (11.6%)<br>417 (8.2%)<br>1,296 (25.3%)<br>217 (4.2%)<br>3.263 (63.8%)<br>1.421 (27.8%)<br>889 (17.4%)<br>661 (12.9%)<br>1,674 (32.7%)<br>303 (5.9%)<br>3,642 (71.2%)<br>168 (3.3%)<br>1,753 (34.3%)<br>2,743 (53.6%) | -(-, -) -(-, - | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>2,392 (72.6%)<br>1,076 (32.6%)<br>1,847 (56.0%) | 1.00, 7.00<br>1.570 (47.6%)<br>827 (25.1%)<br>473 (14.3%)<br>293 (8.9%)<br>882 (26.8%)<br>154 (4.7%)<br>2.144 (65.0%)<br>1.094 (33.2%)<br>699 (21.2%)<br>459 (13.9%)<br>1.150 (34.9%)<br>218 (6.6%)<br>2.363 (71.7%)<br>119 (3.6%)<br>1,089 (33.0%)<br>1,866 (56.6%) | - (-, -) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SDIT-2i; n (%) Past use of SP-4i; n (%) Past use of SP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARN; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1,320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2,139 (40.2%) 1,414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3,923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) | 1.00, 7.00 2,402 (47.0%) 1,089 (21.3%) 592 (11.6%) 417 (8.2%) 1,296 (25.3%) 217 (4.2%) 3,263 (63.8%) 1,421 (27.8%) 889 (17.4%) 661 (12.9%) 1,674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) | -(-, -) -(-, - | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1,100 (33.4%)<br>766 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>2,392 (72.6%)<br>110 (3.3%)<br>1,076 (32.6%)<br>1,847 (56.0%)<br>1,112 (33.7%) | 1.00, 7.00 1,570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 699 (21.2%) 459 (13.9%) 1,150 (34.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) | - (·, ·) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SP-4i; n (%) Past use of Sp-4i; n (%) Past use of S | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1.414 (26.6%) 775 (14.6%) 1.794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3.187 (59.9%) 1,921 (36.1%) 54 (1.0%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) 36 (0.7%) | - (-, -) -1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) 2.3% (-4.2%, 0.5%) 6.2% (4.3%, 8.1%) 4.0% (2.2%, 5.8%) 0.3% (-0.1%, 0.7%) | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>2,132 (72.6%)<br>110 (3.3%)<br>1,076 (32.6%)<br>1,847 (56.0%)<br>1,112 (33.7%)<br>20 (0.6%) | 1.00, 7.00 1.570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 699 (21.2%) 459 (13.9%) 1,150 (34.9%) 2,18 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) | - (·, ·) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2i; n (%) Past | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3,437 (64.6%) 2,139 (40.2%) 1.414 (26.6%) 775 [14.6%) 1,794 (33.7%) 414 (7.8%) 3,923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) 54 (1.0%) 1,226 (23.0%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3.642 (71.2%) 168 (3.3%) 1.753 (34.3%) 2,743 (53.6%) 1.641 (32.1%) 36 (0.7%) 940 (18.4%) | -(-, -) -(-, - | 1.00, 6.00<br>1.564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2.132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>10 (3.3%)<br>1,076 (32.6%)<br>1,847 (56.0%)<br>1,12 (33.7%)<br>20 (0.6%)<br>637 (19.3%) | 1.00, 7.00 1,570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 699 (21.2%) 459 (13.9%) 1,150 (34.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) | - (-, -) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of SP-4i; n (%) Past use of SP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Other diuretics; n (%) Other diuretics; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1,414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) 54 (1.0%) 1,226 (23.0%) 564 (10.6%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) | -(·, -) -(·, - | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>2,132 (64.7%)<br>1,100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>229 (72.6%)<br>110 (3.3%)<br>1,076 (32.6%)<br>1,847 (56.0%)<br>1,112 (33.7%)<br>20 (0.6%)<br>637 (19.3%)<br>352 (10.7%) | 1.00, 7.00 1,570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 459 (13.9%) 1,150 (34.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) | - (-, -) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SQLT-2i; n (%) Concomitant use or initiation of SQLT-2i; n (%) Concomitant use or initiation of SQLT-2i; n (%) Past use of Metformin; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SQLT-2i; n (%) Past use of | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1.414 (26.6%) 775 (14.6%) 1.794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1.700 (31.9%) 3.187 (59.9%) 1.921 (36.1%) 54 (1.0%) 54 (1.0%) 78 (1.5%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3.642 (71.2%) 168 (3.3%) 1.753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) 52 (1.0%) | -(-, -) 1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 1.9% (0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) 2.3% (-4.2%, -0.5%) 6.2% (4.3%, 8.1%) 4.0% (2.2%, 5.8%) 0.3% (-0.1%, 0.7%) 4.6% (3.1%, 6.2%) 0.0% (-1.2%, 1.2%) 0.4% (0.0%, 0.9%) | 1.00, 6.00<br>1,564 (47.4%)<br>833 (25.3%)<br>481 (14.6%)<br>290 (8.8%)<br>871 (26.4%)<br>156 (4.7%)<br>1.100 (33.4%)<br>706 (21.4%)<br>463 (14.0%)<br>1,139 (34.5%)<br>212 (6.4%)<br>2,392 (72.6%)<br>110 (3.3%)<br>1,076 (32.6%)<br>1,847 (56.0%)<br>1,112 (33.7%)<br>20 (0.6%)<br>637 (19.3%)<br>352 (10.7%)<br>33 (1.0%) | 1.00, 7.00 1.570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2.144 (65.0%) 1.094 (33.2%) 699 (21.2%) 459 (13.9%) 1.150 (34.9%) 218 (6.6%) 2.363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) 34 (10.3%) | - (·, ·) - ( |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of SP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of SPP-4i; n (%) Past use of SPP-4i; n (%) Past use of SPP-4i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ACE-is/ARB's; n (%) Thizaides; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Calcium channel blockers; n (%) Unitrates; n (%) Intravenous diuretics; n (%) Nitrates; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1,320 (24.8%) 285 (5.4%) 3,437 (64.6%) 2,139 (40.2%) 1,414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3,923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) 54 (1.0%) 1,226 (23.0%) 564 (10.6%) 78 (1.5%) | 1.00, 7.00 2.402 (47.0%) 1,089 (21.3%) 592 (11.6%) 417 (8.2%) 1,296 (25.3%) 217 (4.2%) 3,263 (63.8%) 1,421 (27.8%) 889 (17.4%) 661 (12.9%) 1,674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) 52 (1.0%) | -(-, -) -(-, - | 1.00, 6.00 1,564 (47.4%) 833 (25.3%) 481 (14.6%) 290 (8.8%) 871 (26.4%) 156 (4.7%) 2,132 (64.7%) 1,100 (33.4%) 706 (21.4%) 463 (14.0%) 2,139 (72.6%) 110 (3.3%) 1,076 (32.6%) 1,12 (33.7%) 20 (0.6%) 637 (19.3%) 352 (10.7%) 33 (1.0%) 414 (12.6%) | 1.00, 7.00 1,570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 699 (21.2%) 459 (13.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) 34 (10.3%) 411 (12.5%) | -(·, ·) -(·, ·) -(·, ·) -(·, ·) -(·, ·) -0.2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.0%) 0.1% (-1.5%, 1.3%) -0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) -0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-1.1%, 2.5%) 0.2% (-1.1%, 2.5%) 0.3% (-2.2%, 2.0%) -0.3% (-2.7%, 2.0%) -0.3% (-1.2%, 0.0%) -0.3% (-1.2%, 0.6%) -0.4% (-2.7%, 1.9%) -0.6% (-2.5%, 0.5%) -0.1% (-0.5%, 0.3%) -0.6% (-2.5%, 0.3%) -0.6% (-2.5%, 0.5%) 0.1% (-1.5%, 1.7%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SOLT-2; n (%) Concomitant use or initiation of SOLT-2; n (%) Concomitant use or initiation of SOLT-2; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Insulins; n (%) Past use of Sulfonylureas; n (%) Past use of PP-4; n (%) Past use of SPP-4; n (%) Past use of Sulfonylureas; n (%) P | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1.414 (26.6%) 775 (14.6%) 1.794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3.187 (59.9%) 1.921 (36.1%) 54 (1.0%) 1.226 (23.0%) 564 (10.6%) 78 (1.5%) 764 (14.4%) 184 (3.5%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1.641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) 521 (10.9%) 171 (3.3%) | -(-, -) 1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) 2.3% (-4.2%, -0.5%) 6.2% (4.3%, 8.1%) 4.0% (2.2%, 5.8%) 0.3% (-0.1%, 0.7%) 4.6% (3.1%, 6.2%) 0.0% (-1.2%, 1.2%) 0.4% (0.0%, 0.9%) 3.5% (2.2%, 4.7%) 0.1% (-0.6%, 0.8%) | 1.00, 6.00 1.564 (47.4%) 833 (25.3%) 481 (14.6%) 290 (8.8%) 871 (26.4%) 156 (4.7%) 2.132 (64.7%) 1.100 (33.4%) 706 (21.4%) 463 (14.0%) 1.139 (34.5%) 212 (6.4%) 2.392 (72.6%) 110 (3.3%) 1.076 (32.6%) 1.847 (56.0%) 1.112 (33.7%) 20 (0.6%) 637 (19.3%) 352 (10.7%) 33 (1.0%) 144 (12.6%) 108 (3.3%) | 1.00, 7.00 1.570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 699 (21.2%) 459 (13.9%) 1,150 (34.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) 341 (10.%) 411 (12.5%) 102 (3.1%) | -(·, ·) -(·, · |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of DPP-4i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of SGLT-2i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SGLT-2i; n (%) Past use of SGLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ARNI; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Beta-blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) Intravenous diuretics; n (%) Intravenous diuretics; n (%) Statins; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3,437 (64.6%) 2.139 (40.2%) 1.414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3,923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) 54 (1.0%) 1,226 (23.0%) 564 (10.6%) 764 (14.4%) 184 (3.5%) 1,87 (59.9%) 184 (3.5%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3.642 (71.2%) 168 (3.3%) 1.753 (34.3%) 2,743 (53.6%) 1.641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) 52 (1.0%) 557 (10.9%) 171 (3.3%) 3,994 (78.1%) | -(·, -) 1.6% (-3.5%, 0.4%) 7.9% (6.2%, 9.6%) 6.9% (5.5%, 8.3%) 0.9% (-0.2%, 2.0%) -0.5% (-2.2%, 1.1%) 1.1% (0.3%, 1.9%) 0.8% (-1.1%, 2.6%) 12.4% (10.6%, 14.2%) 9.2% (7.6%, 10.8%) 1.6% (0.3%, 3.0%) 1.0% (-0.9%, 2.8%) 2.5% (0.7%, 4.2%) 0.2% (-0.5%, 1.0%) -2.3% (-4.2%, -0.5%) 6.2% (4.3%, 8.1%) 4.0% (2.2%, 5.8%) 0.3% (-0.1%, 0.7%) 4.6% (3.1%, 6.2%) 0.0% (-1.2%, 1.2%) 0.4% (0.0%, 0.9%) 3.5% (2.2%, 4.7%) 0.1% (-0.6%, 0.8%) 5.6% (4.1%, 7.1%) | 1.00, 6.00 1,564 (47.4%) 833 (25.3%) 481 (14.6%) 290 (8.8%) 871 (26.4%) 156 (4.7%) 1,132 (64.7%) 1,100 (33.4%) 706 (21.4%) 463 (14.0%) 1,139 (34.5%) 212 (6.4%) 10 (3.3%) 1,076 (32.6%) 1,147 (56.0%) 1,112 (33.7%) 20 (0.6%) 637 (19.3%) 352 (10.7%) 33 (1.0%) 414 (12.6%) 108 (3.3%) 2,666 (80.9%) | 1.00, 7.00 1.570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2.144 (65.0%) 1.094 (33.2%) 699 (21.2%) 459 (13.9%) 1.150 (34.9%) 218 (6.6%) 2.363 (71.7%) 119 (3.6%) 1.089 (33.0%) 1.866 (56.6%) 1.120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) 34 (1.0%) 411 (12.5%) 102 (3.1%) 2,665 (80.8%) | -(·,·) -(·,·) -(·,·) -(·,·) -(·,·) -(·,·) -(·,·) -(.2% (-2.6%, 2.3%) 0.2% (-1.5%, 2.3%) 0.2% (-1.5%, 2.3%) 0.2% (-1.5%, 1.3%) -0.3% (-2.5%, 1.8%) 0.1% (-1.0%, 1.1%) -0.4% (-2.7%, 2.0%) 0.2% (-2.1%, 2.5%) 0.2% (-1.1%, 2.2%) 0.1% (-1.6%, 1.8%) -0.3% (-2.7%, 2.0%) -0.2% (-1.4%, 1.0%) 0.9% (-1.3%, 3.1%) -0.3% (-1.2%, 0.6%) -0.4% (-2.7%, 1.9%) -0.6% (-3.0%, 1.8%) -0.2% (-2.6%, 2.1%) -0.1% (-0.5%, 0.3%) -0.6% (-2.5%, 1.4%) 0.4% (-1.1%, 1.9%) -0.0% (-0.5%, 0.5%) 0.1% (-1.5%, 1.7%) 0.2% (-0.7%, 1.1%) 0.0% (-1.9%, 2.0%) |
| median [IQR]min, max Concomitant use or initiation of Metformin; n (%) Concomitant use or initiation of Insulins; n (%) Concomitant use or initiation of Sulfonylureas; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of SPP-4i; n (%) Concomitant use or initiation of Any other glucose-lowering drugs; n (%) Past use of Metformin; n (%) Past use of Metformin; n (%) Past use of Sulfonylureas; n (%) Past use of Sulfonylureas; n (%) Past use of SOLT-2i; n (%) Past use of SOLT-2i; n (%) Past use of Any other glucose-lowering drugs; n (%) ACE-is/ARB's; n (%) ARNI; n (%) Thiazides; n (%) Beta-blockers; n (%) Calcium channel blockers; n (%) Digoxin / Digitoxin; n (%) Loop diuretics; n (%) Intravenous diuretics; n (%) Nitrates; n (%) Statins; n (%) PCSK9 inhibitors and other lipid-lowering drugs; n (%) | 2.00 [2.00, 3.00] 1.00, 6.00 2.418 (45.4%) 1.554 (29.2%) 984 (18.5%) 481 (9.0%) 1.320 (24.8%) 285 (5.4%) 3.437 (64.6%) 2.139 (40.2%) 1,414 (26.6%) 775 (14.6%) 1,794 (33.7%) 414 (7.8%) 3.923 (73.7%) 188 (3.5%) 1,700 (31.9%) 3,187 (59.9%) 1,921 (36.1%) 54 (1.0%) 1,226 (23.0%) 564 (10.6%) 78 (1.5%) 764 (14.4%) 184 (3.5%) 4,455 (83.7%) 995 (18.7%) | 1.00, 7.00 2.402 (47.0%) 1.089 (21.3%) 592 (11.6%) 417 (8.2%) 1.296 (25.3%) 217 (4.2%) 3.263 (63.8%) 1.421 (27.8%) 889 (17.4%) 661 (12.9%) 1.674 (32.7%) 303 (5.9%) 3,642 (71.2%) 168 (3.3%) 1,753 (34.3%) 2,743 (53.6%) 1,641 (32.1%) 36 (0.7%) 940 (18.4%) 541 (10.6%) 52 (1.0%) 557 (10.9%) 171 (3.3%) 3,994 (78.1%) 923 (18.0%) | -(-, -) -(-, - | 1.00, 6.00 1,564 (47.4%) 833 (25.3%) 481 (14.6%) 290 (8.8%) 871 (26.4%) 156 (4.7%) 1,100 (33.4%) 706 (21.4%) 463 (14.0%) 1,139 (34.5%) 212 (6.4%) 1,107 (33.3%) 1,076 (32.6%) 1,112 (33.7%) 20 (0.6%) 637 (19.3%) 352 (10.7%) 33 (1.0%) 414 (12.6%) 108 (3.3%) 2,666 (80.9%) 606 (18.4%) | 1.00, 7.00 1.570 (47.6%) 827 (25.1%) 473 (14.3%) 293 (8.9%) 882 (26.8%) 154 (4.7%) 2,144 (65.0%) 1,094 (33.2%) 459 (13.9%) 218 (6.6%) 2,363 (71.7%) 119 (3.6%) 1,089 (33.0%) 1,866 (56.6%) 1,120 (34.0%) 24 (0.7%) 656 (19.9%) 340 (10.3%) 34 (1.0%) 411 (12.5%) 102 (3.1%) 608 (18.4%) | -(-, -) -(-, - |

| COPD/Asthma medications; n (%) | 1,878 (35.3%) | 2,006 (39.2%) | -4.0% (-5.8%, -2.1%) | 1,220 (37.0%) | 1,218 (36.9%) | 0.1% (-2.3%, 2.4%) |
|---|---|---|---|---|---|---|
| NSAIDS; n (%) | 1,506 (28.3%) | 1,762 (34.5%) | -6.2% (-8.0%, -4.4%) | 1,052 (31.9%) | 1,040 (31.5%) | 0.4% (-1.9%, 2.6%) |
| Oral corticosteroids; n (%) | 1,359 (25.5%) | 1,571 (30.7%) | -5.2% (-6.9%, -3.5%) | 932 (28.3%) | 894 (27.1%) | 1.2% (-1.0%, 3.3%) |
| Osteoporosis agents (incl. bisphosphonates); n (%) | 110 (2.1%) | 86 (1.7%) | 0.4% (-0.2%, 0.9%) | 66 (2.0%) | 67 (2.0%) | -0.0% (-0.7%, 0.7%) |
| Opioids; n (%) | 1,147 (21.5%) | 1,135 (22.2%) | -0.7% (-2.3%, 1.0%) | 722 (21.9%) | 688 (20.9%) | 1.0% (-1.0%, 3.0%) |
| Anti-depressants; n (%) | 1,928 (36.2%) | 1,981 (38.7%) | -2.5% (-4.4%, -0.6%) | 1,218 (36.9%) | 1,237 (37.5%) | -0.6% (-2.9%, 1.8%) |
| Antipsychotics; n (%) | 170 (3.2%) | 167 (3.3%) | -0.1% (-0.8%, 0.6%) | 107 (3.2%) | 101 (3.1%) | 0.2% (-0.7%, 1.1%) |
| Anxiolytics / hypnotics, benzos; n (%) | 973 (18.3%) | 1,197 (23.4%) | -5.1% (-6.7%, -3.6%) | 668 (20.3%) | 684 (20.7%) | -0.5% (-2.5%, 1.5%) |
| Dementia medications; n (%) | 118 (2.2%) | 36 (0.7%) | 1.5% (1.0%, 2.0%) | 31 (0.9%) | 32 (1.0%) | -0.0% (-0.5%, 0.5%) |
| Urinary tract infections antibiotics; n (%) | 2,479 (46.6%) | 2,571 (50.3%) | -3.7% (-5.6%, -1.8%) | 1,565 (47.5%) | 1,543 (46.8%) | 0.7% (-1.8%, 3.1%) |
| Laxatives; n (%) | 161 (3.0%) | 186 (3.6%) | -0.6% (-1.3%, 0.1%) | 104 (3.2%) | 101 (3.1%) | 0.1% (-0.8%, 1.0%) |
| Number of distinct medications | 101 (6.070) | 100 (0.070) | 0.070 ( 2.070, 0.270) | 10 1 (0.1270) | 101 (0.170) | 0.270 ( 0.070, 2.070) |
| mean (sd) | 15.36 (6.48) | 15.49 (6.74) | -0.14 (-0.39, 0.12) | 15.30 (6.66) | 15.25 (6.43) | 0.04 (-0.27, 0.36) |
| median [IQR] | 15.00 [11.00, 19.00] | 15.00 [11.00, 19.00] | - (-, -) | 15.00 [11.00, 19.00] | 14.00 [11.00, 19.00] | - (-, -) |
| | 1.00, 50.00 | 1.00, 51.00 | - (-, -)<br>- (-, -) | 1.00, 50.00 | 1.00, 51.00 | - (-, -)<br>- (-, -) |
| min, max | 1.00, 50.00 | 1.00, 51.00 | - (-, -) | 1.00, 50.00 | 1.00, 51.00 | - (-, -) |
| Number of office visits | | | | | | |
| mean (sd) | 10.94 (7.17) | 11.00 (7.13) | -0.06 (-0.33, 0.22) | 10.79 (7.26) | 10.69 (6.86) | 0.10 (-0.24, 0.44) |
| median [IQR] | 9.00 [6.00, 14.00] | 9.00 [6.00, 14.00] | - (-, -) | 9.00 [6.00, 14.00] | 9.00 [6.00, 14.00] | - (-, -) |
| min, max | 0.00, 66.00 | 0.00, 101.00 | - (-, -) | 0.00, 66.00 | 0.00, 55.00 | - (-, -) |
| Number of endocrinologist visits | | | | | | |
| mean (sd) | 0.64 (1.70) | 0.52 (1.41) | 0.12 (0.06, 0.18) | 0.56 (1.53) | 0.56 (1.50) | -0.00 (-0.08, 0.07) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 30.00 | 0.00, 27.00 | - (-, -) | 0.00, 20.00 | 0.00, 27.00 | - (-, -) |
| Number of cardiologist visits | | | | | | |
| mean (sd) | 2.43 (4.02) | 2.08 (3.48) | 0.34 (0.20, 0.49) | 2.14 (3.70) | 2.12 (3.51) | 0.02 (-0.16, 0.19) |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max | 0.00, 50.00 | 0.00, 48.00 | - (-, -) | 0.00, 50.00 | 0.00, 44.00 | - (-, -) |
| Number of internal/family medicine visits | | | | | | |
| mean (sd) | 6.33 (7.78) | 5.56 (5.91) | 0.78 (0.51, 1.04) | 5.59 (7.05) | 5.61 (5.90) | -0.03 (-0.34, 0.29) |
| median [IQR] | 4.00 [2.00, 8.00] | 4.00 [2.00, 7.00] | - (-, -) | 4.00 [2.00, 7.00] | 4.00 [2.00, 7.00] | - (-, -) |
| min, max | 0.00, 216.00 | 0.00, 94.00 | - (-, -) | 0.00, 216.00 | 0.00, 60.00 | - (-, -) |
| Number of Electrocardiograms (ECG/EKG) | | | 1 | | | · · · / |
| mean (sd) | 1.43 (2.01) | 1.24 (1.73) | 0.20 (0.12, 0.27) | 1.30 (1.85) | 1.28 (1.79) | 0.02 (-0.07, 0.11) |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) |
| min, max | 0.00, 28.00 | 0.00, 23.00 | - (-, -) | 0.00, 28.00 | 0.00, 23.00 | - (-, -) |
| Number of Echocardiograms | 0.00, 28.00 | 0.00, 23.00 | - (-, -) | 0.00, 28.00 | 0.00, 23.00 | - (-, -) |
| mean (sd) | 0.51 (0.92) | 0.43 (0.81) | 0.08 (0.04, 0.11) | 0.45 (0.84) | 0.44 (0.82) | 0.01 (-0.03, 0.05) |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | |
| | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) | 0.00, 11.00 | 0.00 [0.00, 1.00] | - (-, -)<br>- (-, -) |
| min, max | 0.00, 11.00 | 0.00, 9.00 | - (-, -) | 0.00, 11.00 | 0.00, 9.00 | - (-, -) |
| Out-of-pocket medication cost | COC 07 (1 000 00) | C4454(140440) | 27.57 ( 70.05, 2.75) | CO 4 OO (4 O 40 OE) | COO OC (COO OT) | 0.00 / 41 40 50 0 4) |
| mean (sd) | 606.97 (1,022.30) | 644.54 (1,124.49) | -37.57 (-78.85, 3.71) | 634.32 (1,049.85) | 628.06 (920.97) | 6.26 (-41.42, 53.94) |
| median [IQR] | 379.82 [175.86, 765.84] | 379.12 [150.00, 805.88] | - (-, -) | 385.12 [167.24, 780.44] | 371.38 [154.90, 811.08] | - (-, -) |
| min, max | -33,195.00, 22,108.03 | -1,425.00, 30,361.78 | - (-, -) | -445.00, 22,108.03 | -1,425.00, 19,162.24 | - (-, -) |
| Unique brand medicines | | | | | | |
| mean (sd) | 15.65 (6.70) | 15.77 (6.94) | -0.12 (-0.38, 0.14) | 15.58 (6.88) | 15.53 (6.60) | 0.05 (-0.27, 0.38) |
| median [IQR] | 15.00 [11.00, 19.00] | 15.00 [11.00, 20.00] | - (-, -) | 15.00 [11.00, 19.00] | 15.00 [11.00, 19.00] | - (-, -) |
| min, max | 1.00, 52.00 | 1.00, 54.00 | - (-, -) | 1.00, 52.00 | 1.00, 54.00 | - (-, -) |
| Unique generic medicines | | | | | | |
| mean (sd) | 15.36 (6.48) | 15.49 (6.74) | -0.14 (-0.39, 0.12) | 15.30 (6.66) | 15.25 (6.43) | 0.04 (-0.27, 0.36) |
| median [IQR] | 15.00 [11.00, 19.00] | 15.00 [11.00, 19.00] | - (-, -) | 15.00 [11.00, 19.00] | 14.00 [11.00, 19.00] | - (-, -) |
| min, max | 1.00, 50.00 | 1.00, 51.00 | - (-, -) | 1.00, 50.00 | 1.00, 51.00 | - (-, -) |
| Colonoscopy Sigmoidoscopy; n (%) | 594 (11.2%) | 649 (12.7%) | -1.5% (-2.8%, -0.3%) | 389 (11.8%) | 387 (11.7%) | 0.1% (-1.5%, 1.6%) |
| Flu Pneumococcal vaccine; n (%) | 1,840 (34.6%) | 1,429 (27.9%) | 6.6% (4.8%, 8.4%) | 1,021 (31.0%) | 983 (29.8%) | 1.2% (-1.1%, 3.4%) |
| Pap smear; n (%) | 329 (6.2%) | 503 (9.8%) | -3.7% (-4.7%, -2.6%) | 254 (7.7%) | 256 (7.8%) | -0.1% (-1.4%, 1.3%) |
| PSA test; n (%) | 1,337 (25.1%) | 1,386 (27.1%) | -2.0% (-3.7%, -0.3%) | 864 (26.2%) | 849 (25.8%) | 0.5% (-1.7%, 2.6%) |
| Fecal occult blood test; n (%) | 196 (3.7%) | 202 (3.9%) | -0.3% (-1.0%, 0.5%) | 124 (3.8%) | 128 (3.9%) | -0.1% (-1.1%, 0.8%) |
| Bone mineral density tests; n (%) | 250 (4.7%) | 264 (5.2%) | -0.5% (-1.3%, 0.4%) | 151 (4.6%) | 158 (4.8%) | -0.2% (-1.3%, 0.8%) |
| Mammograms; n (%) | 1.153 (21.7%) | 1.338 (26.2%) | -4.5% (-6.2%, -2.9%) | 794 (24.1%) | 808 (24.5%) | -0.4% (-2.5%, 1.7%) |
| Telemedicine; n (%) | 1,601 (30.1%) | 1,575 (30.8%) | -0.7% (-2.5%, 1.1%) | 1,002 (30.4%) | 985 (29.9%) | 0.5% (-1.7%, 2.8%) |
| HbA1C tests | , () | \/ | ( =.=.:, =.=/0) | , | | |
| mean (sd) | 2.36 (1.49) | 2.34 (1.54) | 0.02 (-0.04, 0.07) | 2.33 (1.46) | 2.35 (1.52) | -0.01 (-0.09, 0.06) |
| mean (sa) | 2.00 (I.TJ) | として (エンマ) | 0.02 ( 0.07, 0.07) | 2.00 (1.70) | L.JJ (1.JL) | 0.01 (-0.00, 0.00) |

| | T | | T | T | | |
|---|---|---|---|---|---|---|
| median [IQR] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | - (-, -) |
| min, max | 0.00, 26.00 | 0.00, 31.00 | - (-, -) | 0.00, 26.00 | 0.00, 31.00 | - (-, -) |
| Lipid panels | | | | | | |
| mean (sd) | 1.60 (1.28) | 1.76 (1.38) | -0.16 (-0.21, -0.11) | 1.69 (1.33) | 1.68 (1.24) | 0.01 (-0.06, 0.07) |
| median [IQR] | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | - (-, -) | 1.00 [1.00, 2.00] | 2.00 [1.00, 2.00] | - (-, -) |
| min, max | 0.00, 22.00 | 0.00, 29.00 | - (-, -) | 0.00, 22.00 | 0.00, 12.00 | - (-, -) |
| Creatinine tests | | | | | | |
| mean (sd) | 0.06 (0.35) | 0.04 (0.28) | 0.02 (0.01, 0.03) | 0.05 (0.31) | 0.05 (0.30) | 0.00 (-0.01, 0.02) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 8.00 | 0.00, 6.00 | - (-, -) | 0.00, 6.00 | 0.00, 6.00 | - (-, -) |
| Natriuretic peptide tests | | | | | | |
| mean (sd) | 0.22 (0.87) | 0.20 (0.98) | 0.02 (-0.02, 0.05) | 0.21 (0.88) | 0.20 (0.94) | 0.01 (-0.03, 0.06) |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 20.00 | 0.00, 28.00 | - (-, -) | 0.00, 18.00 | 0.00, 27.00 | - (-, -) |
| Urine tests | | | | | | |
| mean (sd) | 1.10 (1.85) | 1.13 (1.85) | -0.03 (-0.10, 0.05) | 1.09 (1.86) | 1.06 (1.77) | 0.04 (-0.05, 0.12) |
| median [IQR] | 0.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | - (-, -) | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | - (-, -) |
| min, max | 0.00, 30.00 | 0.00, 33.00 | - (-, -) | 0.00, 29.00 | 0.00, 28.00 | - (-, -) |
| Combined comorbidity score | 0.00,00.00 | 0.00,00.00 | ( , / | 0.00, 20.00 | 0.00, 20.00 | ( , , |
| mean (sd) | 2.34 (2.50) | 1.78 (2.02) | 0.57 (0.48, 0.65) | 1.93 (2.15) | 1.91 (2.10) | 0.02 (-0.08, 0.12) |
| median [IQR] | 2.00 [1.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | - (-, -) |
| min, max | -2.00, 20.00 | -1.00, 16.00 | - (-, -) | -2.00, 15.00 | -1.00, 13.00 | - (-, -) |
| Frailty Score | -2.00, 20.00 | -1.00, 10.00 | - (-, -) | -2.00, 13.00 | -1.00, 13.00 | - (-, -) |
| mean (sd) | 0.18 (0.05) | 0.16 (0.04) | 0.01 (0.01, 0.01) | 0.17 (0.05) | 0.17 (0.05) | 0.00 (-0.00, 0.00) |
| median [IQR] | 0.17 [0.14, 0.20] | 0.16 (0.13, 0.19) | - (-, -) | 0.16 [0.14, 0.19] | 0.16 [0.14, 0.19] | - (-, -) |
| min, max | 0.06, 0.55 | 0.04, 0.47 | - (-, -)<br>- (-, -) | 0.06, 0.48 | 0.04, 0.43 | - (-, -)<br>- (-, -) |
| Number of Hospitalizations | 0.00, 0.55 | 0.04, 0.47 | - (-, -) | 0.00, 0.46 | 0.04, 0.43 | - (-, -) |
| mean (sd) | 10.50 (32.68) | 6.19 (25.28) | 4.31 (3.19, 5.43) | 7.49 (27.27) | 7.19 (26.84) | 0.30 (-1.01, 1.61) |
| ` ' | | | | 0.00 [0.00, 0.00] | | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | - (-, -) | | 0.00 [0.00, 0.00] | - (-, -) |
| min, max | 0.00, 552.00 | 0.00, 482.00 | - (-, -) | 0.00, 552.00 | 0.00, 444.00 | - (-, -) |
| Any hospitalization within prior 91 days; n (%) | 257 (4.8%) | 147 (2.9%) | 2.0% (1.2%, 2.7%) | 122 (3.7%) | 107 (3.2%) | 0.5% (-0.5%, 1.4%) |
| Any hospitalization within prior 92-365 days; n (%) | 752 (14.1%) | 468 (9.2%) | 5.0% (3.7%, 6.2%) | 344 (10.4%) | 343 (10.4%) | 0.0% (-1.5%, 1.5%) |
| Number of hospitalizations (0, 1, 2 or more) | | . === :== ==: | | | | |
| < 1; n (%) | 4,402 (82.7%) | 4,552 (89.0%) | -6.3% (-7.7%, -5.0%) | 2,867 (87.0%) | 2,882 (87.4%) | -0.5% (-2.1%, 1.2%) |
| 1 - <2; n (%) | 45 (0.8%) | 30 (0.6%) | 0.3% (-0.1%, 0.6%) | 17 (0.5%) | 22 (0.7%) | -0.2% (-0.6%, 0.2%) |
| >= 2; n (%) | 877 (16.5%) | 532 (10.4%) | 6.1% (4.7%, 7.4%) | 413 (12.5%) | 393 (11.9%) | 0.6% (-1.0%, 2.2%) |
| Heart failure hospitalization; n (%) | 304 (5.7%) | 144 (2.8%) | 2.9% (2.1%, 3.7%) | 118 (3.6%) | 106 (3.2%) | 0.4% (-0.5%, 1.3%) |
| ED visit; n (%) | 2,230 (41.9%) | 1,894 (37.0%) | 4.9% (3.0%, 6.7%) | 1,267 (38.4%) | 1,249 (37.9%) | 0.5% (-1.8%, 2.9%) |
| Acute MI; n (%) | 164 (3.1%) | 109 (2.1%) | 0.9% (0.3%, 1.6%) | 80 (2.4%) | 82 (2.5%) | -0.1% (-0.8%, 0.7%) |
| Old MI; n (%) | 273 (5.1%) | 236 (4.6%) | 0.5% (-0.3%, 1.4%) | 165 (5.0%) | 159 (4.8%) | 0.2% (-0.9%, 1.3%) |
| Heart failure; n (%) | 944 (17.7%) | 618 (12.1%) | 5.6% (4.3%, 7.0%) | 461 (14.0%) | 452 (13.7%) | 0.3% (-1.4%, 2.0%) |
| A cute heart failure; n (%) | 228 (4.3%) | 136 (2.7%) | 1.6% (0.9%, 2.3%) | 99 (3.0%) | 92 (2.8%) | 0.2% (-0.6%, 1.1%) |
| Microalbuminuria or proteinuria; n (%) | 267 (5.0%) | 207 (4.0%) | 1.0% (0.2%, 1.8%) | 130 (3.9%) | 143 (4.3%) | -0.4% (-1.4%, 0.6%) |
| Ratio of brand to generic medications | | | | | | |
| mean (sd) | 1.02 (0.04) | 1.02 (0.04) | 0.00 (-0.00, 0.00) | 1.02 (0.04) | 1.02 (0.04) | -0.00 (-0.00, 0.00) |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | - (-, -) |
| min, max | 0.89, 1.35 | 0.89, 1.33 | - (-, -) | 0.89, 1.35 | 0.89, 1.33 | - (-, -) |

## Variable\_name

Age

Gender

Race

Region

Smoking / Tobacco use

Underweight

Normal weight, if BMI is 20.0-24.9 Overweight, if BMI is 25.0 to 29.9

Class 1 (low-risk) obesity, if BMI is 30.0 to 34.9

Class 2 (moderate-risk) obesity, if BMI is 35.0 to 39.9

Class 3 (high-risk) obesity if BMI is equal to or greater than 40

Unspecified obesity

Diabetic retinopathy

Diabetic neuropathy

Diabetic nephropathy

Diabetes with other opthalmic complications

Diabetes with peripheral circulatory disorders

Diabetic foot

Erectile dysfuntion

Hypoglycemia

Hyperglycemia/DKA/HONK

Skin infections

Stable angina

Unstable angina

Hypertension

Hypotension

Hyperlipidemia

Atrial fibrillation

Acute myocardial infarction
Old myocardial infarction

Cardiac conduction disorder

Previous cardiac procedure (CABG, PTCA, Stent)

Ischemic stroke

PVD diagnosis or surgery

## Algorithm sources

If region not available, from State, https://www2.census.gov/geo/pdfs/maps-data/maps/reference/us\_regdiv.pdf

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://pubmed.ncbi.nlm.nih.gov/34953068/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9154288/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3721171/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

 $\underline{Investigator\ review\ of\ codes\ based\ on:\ https://pubmed.ncbi.nlm.nih.gov/34338404/}$ 

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34338404/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/books/NBK368403/table/sb203.t5/, https://www.health.mil/Reference-

Center/Publications/2016/03/01/Diabetes-Mellitus, http://www.icd9data.com/2014/Volume1/240-279/249-259/250/default.htm,

https://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-

Investigator review of codes based on: (modified codes) https://pubmed.ncbi.nlm.nih.gov/36102675/

Investigator review of codes based on: the paper then used ICD9/ICD10 website to expand it, https://www.icd10data.com/ICD10CM/Codes/N00-N99/N40-

N53/N52-, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4857901/

 $Investigator\ review\ of\ codes\ based\ on:\ https://pubmed.ncbi.nlm.nih.gov/34953068/,\ https://pubmed.ncbi.nlm.nih.gov/35043165/,\ https://pubmed.ncbi.nlm.nih.gov/34953068/,\ https://pubmed.ncbi$ 

Investigator review of codes based on:

Hyperglycemia: https://pubmed.ncbi.nlm.nih.gov/34953068/, https://pubmed.ncbi.nlm.nih.gov/35043165/

DKA: https://pubmed.ncbi.nlm.nih.gov/29773640/, https://pubmed.ncbi.nlm.nih.gov/38262528/

HONK: https://dam.assets.ohio.gov/image/upload/medicaid.ohio.gov/Providers/PaymentInnovation/DEF/DKA.pdf

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/34953068/, ICD9 to ICD10 conversion

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/19337843/, https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/

 $Investigator\ review\ of\ codes\ based\ on:\ https://pubmed.ncbi.nlm.nih.gov/19337843/,\ https://pmc.ncbi.nlm.nih.gov/articles/PMC9172873/nd-ncbi.nlm.nih.gov/articl$ 

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC8064679/

 $Investigator\ review\ of\ codes\ based\ on:\ https://pubmed.ncbi.nlm.nih.gov/35043165/,\ https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-approximation and the sentinels of the sentinels of$ 

 $packages/browse? at = refs\%2 Fheads\%2 Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_sir\_wp002, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse.$ 

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/31933524/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/24682186/

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html,

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1.pdf, ICD9 to ICD10 conversion

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes, https://www.icd10data.com/

Other cardiac dysrhythmia

Heart failure

Acute heart failure

Microalbuminuria/proteinuria

Cardiomyopathy

Valve disorders

Valve replacement

TIA

Edema

Venous thromboembolism/ pulmonary embolsim

Pulmonary hypertension

Implantable cardioverter defibrillator

Hyperkalemia

Coronary atherosclerosis

Cerebrovascular procedure

Insertion of pacemakers / removal of cardiac lead

CKD stage 1-2

CKD stage 3-4

Unspecified CKD

Acute kidney injury

Hypertensive nephropathy

Urinary tract infections

Genital infections

Urolithiasis (kidney or urinary stones)

COPD

Asthma

Obstructive sleep apnea

Serious bacterial infections

Pneumonia Liver disease

MASH/MASLD

Fractures / Falls

Osteoporosis

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf,

 $https://www.health.ny.gov/health\_care/medicaid/redesign/dsrip/vbp\_library/docs/arrblk.pdf, https://www.cdc.gov/dhdsp/maps/atlas/data-sources.html, https://www.cdc.gov/dhdsp/maps/atlas/data-sources$ 

https://www.cms.gov/medicare/coding/icd10/downloads/icd10clinicalconceptscardiology1.pdf, ICD9 to ICD10 conversion

Investigator review of codes

Investigator review of codes

Modified codes based on inclusion criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

Investigator review of codes based on: https://stacks.cdc.gov/view/cdc/31381/cdc\_31381\_DS8.pdf, https://pubmed.ncbi.nlm.nih.gov/38440888/,

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8751938/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

 $packages/browse? at = refs\%2 Fheads\%2 Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse? at = refs\%2 Fheads\%2 Fcder\_mpl2p\_wp015, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse.$ 

packages/browse?at=cder\_mpl2p\_wp009

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleid=52993&ver=45&

Investigator review of codes based on: https://www.sciencedirect.com/science/article/pii/S2666572723000251

Investigator review of codes

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

https://pmc.ncbi.nlm.nih.gov/articles/PMC4399109/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC10251803/

Investigator review of codes, https://www.icd10data.com/

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC2978782/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC5888226/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8929186/

Investigator review of codes based on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637,

https://www.kidneymedicinejournal.org/cms/10.1016/j.xkme.2022.100414/attachment/5e29ab67-7a7d-4621-9af3-81bd071bbc67/mmc1.pdf,

https://www.icd10data.com/ICD10CM/Codes/I00-I99

Investigator reviewed code based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7558992/#app1-antibiotics-09-00536

Investigator reviewed codes based on: https://pubmed.ncbi.nlm.nih.gov/30207042/

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC7793999/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/, modified CCW algorithm (any care setting, any diagnosis

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8636332/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7927325/

https://pubmed.ncbi.nlm.nih.gov/29921683/, https://pubmed.ncbi.nlm.nih.gov/17346615/, https://pubmed.ncbi.nlm.nih.gov/23335588/

Investigator review of codes based on: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10203971/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002,

 $\frac{https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs\%2Fheads\%2Fcder\_mpl2p\_wp015, Modified algorightm from https://pubmed.ncbi.nlm.nih.gov/34256144/, Modified CCW algorithm$ 

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/32300995/, https://pubmed.ncbi.nlm.nih.gov/39316292/

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp009,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015,

https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=cder\_mpl2p\_wp010

https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8202643/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-likely-like

packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, CCW Algorithms

Osteoarthritis Depression

Dementia

Delirium or psychosis

Anxiety

Sleep disorder

Anemia

Influenza

COVID-19

Hyperthyroidism and other thyroid gland disorders

Hypothyroidism Nephrotic syndrome

Urinary incontinence

Biliary disease

Pancreatitis

Bowel obstruction

Gastroparesis

Number of antidiabetic drugs on CED

Concomitant use or initiation of metformin

Concomitant use or initiation of insulin

Concomitant use or initiation of sulfonylureas

Concomitant use or initiation of DPP4i

Concomitant use or initiation of SGLT2i

Concomitant use or initiation of other glucose-lowering drugs

Past use of metformin

Past use of insulin

Past use of sulfonylureas

Past use of DPP4i

Past use of SGLT2i

Past use of other glucose-lowering drugs

ACEi / ARB

ARNI

Thiazides

Beta-Blockers

Calcium channel blockers

Digoxin / Digitoxin

Loop diuretics

Other diuretics

Intravenous diuretics

Nitrates

Modified CCW algorithm

https://pubmed.ncbi.nlm.nih.gov/35043165/, CCW Algorithms

https://pubmed.ncbi.nlm.nih.gov/35043165/, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-

packages/browse?at=refs%2Fheads%2Fcder\_mpl2p\_wp015

https://pubmed.ncbi.nlm.nih.gov/28485014/, https://pubmed.ncbi.nlm.nih.gov/35043165/

https://pubmed.ncbi.nlm.nih.gov/35043165/

Investigator review of codes based on https://www.verywellhealth.com/sleeping-disorders-list-and-diagnostic-codes-3014779

Modified codes based on eligibility criteria, here we implement any care setting, any diagnosis position

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38556924/

https://pubmed.ncbi.nlm.nih.gov/34913208/, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8427377/

 $\underline{Investigator\ review\ of\ codes\ based\ on:\ https://www.cms.gov/icd10m/version37-fullcode\_cms/P0244.html}$ 

Investigator review of codes based on: https://pmc.ncbi.nlm.nih.gov/articles/PMC10478599/

 $Investigator\ review\ of\ codes\ based\ on: https://nccd.cdc.gov/ckd/Methods.aspx?Qnum=Q637, https://www.cms.gov/icd10m/FY2024-nprmversion41.0-fullcode-linearity-f$ 

cms/fullcode\_cms/P2401.html

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/38527324/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/37796527/, https://pubmed.ncbi.nlm.nih.gov/35851329/,

https://pmc.ncbi.nlm.nih.gov/articles/PMC3985913/, https://pubmed.ncbi.nlm.nih.gov/38503905/, https://pubmed.ncbi.nlm.nih.gov/35513234/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/36222554/, https://pubmed.ncbi.nlm.nih.gov/30287807/,

https://pubmed.ncbi.nlm.nih.gov/22262606/

Investigator review of codes based on: https://pubmed.ncbi.nlm.nih.gov/36798959/, https://pubmed.ncbi.nlm.nih.gov/28438588/,

https://pubmed.ncbi.nlm.nih.gov/31095068/

Investigator review of codes: https://pubmed.ncbi.nlm.nih.gov/34624355/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK513225/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK518983/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK278938/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK542331/

 $Investigator\ review\ of\ codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/NBK576405/nlm.nih.gov/books/nlm.nih.gov/boo$ 

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK551656/, https://pmc.ncbi.nlm.nih.gov/articles/PMC4882495/,

https://www.ncbi.nlm.nih.gov/books/NBK557848/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK507904/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK556025/, https://pubchem.ncbi.nlm.nih.gov/compound/441207

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Investigator review of codes

Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK9626/table/A66/

Anti-arrhythmics Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK482322/ (using class I and class II as class 2 is beta blockers and class 4 is calcium channel blockers) Statins Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterol-PCSK9 inhibitors and other lipid-lowering drugs Investigator review of codes, https://www.drugs.com, https://www.heart.org/en/health-topics/cholesterol/prevention-and-treatment-of-high-cholesterolhyperlipidemia/cholesterol-medications Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK537062/ Antiplatelet agents Oral anticoagulants Investigator review of codes, https://www.drugs.com, https://www.ahajournals.org/doi/full/10.1161/JAHA.120.017559 COPD/Asthma medication Investigator review of codes, https://www.copdfoundation.org/Learn-More/I-am-a-Person-with-COPD/Treatments-Medications.aspx, https://getasthmahelp.org/medications-list.aspx **NSAIDs** Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK547742/ Oral corticosteroids Investigator review of codes, https://www.drugs.com, https://www.aaaai.org/tools-for-the-public/drug-guide/oral-corticosteroid-medications Osteoporosis agents (incl. bisphosphonates) Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK470248/ Opioids Investigator review of codes, https://www.drugs.com, https://pubmed.ncbi.nlm.nih.gov/31643200/#:~:text=They%20can%20also%20be%20informally,%2C%20codeine%2C%20oxycodone%2C%20hydrocodone Anti-depressants Investigator review of codes, https://www.drugs.com, https://www.ncbi.nlm.nih.gov/books/NBK538182/ Antipsychotics Investigator review of codes, https://www.drugs.com Anxiolytics/hypnotics, benzodiazepines Investigator review of codes, https://www.drugs.com, https://www.dea.gov/sites/default/files/2020-06/Benzodiazepenes-2020.pdf, https://www.ncbi.nlm.nih.gov/books/NBK470159/, https://www.drugs.com Medication for dementia Investigator review of codes based on: https://www.drugs.com, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7462122/, https://go.drugbank.com/drugs/DB00382 Urinary tract infections antibiotics https://pubmed.ncbi.nlm.nih.gov/35790044/ Investigator review of codes, https://www.drugs.com Laxatives Number of distinct medications, median (iqr), mean (sd) N/A Number of office visits median (igr), mean (sd) https://www.cms.gov/files/document/mm13473-how-use-office-and-outpatient-evaluation-and-management-visit-complexity-add-code-g2211.pdf, https://www.cms.gov/files/document/physician-fee-schedule-pfs-payment-officeoutpatient-evaluation-and-management-em-visits-fact-sheet.pdf Number of endocrinologist visits, median (igr), mean (sd) Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-andcertification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Number of cardiologist visits, median (iqr), mean (sd) Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/MedicareProviderSupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-andcertification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf Number of internal medicine/family medicine visits, median (igr), mean (sd) Data dictionary of Optum, Marketscan and https://www.cms.gov/Medicare/Provider-Enrollment-and-Certification/Medicare Provider SupEnroll/downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-and-downloads/taxonomy.pdf, https://www.cms.gov/medicare/provider-enrollment-andcertification/medicareprovidersupenroll/downloads/taxonomycrosswalk.pdf https://www.cms.gov/medicare-coverage-database/view/article.aspx?articleld=57326, https://firstcoastbillinggroup.com/ekg-billing-and-reimbursement/, Number of electrocardiograms, median (iqr), mean (sd) https://www.aapc.com/codes/coding-newsletters/my-cardiology-coding-alert/cpt-answer-5-common-ecg-coding-questions-175952-article Number of echocardiograms, median (iqr), mean (sd) https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8511132/, https://pubmed.ncbi.nlm.nih.gov/34778785/, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56625&ver=27&, https://www.medicalbillgurus.com/echocardiogram-cpt-code/ Pharmacy out-of-pocket cost, median (igr), mean (sd) N/A Unique brand medications Investigator review of codes, https://www.drugs.com Unique generic medications Investigator review of codes, https://www.drugs.com Investigator review of codes, https://www.drugs.com Ratio of unique brand to generic medications https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002 Colonoscopy/ Sigmoidoscopy

Flu vaccine / Pneumococcal vaccine https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicarecoverage-database/view/article.aspx? article Id=54767&DocID=A54767, https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-aps/sentinel-analpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleId=54767&DocID=A54767 Pap smear test https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V72/default.htm, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htm, http://www.icd9data.com/2012/V01-V91/V70-V82/V76/default.htm, http://www.icd9data.com/2012/V01-V91 $\underline{https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analytic-packages/browse?at=refs\%2Fheads\%2Fcder\_sir\_wp002$ PSA test Fecal occult blood test Investigator review of codes N/A Bone mineral density tests Mammograms Investigator review of codes based on: https://dev.sentinelsystem.org/projects/AP/repos/sentinel-analyticpackages/browse?at=refs%2Fheads%2Fcder\_sir\_wp002, https://www.cms.gov/medicare-coveragedatabase/view/article.aspx?articleid=56448&ver=16&bc=0, http://www.icd9data.com/2012/Volume1/V01-V91/V70-V82/V76/default.htmTelemedicine  $Investigator\ review\ of\ codes\ based\ on:\ https://pubmed.ncbi.nlm.nih.gov/33151319/, https://www.cms.gov/newsroom/fact-sheets/medicare-telemedicine-health-newsroom/fact-sheets/medicare-teleme$ care-provider-fact-sheet, https://www.aafp.org/family-physician/practice-and-career/getting-paid/coding/coding-telehealth-audio-virtual-digital-visits.html Number of HbA1c tests, median (iqr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of lipid panels, median (iqr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of creatinine tests, median (igr), mean (sd) https://pubmed.ncbi.nlm.nih.gov/34953068/ Number of natriuretic peptide tests, median (iqr), mean (sd) Investigator review of codes Number of urine tests, median (iqr), mean (sd) Investigator review of codes HbA1c N/A N/A Glucose Creatinine N/A Systolic blood pressure N/A Heart rate N/A BMI N/A eGFR N/A LDL N/A HDL N/A Total cholesterol N/A N/A Triglycerides A combined comorbidity score predicted mortality in elderly patients better than existing scores, https://pubmed.ncbi.nlm.nih.gov/21208778/ Combined comorbidity score Frailty score Measuring Frailty in Medicare Data: Development and Validation of a Claims-Based Frailty Index, https://pubmed.ncbi.nlm.nih.gov/29244057/ Number of any hospitalization, median (iqr), mean (sd) N/A N/A Any hospitalization within prior 90 days; n (%) Any hospitalization within prior 91-365 days; n (%) N/A 0, 1, >1 hospitalizations (any) N/A Hospitalization for heart failure; n (%) N/A Number of emergency department visit median (igr), mean (sd) Different in all 3 databases and measure already created in all 3 as well; ED visit (Medicare): Revenue center codes: 0450, 0451, 0452, 0456, 0459, 0981; Place of service: 23 ED visit (Optum): Place of service: 23 ED visit (Marketscan): Service sub-category codes: 10120, 10220, 10320, 10420, 10520, 12220, 20120, 20220, 21120, 21220, 22120, 22320, 30120, 30220, 30320, 30420, 30520, 30620, 31120, 31220, 31320, 31420, 31520, 31620; Place of service: 23 Calendar year N/A